## PROTOCOL N01349 AMENDMENT 7

# ation and any extensions or variations thereof. A MULTICENTER, OPEN-LABEL, SINGLE-ARM STUDY TO **EVALUATE THE PHARMACOKINETICS, EFFICACY, AND** SAFETY OF BRIVARACETAM IN NEONATES WITH REPEATED ELECTROENCEPHALOGRAPHIC SEIZURES

## **PHASE 2/3**

EudraCT Number: 2015-002756-27

Sponsor:

UCB Biopharma SRL Allée de la Recherche 60 1070 Brussels **BELGIUM** 

| Protocol/Amendment number | Date | Type of amendment |
|---|---|---|
| Final Protocol | 14 Oct 2016 | Not applicable |
| Protocol Amendment (1.0) | 14 Dec 2016 | Non-Substantial |
| Protocol Amendment (2.0) | 28 Feb 2017 | Non-Substantial |
| Protocol Amendment (2.1, Germany) | 19 Jul 2017 | Non-Substantial |
| Protocol Amendment (2.2, Czech Republic) | 19 Jul 2017 | Non-Substantial |
| Protocol Amendment (3.0) | 23 Oct 2017 | Non-Substantial |
| Protocol Amendment (4.0) | 22 Jan 2018 | Non-Substantial |
| Protocol Amendment (5.0) | 10 Oct 2019 | Substantial |
| Protocol Amendment (6.0) | 28 Oct 2019 | Non-Substantial |
| Protocol Amendment (6.1, Germany) | 08 Nov 2019 | Non-Substantial |
| Protocol Amendment (6.2, Czech Republic) | 08 Nov 2019 | Non-Substantial |
| Protocol Amendment (6.3, France) | 07 Oct 2020 | Substantial |
| Protocol Amendment (6.4, Czech Republic) | 10 Nov 2020 | Substantial |
| Protocol Amendment (6.5, Germany) | 02 Dec 2020 | Substantial |
| Protocol Amendment (7.0) | 24 May 2021 | Substantial |

#### **Confidential Material**

#### Confidential

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


24 May 2021 N01349

## STUDY CONTACT INFORMATION

## **Sponsor**

UCB Biopharma SRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

## **Principal/Coordinating Investigator**

| | | 6. |
|---|---|---|
| _ | | reox. |
| e 60 | | ille, |
| | | ions |
| | | or variati |
| nating Investigator | ione | |
| Ronit Pressler, | , tens | |
| University College London | OT OT | |
| Gower Street 1 | dall | |
| London, WC1E 6BT | diffe | |
| United Kingdom | ion | |
| il C | 3 | |
| 27 200 | | |
| 2 | Ronit Pressler, University College London Gower Street 1 London, WC1E 6BT | Ronit Pressler, University College London Gower Street 1 London, WC1E 6BT |

## **Sponsor Study Physician**

| Name: | , <b>B</b> |
|----------|-------------------------------------------------------------------|
| Address: | UCB BioSciences, Inc. 8010 Arco Corporate Drive Raleigh, NC 27617 |
| | USA ACT |
| Phone: | |
| Fax: | |

## **Clinical Project Manager**

| Name. | , |
|----------|-----------------------------------------------|
| Address: | Alfred-Nobel-Strasse 10 40789 Monheim GERMANY |
| Phone: | |
| Fax: | |

## **Clinical Trial Biostatistician**

| Name: | , |
|---|---|
| Address: | UCB BioSciences, Inc. 8010 Arco Corporate Drive, Raleigh, NC 27617 |
| Phone: | USA |
| Fax: | |

## **Clinical Monitoring Contract Research Organization**

| Name: | PRA Health Sciences | of |
|----------|---------------------|---------|
| Address: | Green Park | Sill |
| | 500 South Oak Way | ario |
| | Reading, RG2 6AD | 700: |
| | United Kingdom | :;CALL |
| Phone: | +44 118 918 1000 | 1 appli |
| Fax: | +44 118 918 1001 | OR ion |

## **Data Monitoring Committee**

| Name: | BOLDIN | Affiliation/Job title: |
|-------|--------|-----------------------------------|
| | eting | Pediatric Clinical Pharmacologist |
| | diffe | Pediatric Neonatologist |
| 30 | | Pediatric Neonatologist |

| UCB<br>Clinical Study Protocol | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|
| SERIOUS ADVER | RSE EVENT REPORTING | |
| | Serious adverse event reporting (24h) | .0 |
| Fax | Europe: +32 238 66561 | Silver |
| Email | PSRapidalert@ucb.com | iation |
| ocument cannot be used to | Serious adverse event reporting (24h) Europe: +32 238 66561 PSRapidalert@ucb.com PSRapidalert@ucb.com | and any extensions |

## **TABLE OF CONTENTS**

| LIST OF ABBREVIATIONS | 10 |
|---|---|
| 1 SUMMARY | 12 |
| 2 INTRODUCTION | 15 |
| 2.1 Epidemiology and treatment of targeted disease | 15 |
| 2.2 Background information regarding product | 15 |
| 2.3 Rationale for the study | 17, |
| 3 STUDY OBJECTIVES | 48 |
| 3.1 Primary objective | |
| 3.2 Secondary objectives | 18 |
| 4 STUDY VARIABLES | 18 |
| 4.1 PK variables (Exploratory and Confirmatory Cohorts | 3)18 |
| 4.1.1 Primary PK variable | 18 |
| 4.1.2 Other PK variables | 18 |
| 4.2 Efficacy variables (Confirmatory Cohorts only) | 19 |
| 4.2.1 Secondary efficacy variables | <u>.;;;</u> ;;;;;;;;;;;;;;;;;;;;;;;;;;;;;; |
| 4.2.2 Other efficacy variables | 20 |
| 4.3 Safety variables (Exploratory and Confirmatory Coh | orts)21 |
| 4.3.1 Secondary safety variable | 21 |
| 4.3.2 Other safety variables | 21 |
| 5 STUDY DESIGN | 22 |
| 4.3 Safety variables (Exploratory and Confirmatory Coh 4.3.1 Secondary safety variable 4.3.2 Other safety variables 5 STUDY DESIGN 5.1 Study description 5.1.1 Exploratory Cohort | 22 |
| 5.1.1 Exploratory Cohort | 24 |
| 5.1.2 Confirmatory Cohorts | 25 |
| 5.1.3 Study duration per subject | 28 |
| 5.1.4 Planned number of subjects and sites | 28 |
| 5.1.5 Anticipated regions and countries | |
| 5.2 Schedule of study assessments | 29 |
| 5.3 Schematic diagrams | 40 |
| 5.4 Rationale for study design and selection of dose | 45 |
| 5.4.1 Rationale for study design | |
| 5.4.2 Rationale for dose selection | 45 |
| 6 SELECTION AND WITHDRAWAL OF SUBJECTS. | 47 |
| 61 Inclusion criteria | 47 |
| 6.2 Exclusion criteria | 47 |
| 6.3 Withdrawal criteria | 48 |
| 6.3.1 Potential drug-induced liver injury IMP discont | inuation criteria49 |
| 7 STUDY TREATMENTS | 50 |

| 7.1 | Description of investigational medicinal products | 50 |
|---|---|---|
| 7.2 | Treatments to be administered | 50 |
| 7.3 | Packaging | 51 |
| 7.4 | Labeling | 51 |
| 7.5 | Handling and storage requirements | 51 |
| 7.6 | Drug accountability | 51 |
| 7.7 | Procedures for monitoring subject compliance | 52 |
| 7.8 | Concomitant treatments and medications | 5210 |
| 7.8 | Permitted concomitant treatments (medications and therapies) | s 52 |
| 7.8 | Prohibited concomitant treatments (medications and therapies) | 53 |
| 7.8 | 8.3 Rescue medication | 53 |
| 7.9 | Blinding. | 53 |
| 7.10 | Randomization and numbering of subjects | 53 |
| 8 | STUDY PROCEDURES BY VISIT | 53 |
| 8.1 | Exploratory Cohort | 54 |
| 8.1 | 1.1 Screening Period | 54 |
| 8.1 | 1.2 Evaluation Period | 55 |
| 8.1 | 1.3 BRV Extension Period | 56 |
| | 8.1.3.1 Extension Period Visit 1 | 57 |
| | Rescue medication Blinding | 57 |
| | 8.1.3.3 Unscheduled Visit | 58 |
| | 8.1.3.4 Telephone Contact | 58 |
| 8.1 | 1.4 Safety Follow-Up Period | 58 |
| 8.2 | Confirmatory Cohorts | 59 |
| 8.2 | 2.1 Screening Period | 59 |
| | 8.2.1.1 Baseline Period | 59 |
| 8.2 | 2.2 Evaluation Period | |
| 8.2 | 2.3 BRV Extension Period | |
| | 8.2.3.1 Extension Period Visit 1 | |
| | 8.2.3.2 Extension Period Visit 2 | |
| | 8.2.3.3 Unscheduled Visit | |
| | 8.2.3.4 Telephone Contact | |
| 8.2<br>8.2 | Down-Titration Period | |
| 8.2 | 2.5 Safety Follow-Up Period | 65 |
| 9 | | |
| 9.1 | Pharmacokinetic sampling and handling | |
| 9.2 | Pharmacokinetic sample shipment | |
| 10 | ASSESSMENT OF EFFICACY | 67 |

| 10.1 | Asse | essment of the secondary efficacy variables (Confirmatory Cohort[s] only) | 67 |
|---|---|---|---|
| 10.2 | Asse | essment of other efficacy variables | 68 |
| 10.3 | Seiz | ure burden | 69 |
| 11 A | ASSES | SSMENT OF SAFETY | 69 |
| 11.1 | Adve | erse events | 69 |
| 11. | 1.1 | Definitions | 69 |
| | 11.1.1 | .1 Adverse event | 69 |
| | 11.1.1 | | 70 |
| | 11.1.1 | .3 Adverse events of special interest | 72 |
| 11. | 1.2 | Procedures for reporting and recording adverse events 2.1 Description of adverse events 2.2 Rule of repetition of an adverse event 2.3 Additional procedures for reporting serious adverse events | 72 |
| | 11.1.2 | 2.1 Description of adverse events | 75 |
| | 11.1.2 | 2.2 Rule of repetition of an adverse event | 75 |
| | 11.1.2 | 2.3 Additional procedures for reporting serious adverse events | 75 |
| | 11.1.2 | 2.4 Immediate reporting of adverse events | 76 |
| 11. | 1.3 | Follow-up of adverse events | 76 |
| 11. | 1.4 | Suspected transmission of an infectious agent | 76 |
| 11. | 1.5 | Overdose of investigational medicinal product | 76 |
| 11. | 1.6 | Safety signal detection | 77 |
| 11.2 | Labo | oratory measurements | 77 |
| 11. | 2.1 | 2.4 Immediate reporting of adverse events | <del>79</del> |
| | 11.2.1 | .1 Consultation with Medical Monitor and local hepatologist | 81 |
| | 11.2.1 | 1.2 Immediate action: determination of IMP discontinuation | 81 |
| | 11.2.1 | Testing: identification/exclusion of alternative etiology | 81 |
| | 11.2.1 | 1 | |
| 11.3 | Othe | er safety measurements. | |
| 11. | | Physical and neurological examinations | 83 |
| 11. | 3.2 | Medical history including Apgar score | |
| 11. | 3.3 | Vital signs | 84 |
| 11. | 3.4 | Biometric parameters | |
| 11. | 3.5 | N-PASS | 84 |
| | X | Video-EEG Parameters | |
| | 3.70 | HIE (Thompson score) | 85 |
| 110 | 3.8 | Withdrawal and rebound phenomena | |
| | 3.9 | Mechanical ventilation. | |
| 11. | 3.10 | Bayley Scales of Infant and Toddler Development, Third Edition | |
| 12 S | | Y MANAGEMENT AND ADMINISTRATION | |
| 12.1 | | erence to protocol | 86 |
| 12.2 | Mon | itoring | 86 |

| 12. | 2.1 Definition of source data | 86 |
|---|---|---|
| 12. | 2.2 Source data verification | 87 |
| 12.3 | Data handling | 87 |
| 12. | 3.1 Case Report form completion | 87 |
| 12. | 3.2 Database entry and reconciliation | 87 |
| 12. | 3.3 Subject Screening and Enrollment log/Subject Identification Code list | 87 |
| 12.4 | Termination of the study | |
| 12.5 | Archiving and data retention. | 88 |
| 12.6 | Audit and inspection | . 88 |
| 12.7 | Good Clinical Practice | 88 |
| 13 | STATISTICS | 89 |
| 13.1 | Definition of analysis sets | 89 |
| 13.2 | General statistical considerations | 89 |
| 13.3 | Pharmacokinetic variable analysis | 89 |
| 13. | 3.1 Exploratory Cohort | 89 |
| 13. | 3.2 Confirmatory Cohorts | 90 |
| 13.4 | Safety analyses | 90 |
| 13.5 | Planned efficacy analyses | 90 |
| 13. | | 90 |
| 13. | 5.2 Analysis of the other efficacy variables | 92 |
| 13.6 | Handling of protocol deviations. | 93 |
| 13.7 | Handling of dropouts or missing data | 93 |
| 13.8 | Planned PK data review and safety data monitoring | 93 |
| 13. | | 93 |
| 13. | 8.2 Confirmatory Cohorts | 93 |
| 13. | 8.3 DMC and stopping rules | 94 |
| 13.9 | Determination of sample size. | 94 |
| 14 I | ETHICS AND REGULATORY REQUIREMENTS | 94 |
| 14.1 | Informed consent | |
| 14.2 | Subject identification cards | 95 |
| 14.3 | Independent Ethics Committees | 95 |
| 14.4 | Subject privacy | 96 |
| - Y - | Protocol amendments | |
| $\sim$ | FINANCE, INSURANCE, AND PUBLICATION | |
| 16 I | REFERENCES | 97 |
| 17 | APPENDICES | |
| 17.1 | Protocol Amendment 1 | 100 |
| 17.2 | Protocol Amendment 2 | 122 |

## LIST OF ABBREVIATIONS

AΕ adverse event

**AED** antiepileptic drug ALP alkaline phosphatase

ALT alanine aminotransferase AST aspartate aminotransferase

**AUC** area under the curve

and any extensions of variations thereof.

Aication and any extensions Bayley-III® Bayley Scales of Infant and Toddler Development®, Third Edition

bid (bis in die) twice daily

**BRV** brivaracetam **BZD** benzodiazepine

**CDMS** clinical data management system

CI confidence interval

CGA corrected gestational age **CNS** central nervous system

Committee for Proprietary Medicinal Products **CPMP** 

contract research organization CRO

CTD Clinical Trials Directive

Data Monitoring Committee **DMC** 

**ECG** electrocardiogram

eCRF electronic Case Report form

**EEG** electroencephalogram

**EMA** European Medicines Agency

**ENS** electroencephalographic neonatal seizures

**EPV Extension Period Visit** 

**EudraCT** European Union Drug Regulating Authorities Clinical Trials

GA gestational age

**GCP** Good Clinical Practice

Good Manufacturing Practice

HIE hypoxic-ischemic encephalopathy

Investigator's Brochure **ICF** Informed Consent form

**ICH** International Council for Harmonisation

**IEC Independent Ethics Committee** 

| investigational medicinal product |
|---|
| interactive response technology |
| intravenous(ly) |
| lidocaine |
| levetiracetam |
| liver function test |
| midazolam |
| neonatal pain, agitation and sedation scale |
| phenobarbital |
| Paediatric Committee |
| potential drug-induced liver injury |
| phenytoin |
| postnatal age |
| pharmacokinetic |
| partial-onset seizure |
| Patient Safety |
| serious adverse event |
| midazolam neonatal pain, agitation and sedation scale phenobarbital Paediatric Committee potential drug-induced liver injury phenytoin postnatal age pharmacokinetic partial-onset seizure Patient Safety serious adverse event Statistical Analysis Plan standard of care Standard Operating Procedure Safety Set synaptic vesicle protein 2A |
| standard of care |
| Standard Operating Procedure |
| Safety Set |
| synaptic vesicle protein 2A |
| treatment-emergent adverse event |
| upper limit of normal |
| (multichannel) video-electroencephalography |
| Safety Set synaptic vesicle protein 2A treatment-emergent adverse event upper limit of normal (multichannel) video-electroencephalography |

#### 1 SUMMARY

N01349 is a Phase 2/3, multicenter, open-label, single-arm study to evaluate the pharmacokinetics (PK), seizure activity/efficacy (interpreted as "efficacy on seizure activity" and referred to as "efficacy" in the protocol), and safety of brivaracetam (BRV) in neonates with repeated electroencephalographic (EEG) seizures. Subjects will first receive antiepileptic drugs (AEDs) for the treatment of electroencephalographic neonatal seizures (ENS) (first-line, second-line, or subsequent treatment, which may have started prior to the subject's admission into the study site; dose and dosing regimen at the Investigator's discretion). If they do not have adequate seizure control after the treatment with AEDs, they may be enrolled into N01349.

As the patient population of neonates with ENS is limited, N01349 is designed with a 2-step approach to allow for confirmation (or adjustment) of BRV dosing based on results from the first step (Exploratory Cohort) and evaluation of BRV efficacy in the second step (Confirmatory Cohorts). This adaptive design allows for the determination of dose and the collection of PK, safety, and efficacy data, thereby potentially providing rapid access to alternative treatment in neonates.

For the Exploratory Cohort (first step), enrolled subjects will receive 1 or more of the following AEDs prior to or at the time of enrollment: phenobarbital (PB), midazolam (MDZ), phenytoin (PHT), levetiracetam (LEV), or lidocaine (LDC) for the treatment of ENS (first-line, second-line, or subsequent treatment; choice of treatment, dose, and dosing frequency is at the discretion of the Investigator) prior to receiving BRV. Subsequently, an initial low dose of BRV intravenous (iv) solution for injection will be administered. At the discretion of the Investigator, 3 additional iv BRV doses can be administered, up to a total of 4 iv BRV doses (0.5mg/kg twice daily [bid]), during the 48-hour Evaluation Period to determine the PK of BRV in neonates. This treatment represents the first use of BRV in neonates (0.5mg/kg bid), which is 4-fold less than the highest dosage of 4mg/kg/day that has been used previously in study N01263 (Section 2.2).

In BRV PK modeling studies CL0187 and N01331, PK profiles were extrapolated allometrically to the neonatal age group from the pediatric data collected in N01263 (age range of  $\geq 1$  month to < 16 years). A total of 600 samples from 96 subjects were used for this modeling. The results of this modeling suggest that a dosing regimen of 2mg/kg bid in pediatric subjects  $\geq 1$  month to < 16 years of age with a maximum of 100mg bid (for patients with a bodyweight of 50kg or more) would result in plasma concentration profiles similar to those attained in older children and adults who received therapeutic doses of BRV (up to 100mg bid). Since extrapolation of data from subjects  $\geq 1$  month to subjects  $\leq 2$  weeks may be imprecise due to variability in ontogeny in the metabolic and excretory functions in neonates, actual PK measurements conducted in the Exploratory Cohort of N01349 will be used to confirm the relationship between dose and plasma concentration in neonates.

For the Confirmatory Cohorts (second step with 3 consecutive cohorts planned), the efficacy of BRV will be evaluated. Subjects may have received 1 or more of the following AEDs prior to or at the time of enrollment: PB, MDZ, LEV (≤60mg/kg/day), PHT, or LDC. The iv dose and dosing frequency of BRV selected for the Confirmatory Cohorts will be determined by the evaluation of BRV plasma concentrations from the Exploratory Cohort, as well as by the PK modeling of N01263 data described above, to be within the range of plasma concentrations observed in children ≥1 month old who received BRV 4mg/kg/day. A dosage of BRV 4mg/kg/day for neonates is predicted to be approximately equivalent to the highest BRV dose


(200mg/day) approved as adjunctive therapy for partial-onset seizures (POS) in patients ≥16 years of age.

The recommendation to confirm or adjust the originally calculated BRV dose of the Confirmatory Cohorts of study N01349 will be given by the Data Monitoring Committee (DMC) after review of PK and safety data of the Exploratory Cohort. Based on the DMC meeting held on 05 Nov 2020, the BRV dose and frequency selected for the Confirmatory Cohorts is 1mg/kg bid (2mg/kg/day). Based on data from the Confirmatory Cohorts, the BRV dose may be further adjusted in a staggered approach as determined by the DMC.

The safety and PK of BRV will be evaluated in all 4 cohorts. At the end of the Evaluation Period, subjects from both the Exploratory and Confirmatory Cohorts may enter the BRV Extension Period.

The primary objective of this study is to evaluate the PK of BRV in neonates who have seizures that are not adequately controlled with previous AED treatment, and to identify the optimal BRV dose (Exploratory Cohort) for the treatment of subjects enrolled into the Confirmatory Cohorts of this study. Secondary objectives include the evaluation of the short-term safety and tolerability of BRV in neonates and the evaluation of the efficacy of BRV in severe and nonsevere seizure burden (defined as total minutes of ENS per hour) in neonates with seizures that are not adequately controlled with previous AED treatment.

This study will enroll at least 42 evaluable subjects (at least 6 subjects in the Exploratory Cohort, at least 36 subjects in the Confirmatory Cohorts, including at least 2 subjects undergoing hypothermia treatment in the Exploratory Cohort and each of the 3 Confirmatory Cohorts). At enrollment, subjects must be at least 34 weeks of corrected gestational age (CGA). In addition, term neonates up to 27 days of postnatal age (PNA) and preterm neonates up to 40 weeks of CGA and 27 days of PNA can be enrolled.

Subjects must have a confirmed diagnosis of ENS by multichannel video-electroencephalography (VEEG) of  $\geq 2$  minutes of cumulative ENS or  $\geq 3$  identifiable ENS prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite receiving AED treatment. The maximum study duration per subject is expected to be up to 75 days, which consists of a Screening Period, Baseline Period (Confirmatory Cohorts only), Evaluation Period, BRV Extension Period, Down-Titration Period (Confirmatory Cohorts only), and Safety Follow-Up Period. There is a possibility that in certain regions sites may not be ready to transition subjects to EP0156 at the time enrollment into N01266 will be closed. To avoid that enrollment into N01349 must pause from early Sep 2021 onwards, subjects will then be allowed to stay in N01349 for up to 90 days of PNA until rollover to the long-term study is possible. In this event, the maximum study duration for subjects who remain in the study for up to 90 days of PNA and do not enter the long-term study will then be up to 130 days (90 days of PNA, up to 7 days for the Down-Titration Period, and up to 33 days for the Safety Follow-Up Period). All subjects who participate in the BRV Extension Period must be offered entry into a long-term study, if they meet the eligibility criteria. Before entering the long-term study, subjects must be on oral BRV.

The PK variables are the plasma concentrations of BRV, the area under the curve (AUC), volume of distribution, and clearance of BRV in neonates. Further, PK assessments will include plasma concentrations of concomitant PB and/or PHT if administered.

The safety variables are adverse events (AEs) as reported by the Investigator, withdrawal and rebound phenomena, and mechanical ventilation over the Evaluation Period of the Exploratory The efficacy of BRV will be analyzed for the Confirmatory Cohorts based on the following variables:

The proportion of responders to BRV treatment from Baseline to 3 hours dose. A BRV responder is defined as a subject who act in minutes per hour), without need for neasured during the B. Cohort and the Confirmatory Cohorts. In addition, safety variables also include the change from

2-hour period starting 1 hour after the start of initial BRV treatment. Reduction in seizure burden is defined as at least 80% reduction in nonsevere seizure burden (nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in all 30-minute timespans) or at least 50% reduction in severe seizure burden (severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan). Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to  $\leq$ 30 minutes,  $\geq$ 30 to  $\leq$ 60 minutes,  $\geq$ 60 to  $\leq$ 90 minutes, and  $\geq$ 90 to <120 minutes.

Secondary efficacy variables will also include the proportion of subjects with at least 80% reduction in nonsevere seizure burden from Baseline to 3 hours after the initial BRV treatment, the proportion of subjects with at least 50% reduction in severe seizure burden from Baseline to 3 hours after the initial BRV treatment, the absolute and percentage reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period, the proportion of BRV responders at the end of the 96-hour Evaluation Period, the proportion of subjects who are seizure-free (100% reduction in seizure burden from Baseline) at 24 hours following the start of initial BRV treatment, categorized by subjects with nonsevere or severe seizure burden at Baseline, the time to reduction in seizure burden for BRV responders (defined as the first timepoint when BRV responder criteria are met), seizure freedom at the end of the Down-Titration Period, rate of at least 50% reduction in ENS frequency per hour from Baseline to the end of the 96-hour Evaluation Period, the proportion of subjects who are seizure-free by time interval (at 3 hours, at 3 hour intervals thereafter through 24 hours, and every 12 hours to 24 hours following the start of the initial BRV treatment), and the absolute and percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline

burden at the defined evaluation periods, the categorized percentage reduction from Baseline to the end of the 96-hour Evaluation Period in seizure burden, the proportion of PDV time interval at the defined evaluation period. the end of the 96-hour Evaluation Period in seizure burden, the proportion of BRV responders by BRV to another AED during the 96-hour Evaluation Period, and the proportion of responders to other treatment during the 96-hour Evaluation Period.

#### 2 INTRODUCTION

## 2.1 Epidemiology and treatment of targeted disease

Seizures occur more often during the neonatal period than at any other time during life (Volpe, 2008). The most common cause of neonatal seizures is HIE as a result of perinatal asphyxia (van Rooij et al, 2013a). A population-based study suggested that 42% of neonatal seizures were observed following HIE (van Rooij et al, 2013a). Other causes include intracranial hemorrhage and stroke, infections of the central nervous system (CNS), congenital malformations, inborn errors of metabolism, transient metabolic disturbances, maternal drug abuse, or rare neonatal epilepsy syndromes (benign familial neonatal-infantile seizures or fifth-day seizures) (Volpe, 2008; Ronen et al, 1999).

Clinical recognition of seizures in newborns is not always simple due to a highly variable clinical expression (Volpe, 2008; Mizrahi and Kellaway, 1987). As demonstrated by prolonged VEEG recordings, especially following AED treatments, ENS patterns are not always accompanied by clinical signs (Scher et al, 2003; Boylan et al, 2002; Clancy et al, 1988; Mizrahi and Kellaway, 1987).

First-generation AEDs, such as PB and PHT, remain the drugs of first (and second) choice because of extensive clinical experience, despite their limited clinical effectiveness and potential neurotoxicity (van Rooij et al, 2013b).

In addition to MDZ, other benzodiazepines (BZDs; eg, lorazepam and clonazepam) are used for the treatment of neonatal seizures, often in PB-refractory cases. As one of the most lipophilic BZDs, MDZ readily crosses the blood-brain barrier and provides the advantage of very rapid onset of action. The formation of pharmacologically active (glucuronidated) metabolites of MDZ is considered a disadvantage of MDZ use since drug-drug interactions or renal impairment could cause an undesired accumulation of these metabolites (van Rooij et al, 2013a).

Current treatments for neonatal seizure include PB, PHT, LEV, LDC, and MDZ (Slaughter et al, 2013).

## 2.2 Background information regarding product

Brivaracetam ((2S)-2-[(4R),2-oxo-4-propyltetrahydro-1H-pyrrol-1-yl] butanamide) displays a high and selective affinity for the synaptic vesicle protein 2A (SV2A) in the brain. Binding to SV2A is believed to be the primary mechanism for BRV anticonvulsant activity. Between 2016 and 2018, marketing authorization for the use of oral and iv BRV as adjunctive treatment for POS was granted in the EU, US, Russia, Turkey, Mexico, Australia, India, Argentina, Israel, United Arab Emirates, Qatar, Hong Kong, and Korea (film coated tablet, oral solution) for patients 16 years of age and older with epilepsy and in Switzerland and Canada for patients 18 years of age and older with epilepsy. Brivaracetam is approved in the US as monotherapy, based on extrapolation, for the treatment of POS in patients with epilepsy aged 16 years and older. An application for the extension of indication to the pediatric population from 4 years of age in the EU (adjunctive) and the US (adjunctive and monotherapy) based on the concept of extrapolation of efficacy data from the adult population was approved in 2018. Of note, in the US, BRV injection is indicated for the treatment of POS only in adult patients (16 years of age and older).


Brivaracetam is weakly bound ( $\leq 20\%$ ) to plasma proteins. The volume of distribution is 0.5L/kg, a value close to that of the total body water.

Brivaracetam is rapidly and evenly distributed in most tissues and penetrates rapidly into the brain. The main metabolic pathway of BRV is by hydrolysis of the acetamide group to the corresponding carboxylic acid, ucb-42145, while a second pathway is the  $\omega$ 1-hydroxylation into ucb-100406-1 mediated by cytochrome P450 (CYP)2C19. The combination of these 2 pathways results in the terminal metabolite (hydroxyacid), ucb-107092-1. These metabolites are not pharmacologically active. Brivaracetam is eliminated primarily by metabolism and by excretion in the urine. More than 95% of the dose, including metabolites, is excreted in the urine within 72 hours after dosing in adults. The terminal half-life is approximately 9 hours.

The first BRV pediatric study was N01263, which is described as follows:

N01263 was a completed open-label, multicenter, fixed 3-step up-titration, adjunctive therapy study of the PK, safety, and efficacy of BRV in subjects ≥1 month old to <16 years of age with epilepsy. The study enrolled 100 subjects with either focal or generalized epilepsy. Doses of BRV (oral solution) were adjusted by body weight and did not exceed a maximum of 50mg/day, 100mg/day, and 200mg/day for each titration step.

A total of 100 subjects were enrolled in N01263: 99 subjects received the study drug and were included in the Safety Set (SS). Results from N01263 indicate that BRV was generally well-tolerated and that the safety profile in pediatric subjects was consistent with the known safety profile in adult subjects. Six subjects discontinued the study due to treatment-emergent adverse events (TEAEs), including 1 serious adverse event (SAE) that was moderate in intensity. All severe TEAEs and 11 out of 12 treatment-emergent SAEs were considered to be not related to study drug by the Investigator. No deaths were reported. The TEAE profile in pediatric subjects in this study was consistent with the known BRV safety profile in adults with a low incidence of dizziness as the main difference. There was no dose dependency observed in the overall incidence of TEAEs. In general, there were no clinically meaningful changes in laboratory parameters, vital signs, or electrocardiograms (ECGs).

Pharmacokinetic analyses performed for N01263 demonstrated that BRV plasma concentrations increased with increasing age and increased proportionally to the dose, which was indicated by the approximate doubling of trough BRV plasma concentration with every doubling of the BRV dose. Trough plasma concentration in the  $\geq 1$  month to  $\leq 2$  years age group was approximately 30% to 45% lower than in adolescents.

For the 97 subjects included in the efficacy analysis, 47 subjects (58.8%) had a -25% to <25% reduction in the number of seizure days from Baseline to the end of the Evaluation Period, and 26 subjects (32.5% of all subjects) had a ≥25% reduction. Similar observations were made overall across age groups and by seizure category. Six subjects (7.5% of all subjects) experienced a 100% reduction in the number of seizure days from Baseline to the end of the Evaluation Period, and 7 subjects (8.8% of all subjects) experienced a <-25% reduction.

Overall, 14 subjects (14.4%) experienced seizure freedom over the Evaluation Period, based on the Data Record Card data. The number of subjects with seizure freedom was highest in the ≥2 years to <12 years age group (9 subjects [18.0%]), with a similar number of subjects in the ≥1 month to <2 years and ≥12 years to <16 years age groups (3 subjects [10.0%] and 2 subjects

[11.8%], respectively). The overall mean proportion of seizure-free days was 0.5 days (±0.4 days) and was similar regardless of age group or seizure type (range: 0.3 days to 0.7 days).

N01266, an ongoing, open-label, multicenter study, was designed as a long-term follow-up study for subjects who had enrolled in N01263 and the other studies conducted with BRV in the pediatric population from birth to 18 years of age. The objectives of this study include evaluation of the long-term safety and efficacy of bid administration of BRV oral solution and tablets in pediatric subjects with epilepsy; the maximum allowable BRV dosage is 5mg/kg/day, not to exceed 200mg/day in subjects with body weights >40kg.

Based on the results of population PK modeling studies CL00187 and N01331, it was concluded that a dosing regimen of 2.0mg/kg bid in pediatric subjects ≥1 month to <16 years of age with a maximum of 100mg bid should result in plasma concentration profiles similar to those attained in older children and adults who receive therapeutic doses of BRV (up to 200mg per day). Extrapolation of the model to neonates suggested that doses of 2mg/kg to 3mg/kg bid might be required to achieve exposure similar to adults receiving the maximum dose of 200mg bid. Since extrapolation of data from subjects more than 1 month old to subjects 2 weeks of age or younger may be imprecise due to variability in ontogeny in the metabolic and excretory functions in neonates, actual PK measurements (ie, those conducted in the Exploratory Cohort of N01349) are needed to confirm the relationship between dose and plasma concentration in neonates.

Additional information about BRV, including the current information pertaining to the pediatric development program, is provided in the Investigator's Brochure (IB).

## 2.3 Rationale for the study

Neonatal seizures are described in the International League Against Epilepsy report as "subtle because the manifestations are often overlooked." Most neonatal seizures do not comply with the usual term epilepsy (enduring predisposition to seizures) because they are symptomatic (provoked, reactive) seizures most commonly caused by HIE, cerebral infarction, or infection.

Due to growing evidence that neonatal seizures contribute to an adverse neurodevelopmental outcome, physicians are increasingly focused on the diagnosis and treatment of this condition (Glass et al, 2012). The current available data from randomized controlled studies to support the choice of AEDs for this indication are limited, and there are currently no definite recommendations on the most suitable treatment option to use (Pressler and Mangum, 2013; van Rooij et al, 2013a). Thus, there is a need to investigate which AEDs should be used to treat neonatal seizures and their most appropriate dosages (Pressler and Mangum, 2013; Glass et al, 2012). Furthermore, although newer AEDs are efficacious for the treatment of seizures in adults and older children, limited progress has been made in the treatment of neonatal seizures (Pressler et al, 2015; Tulloch et al 2012). Therefore, clinical studies to assess the efficacy and safety of new treatment options in neonates are warranted.

Thus far, BRV is well-tolerated orally up to 200mg/day in adult subjects with epilepsy and in children 1 month old to 16 years of age receiving up to 4mg/kg/day. Intravenously administered BRV is bioequivalent to the same dosage given orally in healthy adults when given as a bolus or as a 15-minute infusion. Results have shown that a single iv BRV dose of up to 150mg as a 15-minute infusion or as a bolus dose is well-tolerated in adults. Based on these results, the iv route of administration and the proposed dosages to be used in N01349 are justified.

N01349 represents the first study of BRV in neonatal subjects, and will evaluate the PK, efficacy, and safety of BRV in neonates (up to 27 days of PNA and preterm neonates up to 40 weeks of CGA and 27 days of PNA).

#### 3 STUDY OBJECTIVES

## 3.1 Primary objective

The primary objective is to evaluate the PK of BRV in neonates who have seizures that are not adequately controlled with previous AED treatment, and to identify the optimal BRV dose (Exploratory Cohort) for the treatment of subjects enrolled into the Confirmatory Cohorts of this study.

## 3.2 Secondary objectives

The secondary objectives are:

- To evaluate the efficacy of BRV in severe and nonsevere seizure burden (defined as total minutes of ENS per hour) in neonates with seizures that are not adequately controlled with previous AED treatment
- To evaluate the short-term safety and tolerability of BRV in neonates

#### 4 STUDY VARIABLES

## 4.1 PK variables (Exploratory and Confirmatory Cohorts)

### 4.1.1 Primary PK variable

The primary PK variable is as follows:

• Plasma concentrations of BRV following first dose on Day 1

#### 4.1.2 Other PK variables

- Plasma concentrations of BRV on other occasions
- Plasma concentrations of BRV metabolites ucb-42145 (acid), ucb-100406-1 (hydroxy), and ucb-107092-1 (hydroxyacid)
- AUC, volume of distribution, and clearance of BRV
- Plasma concentrations of concomitant AEDs if administered

  Plasma concentrations of concomitant AEDs if administered

  This document cannot be used.

## 4.2 Efficacy variables (Confirmatory Cohorts only)

The variables for the evaluation of BRV efficacy are described in Section 4.2.1 (Secondary efficacy variables) and Section 4.2.2 (Other efficacy variables).

## 4.2.1 Secondary efficacy variables

The main secondary efficacy variable is as follows:

Proportion of responders to BRV treatment from Baseline to 3 hours after the initial BRV dose

A BRV responder is defined as a subject who achieves the following reduction in seizure burden (ENS in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment:

At least 80% reduction in nonsevere seizure burden
 (Nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in all 30-minute timespans)

OR

At least 50% reduction in severe seizure burden

(Severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan). Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to  $\leq$ 30 minutes, >30 to  $\leq$ 60 minutes, >60 to  $\leq$ 90 minutes, and >90 to  $\leq$ 120 minutes.

For this study, an ENS is defined as an EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug.

In addition, the secondary efficacy variables will include:

- Proportion of subjects with at least 80% reduction in nonsevere seizure burden from Baseline to 3 hours after the initial BRV treatment
- Proportion of subjects with at least 50% reduction in severe seizure burden from Baseline to 3 hours after the initial BRV treatment
- Absolute reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period
- Percent reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period
- Proportion of BRV responders at the end of the 96-hour Evaluation Period
- Proportion of subjects who are seizure-free (100% reduction in seizure burden from Baseline) at 24 hours following the start of initial BRV treatment, categorized by subjects with nonsevere or severe seizure burden at Baseline



- Time to reduction in seizure burden for BRV responders (defined as the first timepoint when BRV responder criteria are met)

- rroportion of subjects who are seizure-free by time interval at 3 hours, at 3-hour intervals thereafter through 24 hours, and every 12 hours to 24 hours thereafter up until the end of the 96-hour Evaluation Period following the start of the initial BRV treatment

  Absolute difference in clinical seizures at the end of the 24 the Baseline for neonates with motor seizure.
- Percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion

The use of rescue medication will affect the analysis of the main secondary efficacy variable(see Section 13.5.1). The factors affecting the definition of BRV responders for the analysis of the secondary efficacy variables are described in Section 10.1.

#### 4.2.2 Other efficacy variables

Other efficacy variables will include:

- Absolute reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
- Percent reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
- Categorized percentage reduction from Baseline to the end of the 96-hour Evaluation Period in seizure burden (<-25% [worsening], -25% to <25% [no change], 25% to <50%, 50% to <80%, and  $\ge 80\%$ )
- Proportion of BRV responders by time interval at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
- Proportion of subjects who switch over from BRV to another AED during the 96-hour **Evaluation Period**
- Proportion of responders to other treatment during the 96-hour Evaluation Period (including at the end of the 96-hour Evaluation Period, and by time intervals: 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment)

(A responder to other treatment is defined as at least 80% reduction in nonsevere seizure burden from start of other treatment to end of other treatment or at least 50% reduction in severe seizure burden from the initiation of other treatment to end of other treatment during the 96-hour Evaluation Period).

## 4.3 Safety variables (Exploratory and Confirmatory Cohorts)

## 4.3.1 Secondary safety variable

The secondary safety variable is as follows:

• AEs as reported by the Investigator

## 4.3.2 Other safety variables

- Change from Baseline in vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Change from Baseline in safety laboratory tests to the end of the Evaluation Period
- Change from Baseline in heart rate at 3 hours, 24 hours, 48 hours, and 96 hours after the start of initial BRV treatment
- Change from Baseline in physical and neurological examination 24 hours, 48 hours, 72 hours, and 96 hours after the start of initial BRV treatment (Sarnat scale; for subjects with HIE only)
- Change from Baseline in EEG-parameters (assessment of sedation) to the end of the Evaluation Period (Confirmatory Cohorts only)
- Change from Baseline in severity of HIE to the end of the Evaluation Period (Thompson score; for subjects with HIE only)
- Change from Baseline in N-PASS score (neonatal pain and agitation measures) to the end of the Evaluation Period
- Change from Baseline in biometric parameters at the Safety Follow-Up Visit: length, body weight, and head circumference (head circumference Baseline measurement should be taken within 7 days prior to drug administration, or at birth for subjects ≤7 days old)
- Withdrawal and rebound phenomena
- Mechanical ventilation:
  - Number and percentage of subjects requiring mechanical ventilation during the Evaluation Period
  - Duration of mechanical ventilation during the Evaluation Period

Neurodevelopmental tests validated for age and language will be done after 1 year for subjects who enter the long-term follow-up study in countries where a validated translation of the Bayley Scales of Infant and Toddler Development<sup>®</sup>, Third Edition (Bayley-III<sup>®</sup>) score is available.

#### 5 STUDY DESIGN

## 5.1 Study description

N01349 is a Phase 2/3, multicenter, open-label, single-arm study to evaluate the PK, efficacy, and safety of BRV in neonates with repeated EEG seizures.

N01349 consists of a 2-step design and includes a descriptive comparison with a historical control group (matched in age and condition) from literature treated with AEDs per SOC and diagnostic methods.

For the Exploratory Cohort (first step), enrolled subjects will have received 1 or more of following AEDs prior to or at the time of enrollment: PB, MDZ, PHT, LEV, or LDC for the treatment of ENS (first-line, second-line, or subsequent treatment; choice of treatment, dose, and dosing frequency are at the discretion of the Investigator) prior to receiving BRV. Subsequently, a low dose of BRV iv solution for injection will be administered. At the discretion of the Investigator, 3 additional iv BRV doses, up to a total of 4 iv BRV doses (0.5mg/kg bid), can be administered during the 48-hour Evaluation Period. This treatment, which is the first use of BRV in neonates, is 4-fold less than the highest dose of 4mg/kg/day dosage (2mg/kg bid) that has been used previously in infants ≥1 month old.

For the Confirmatory Cohorts (second step), 3 consecutive cohorts are planned, and the efficacy of BRV will be evaluated. Subjects may receive 1 or more of the following AEDs prior to or at the time of enrollment: PB, MDZ, PHT, LEV (≤60mg/kg.day), PHT, or LDC. The iv dose of BRV selected for the Confirmatory Cohorts will be determined by the evaluation of BRV plasma concentrations from the Exploratory Cohort, as well as by previous PK modeling of N01263 data, to be within the range of plasma concentrations observed in children ≥1 month old who received 4mg/kg/day. A dosage of BRV 4mg/kg/day for neonates is predicted to be approximately equivalent to the highest BRV dosage (200mg/day) that has been studied in the adult Phase 3 program (eg, N01358 and N01258).

The PK and safety of BRV will be evaluated in all cohorts. The recommendation to confirm or adjust the originally calculated BRV dose of the Confirmatory Cohorts of study N01349 will be given by the DMC after review of PK and safety data of the Exploratory Cohort. Based on the DMC meeting held on 05 Nov 2020, the BRV dose and frequency selected for the Confirmatory Cohorts is 1mg/kg bid (2mg/kg/day). Based on data from the Confirmatory Cohorts, the BRV dose may be further adjusted in a staggered approach as determined by the DMC.

At the end of the Evaluation Period, subjects from both the Exploratory and Confirmatory Cohorts may enter the BRV Extension Period.

All subjects who participate in the BRV Extension Period must be offered entry into a long-term study, if they meet the eligibility criteria. Before entering the long-term study, subjects must be on oral BRV.

Blood samples for routine assay of hematology, biochemistry, liver enzymes, and endocrinology will be collected in line with Section 13.2 of the "Ethical Considerations for Clinical Trials on Medicinal Products Conducted with the Paediatric Population" (European Union Commission ad hoc group, 2008), and according to the schedule of study assessments in Table 5–1 (Exploratory Cohort) and Table 5–2 (Confirmatory Cohorts). The local laboratories will perform the routine analysis of blood samples. For Screening and determination of eligibility, use of laboratory data


acquired prior to Screening per standard of care inside or outside the study site within 36 hours prior to the start of the Evaluation Period is allowed.

Interpretation of VEEGs recorded for the Confirmatory Cohorts will be done by local readers but may be supported by the blinded central reader, as needed. Start and stop of BRV treatment and the administration of rescue medication or alternative AEDs will be digitally marked as treatment events on VEEGs. The VEEG recordings will subsequently be evaluated by a blinded, independent central reader at the end of the study. The independent central reader will be blinded from site-specific information and the subject's medical history.

Subjects assigned to the Confirmatory Cohorts will be evaluated with VEEG monitoring at least during the Baseline, Evaluation, and Down-Titration Period. Interruption of the VEEG is allowed up to 30 minutes per day. Depending on medical needs related to SOC (eg, MRIs to be performed), interruptions longer than this are acceptable. However, every effort should be made to avoid VEEG interruption of the Baseline VEEG and during the first 3 hours after the start of the initial BRV administration. The video portion of the VEEG monitoring will assist Investigators in accurately diagnosing ENS and distinguishing artifacts from epileptiform discharges/seizures.

For subjects undergoing therapeutic hypothermia treatment, the target low body temperature achieved and age since birth when cooling began will be recorded. Rewarming of subjects will be documented in the same way.

If appropriate (in the event of screening failures), re-screening will be allowed for the study. Re-screening for screen-failed subjects will be allowed with prior consultation of the Medical Monitor whenever feasible. Subjects can be re-screened only once. Once a subject has received at least one dose of BRV or has left the study because a "must withdrawal" criterion is met, re-screening will no longer be possible.

A continuous consent process will be followed. Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the Informed Consent form (ICF) after the occurrence of seizures has been confirmed by VEEG; subjects will then be considered to be enrolled. During the course of the study, parent(s) or legal representative(s) will be updated about the care of their neonate, and continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s). Parent(s) or legal representative(s) will not be asked to re-sign and re-date the ICF, but they will be informed that they can withdraw their neonate from the study at any time and that this decision will not affect the care of their neonate. Continuous consent will be documented in the subjects' medical charts and electronic Case Report form (eCRF).

A DMC will be in place for the duration of this study. The DMC will meet after completion of the 6 subjects in the Exploratory Cohort and after completion of each of the 3 Confirmatory The schedules of assessments during the Screen and Confirmatory C. Cohorts (12 subjects each). Although it was planned that the DMC will meet at no longer than 6-month intervals between meetings, due to the low enrollment rate observed, the intervals

The schedules of assessments during the Screening and Evaluation Periods for the Exploratory and Confirmatory Cohorts are presented in Table 5–1 and Table 5–2, respectively. The schedule of assessments during the BRV Extension, Down-Titration (Confirmatory Cohorts only), and

Safety Follow-Up Periods for both the Exploratory and Confirmatory Cohorts are presented in Table 5-3.

Details of the study periods for the Exploratory and Confirmatory Cohorts are described in Section 5.1.1 and Section 5.1.2, respectively.

#### **5.1.1** Exploratory Cohort

For the Exploratory Cohort, at least 6 subjects who do not have adequate seizure control after they received 1 or more of the following AEDs: PB, MDZ, PHT, LEV, or LDC prior to or at the time of enrollment for the treatment of ENS (first-line, second-line, or subsequent treatment, which may have started prior to the subject's admission into the study site; choice of treatment, dose, and dosing regimen at the Investigator's discretion) will be enrolled. The AED treatment per SOC can be continued when BRV dosing is initiated. Alternatively, another AED treatment (choice of treatment, dose, and dosing regimen at the Investigator's discretion) must be initiated and continue in parallel with BRV treatment.

At any time after AED treatment per SOC for the treatment of ENS (first-line, second-line, or subsequent treatment) was initiated, an initial low dose of BRV (0.5mg/kg [bid]) will be administered at the Investigator's discretion. After the Exploratory Cohort completes the study, a PK and safety data review will be performed by the DMC. During the review of data from the Exploratory Cohort, the enrollment of subjects will be on hold.

At least 2 subjects undergoing hypothermia treatment will be included. Subjects in the Exploratory Cohort might be replaced due to lack of data, as deemed necessary following the review of PK and safety data by the DMC.

The study periods for the Exploratory Cohort are as follows:

Screening Period: from signing and dating of the written ICF up to initiation of the first BRV dose.

The Screening Period starts up to 36 hours prior to the first administration of BRV. Phenobarbital, MDZ, PHT, LEV, or LDC may have been administered prior to the subject's enrollment into the study and/or at a location other than the study site.

Subjects will enter the Evaluation Period and start BRV treatment as soon as the occurrence of ENS per inclusion criterion 2a is confirmed by the Investigator based on local EEG. If preferred by the Investigator, the central VEEG reader can be consulted to confirm the required ENS.

• Evaluation Period (48 hours): The first BRV infusion marks the starting point of the Evaluation Period. At any time after AED treatment per SOC for the treatment of ENS (first-line, second-line, or subsequent treatment) was initiated, a low dose of BRV (0.5mg/kg) will be administered as an approximately 15-minute iv infusion; additional 3 doses of BRV(0.5mg/kg) can be administered every 12 hours for 48 hours (at the discretion of the Investigator). The AED treatment per SOC can be continued when BRV dosing is initiated. Otherwise, another AED treatment (choice of treatment, dose, and dosing regimen at the Investigator's discretion) must be initiated and continue in parallel with BRV treatment.

Following the first BRV infusion, 3 to 6 PK blood microsamples (60µL/sample) will be collected during the 48-hour Evaluation Period from each subject for the determination of

plasma concentrations of BRV and its metabolites, as described in Table 5-4. The first set of 3 PK samples will be collected on the first day within specific timeframes (Table 5–4), with the second set of 3 PK samples to be collected within the same timeframes on the second day DRV infusion. The AED PK sample should be collected 3 hours after the start of the initial BRV administration. The number of subjects in the Exploratory Cohort may be increased, if deemed necessary following the analysis of PK data.

At the end of the Evaluation Period, subjects who benefit for BRV Extension Period in accordance the BRV Extension Period in accordance.

the BRV Extension Period will proceed immediately to the Safety Follow-Up Period (a visit will occur 30±3 days after the final BRV administration).

BRV Extension Period (up to 28 days of postnatal age [+7 days]): Subjects can proceed to the BRV Extension Period if they benefit from BRV treatment during the Evaluation Period, in accordance with the Investigator's opinion. All subjects who participate in the BRV Extension Period must be offered entry into the long-term study of they meet the eligibility criteria. Subjects will participate in the BRV Extension Period until they reach a stable condition that will allow them to enter the long-term study. The anticipated duration of the BRV Extension Period per subject is up to 28 days of postnatal age (+7 days). Subjects must switch to BRV oral solution before entering the long-term study. The timing of the switch from iv to oral solution will be at the discretion of the Investigator; subjects who are not able to be dosed with BRV oral solution when they reach 28 days of postnatal age may continue in the BRV Extension Period for an additional 7 days; subjects who are not able to be switched to BRV oral solution by the end of the additional 7 days of the BRV Extension Period will not be eligible for enrollment in the long-term study.

During the BRV Extension Period, subjects may continue receiving the same BRV dose administered at the end of the Evaluation Period (ie, BRV 0.5mg/kg bid); the BRV dose should not be increased but may be decreased at the discretion of the Investigator.

Safety Follow-Up Period: Subjects will proceed to the Safety Follow-Up Period if they do not enter the BRV Extension Period. The visit will occur 30±3 days after the final administration of BRV.

#### 5.1.2 **Confirmatory Cohorts**

For the Confirmatory Cohorts, enrollment will only start after the dosing of BRV is determined based on the PK findings of the Exploratory Cohort and an existing PK model from N01263. A total of at least 36 subjects without adequate seizure control after receiving one or more of the stable dose for at least 1 hour at the time the form. PB, MDZ, PHT, LEV (≤60mg/kg/day), or will enter the Confirmatory Cohorts. The AED treatment can be continued if the subject to the stable dose for at least 1 hour at the time the form.

Three consecutive Confirmatory Cohorts (n=12 each) are planned; each cohort must have at least 2 subjects undergoing hypothermia treatment. A PK and safety data review will be performed by

the DMC after completion of each of the 3 Confirmatory Cohorts. Based on the DMC meeting held on 05 Nov 2020, the BRV dose and frequency selected for the Confirmatory Cohorts is 1mg/kg bid (2mg/kg/day). Based on data from the Confirmatory Cohorts, the BRV dose may Screening Period: from signing and dating of the written ICF up to initiation of the first BRV dose.

The Screening Period starts up to 36 hours prior to the first Phenobarbital, MDZ, PHT, LEV (CCC) prior to the goal.

- site.
- Baseline Period (included in the Screening Period):
  - o For subjects with intermittent ENS: at least 1 hour prior to entering the Evaluation Period
  - For subjects in **status epilepticus:** up to 30 minutes prior to entering the Evaluation Period. At least 15 minutes of continuous seizures, or 50% of cumulative seizure activity during a 30-minute interval are to be confirmed on EEG before the administration of BRV can start.

As soon as subjects are considered to be in status epilepticus, steps required for the preparation of the initial BRV infusion can be initiated (eg, assignment of BRV kits through interactive response technology [IRT] and the dilution of BRV solution for iv infusion), even if the required EEG recording is not completed by that time.

Status epilepticus in neonates for the purpose of this study is defined as follows:

15 minutes of continuous or cumulative electrographic or electroclinical seizure within 30 minutes

The occurrence of ENS during the Baseline Period must be confirmed either by the local or central VEEG reader prior to BRV administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements (eg, ability for immediate cloud-based central review) can be used as part of the Baseline assessment VEEG.

Evaluation Period (96 hours): The first administration of BRV marks the starting point of the Evaluation Period. Subjects in the Confirmatory Cohorts will receive iv BRV 1mg/kg bid (2mg/kg/day), as recommended by the DMC on 05 Nov 2020 based on the results of the PK analysis of the Exploratory Cohort as well an existing PK model from N01263. The DMC will continue to monitor the PK and safety of the subjects and dosing may be adjusted as new data are available. If subjects do not benefit from BRV treatment after 96 hours of BRV administration, BRV administration will be stopped and replaced by another AED.

Following the first BRV infusion, 6 PK blood microsamples (60µL/sample) will be collected during the 96-hour Evaluation Period for each subject for the determination of plasma concentrations of BRV and its metabolites, as described in Table 5–5. Blood for PK samples should be drawn from a line different to that of the BRV infusion.

The AED PK sample should be collected 3 hours after the start of the initial BRV administration. In addition, opportunistic blood samples for the PK analysis may be used at the Investigator's discretion at any time during the Evaluation Period (see Section 9.1).

At the end of the Evaluation Period, subjects who benefit from BRV treatment may enter the BRV Extension Period in accordance with the Investigator's opinion. Subjects not entering the BRV Extension Period will proceed to the Down-Titration Period.

• BRV Extension Period (28 days [up to 90 days] of PNA): Subjects can proceed to the BRV Extension Period if they benefit from BRV treatment during the Evaluation Period, in accordance with the Investigator's opinion. All subjects who participate in the BRV Extension Period must be offered entry into the long-term study, if they meet the eligibility criteria. Subjects will participate in the BRV Extension Period until they reach a stable condition that will allow them to enter the long-term study, if epilepsy is confirmed.

The anticipated duration of the BRV Extension Period per subject is up to 28 (+7) days of PNA. Subjects who are not able to be dosed with BRV oral solution at a PNA of 28 days may continue in the BRV Extension Period for an additional 7 days; subjects who are not able to be switched to BRV oral solution by the end of the additional 7 days of the BRV Extension Period will not be eligible for enrollment in the long-term study.

In the event that a long-term study is temporarily not available, subjects are allowed to remain in the BRV Extension Period until they reach a PNA of up to 90 days. For those subjects, the assessments planned for Unscheduled Visits (see Section 8.1.3.3) will be conducted in intervals of approximately 30 days during the prolonged Extension Period. The treatment with BRV will be managed through IVRS. Before subjects can roll-over to the long-term study, they must have switched to BRV oral solution.

- Subjects must switch to BRV oral solution before entering the long-term study. The timepoint of the switch from iv to oral solution will be at the discretion of the Investigator.
  - During the BRV Extension Period, subjects may continue receiving the same BRV dose administered at the end of the Evaluation Period; the BRV dose should not be increased, but may be decreased at the discretion of the Investigator.
  - Down-Titration Period (up to 1 week): A Down-Titration Period of up to 1 week is recommended for subjects in the Confirmatory Cohorts who discontinue BRV treatment prior to completion of the Evaluation Period, who do not proceed to the BRV Extension Period, or start the BRV Extension Period but do not enter the long-term study. The Down-Titration steps and duration may be adjusted at the Investigator's discretion.
- Safety Follow-Up Period: Subjects will proceed to the Safety Follow-Up Period once they complete the Down-Titration Period. The visit will occur 30±3 days after the final administration of BRV.

Rescue medication should be given if the following occurs:

- There is no improvement in seizure burden within the first 3 hours after administration of BRV.
- Seizure burden is unacceptable to the Investigator, in which case rescue medication can be given earlier at any time, but ideally not in the first 3 hours after the initial administration of BRV.

Subjects in the Confirmatory Cohorts are allowed to switch over from BRV to another AED (eg, MDZ or PHT), if needed. Subjects discontinuing BRV treatment during the Evaluation Period should start the Down-Titration Period while completing the Evaluation Period in parallel for the full 96 hours. In this case, subjects will complete all study assessments, except the collection of blood microsamples for the determination of BRV plasma concentrations. Ideally, changing or adding a new treatment should not occur during the first 3 hours after the initial administration of BRV. Subjects who are switched from BRV to another AED will not be eligible to participate either in the BRV Extension Period or the long-term study.

## 5.1.3 Study duration per subject

The maximum study duration per subject is expected to be up to 75 days (Screening Period [including Baseline Period (Confirmatory Cohorts only)], Evaluation Period, BRV Extension Period, Down-Titration Period [Confirmatory Cohorts only], and Safety Follow-Up Period). In the event that a long-term study is not available at the time of a subject's planned transition, the maximum study duration for subjects who remain in the study for up to 90 days of PNA and do not enter the long-term study will then be up to 130 days (90 days of PNA, up to 1 week for the Down-Titration Period, and up to 33 days for the Safety Follow-Up Period). The individual study duration will be shorter depending on the type of cohort to which subjects will be assigned, the age at enrollment, and the decision to enter the BRV Extension Period.

The maximum BRV exposure per subject is expected to be up to 42 days, which comprises up to 4 days during the Evaluation Period (depending on type of cohort), up to 28 (+7) days of PNA during the BRV Extension Period, and up to 1 week during the Down-Titration Period for subjects in the Confirmatory Cohorts only. For subjects who remain in the study for up to 90 days of PNA and do not enter the long-term study, maximum BRV exposure per subject is expected to be up to 97 days (up to 90 days of PNA and up to 1 week for the Down-Titration Period).

All subjects who do not continue into the long-term study will proceed to the Safety Follow-Up Period, and a visit will occur 30±3 days after the final dose of BRV.

The end of the study is defined as the date of the last visit of the last subject in the study.

# 5.1.4 Planned number of subjects and sites

At least 42 evaluable subjects will be enrolled in this study, with at least 6 subjects in the Exploratory Cohort evaluable for the determination of BRV plasma concentrations and at least 36 subjects with evaluable PK data in the Confirmatory Cohorts (at least 12 subjects in each of the 3 Confirmatory Cohorts). At least 2 subjects undergoing hypothermia treatment will be included in the Exploratory Cohort and each of the 3 Confirmatory Cohorts.

The number of subjects in the Exploratory Cohorts might be increased, if deemed necessary, following the analysis of PK data.

#### 5.1.5 Anticipated regions and countries

Only sites in Europe are planned.

and Evaluation Periods for the Table 5–1 and Table 5–2, respectively.

Some performed according to the schedule provided in Table 5–4 for the Exproratory Cohort and in Table 5–5 for each Confirmatory Cohort.

The schedule of study assessments during the BRV Extension, Down-Titration (Confirmatory Cohorts only), and Safety Follow-Up Periods are presented in Table 5–3. Jon (Confirmate John Andrews of Support any marketing authorization and any extensions of the sead to support any marketing authorization and the support and support any marketing authorization and the support any marketing authorization and the support and support any marketing authorization and support and support any marketing authorization and support and support and support and support any marketing authorization and support and supp


24 May 2021 N01349

Table 5–1: Schedule of study assessments – Screening and Evaluation Periods (Exploratory Cohort)

| | | Screening Period <sup>a</sup> | | | | | | Ev | aluati | on Per | iod | 1 | y Comment | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Up to 36h | | | | | | | | | | OL 1 | | | | |
| Assessments | -36h<br>to 0h | Timepoint immediately before first BRV administration | Oh | 1h | 2h | 3h | 4h | 6h | | RV<br>10h | 12h | 24h | 27h | 34h | 36h | 48h |
| (Assessment window) | _ | - | VII | - | 211 | (±15min) | 711 | UII | W (10) | <u> </u> | | 30min) | | 3411 | 3011 | 4011 |
| Informed consent <sup>b</sup> | X | | | | | , | | 7 | <u></u> | X- | | | | | | |
| Subject identification card dispensing | X | | | | | | | 7/0 | | | | | | | | |
| Inclusion/exclusion criteria | X | X° | | | | × | 101 | | | | | | | | | |
| Demographic data | X | | | | | dico | | | | | | | | | | |
| Medical history including Apgar score and HIE | X | | | Ö | 7 | 366 | | | | | | | | | | |
| Vital signs | | X | Χ ( | .0. | dilo | X | | X | | | X | X | | | | X |
| Physical and neurological examination:<br>Sarnat scale for subjects with HIE | | X | 70 | oii | / | | | | | | | X | | | | X |
| Length | | X O | 37 | , | | | | | | | | | | | | |
| Body weight <sup>d</sup> | X | X iii | ) | | | | | | | | | X | | | | X |
| Head circumference <sup>e</sup> | | X | | | | | | | | | | | | | | |
| Primary cause of seizure | X | Mai | | | | | | | | | | | | | | X |
| Psychometric parameters:<br>N-PASS and EEG-parameters | X | and | | | | | | | | | | | | | | X |
| AED treatment (PB, MDZ, PHT, LEV, or LDC) | X <sup>j</sup> | 1000 | | | | | -X - | | | | | | | | | |
| Cohort Assignment | | S | X | | | | | | | | | | | | | |
| BRV infusion | 69 | | X | | | | | | | | X | X | | | X | |
| Heart rate monitoring | 150 | X | | X | X | X | | X | | X | X | X | X | X | X | X |
| BRV PK samples <sup>f</sup> | | | Xg | | | X | | | | X | ı | X | X | X | | |
| AED PK sample (only when PB and PHT are used) | | | | | | X | | | | | | | | | | |

## Table 5–1: Schedule of study assessments – Screening and Evaluation Periods (Exploratory Cohort)

| | | Screening Period <sup>a</sup> | | | | | | Ev | aluati | ion Per | iod | 170 | )" | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Up to 36h | | | | | | | | | C | )<br>O, | | | | |
| | -36h<br>to 0h | Timepoint immediately before first BRV | | | | | | | В | RV | Siori | | | | | |
| Assessments | toon | administration | 0h | 1h | 2h | 3h | 4h | 6h | | T0h | 12h | 24h | 27h | 34h | 36h | 48h |
| (Assessment window) | - | - | | - | | (±15min) | | | 6 | | (±3 | 30min) | | | | |
| Laboratory assessments (safety) | | $X^{\mathrm{h}}$ | | | | | | 6. | <i>y</i> . | | | | | | | X |
| Thompson scorei | | X | | | | | ( | 3/1 | | | | | | | | X |
| Mechanical ventilation | | | | • | | × | X- | | | • | | | • | | | |
| AE(s) | | | | | | //-X- | | | | | | | | | | |
| Concomitant medications | | | | , | 7 | ∂Q -X- | | | | | | | | | | |
| Medical procedures | | | | -OX | ,;(C | -X- | | | | | | | | | | |
| Infusion site reaction monitoring <sup>k</sup> | | | (X) | X | X | X | | X | | | X | X | | | X | X |
| Dispense BRV dosing diary | | P | V .X | 0, | | | | | | | | | | | | X <sup>l</sup> |
| Dispense BRV for the BRV Extension Period <sup>m</sup> | | \$0° | 200 | | | | | | | | | | | | | X |

AE(s)=adverse event(s); AED(s)=antiepileptic drug(s); BRV=brivaracetam; BZD(s)=benzodiazepine(s); COVID-19=coronavirus disease 2019; ENS=electroencephalographic neonatal seizures; HIE=hypoxic-ischemic encephalopathy; ICF=Informed Consent form; LDC=lidocaine; LEV=levetiracetam; MDZ=midazolam; N-PASS=neonatal pain, agitation, and sedation scale; PB=phenobarbital; PHT=phenytoin; PK=pharmacokinetic(s); SOC=standard of care

- <sup>a</sup> Screening Period is from signing and dating of the written ICF up to initiation of the first BRV dose.
- b Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the informed consent after the occurrence of seizures is confirmed on local VEEG. Continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s), during the conduct of the study.
- <sup>c</sup> The occurrence of ENS prior to entering the Evaluation Period must be confirmed by the local VEEG reader prior to initial BRV administration.
- <sup>d</sup> Measurement of body weight is mandatory prior to BRV treatment and optional at 24 and 48 hours. Dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the Evaluation Period.
- <sup>e</sup> Head circumference Baseline measurement should be taken within 7 days prior to drug administration, or at birth for subjects ≤7 days old.
- $^{\rm f}$  Following the first BRV infusion, 3 to 6 blood microsamples (60  $\mu$ L/sample) will be collected from each subject in the Exploratory Cohort.
- <sup>g</sup> The schedule of PK sampling for the Exploratory Cohort is also provided in Table 5–4.

## Table 5–1: Schedule of study assessments – Screening and Evaluation Periods (Exploratory Cohort)

| | | Screening Period <sup>a</sup> | | | | Eva | aluati | ion Per | riod | ~ 7.0 | 7 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Up to 36h | | | | | | | C | )<br>O, | | | | |
| | -36h | Timepoint immediately | | | | | | | ion | | | | | |
| | to 0h | to 0h before first BRV | | | | | В | RV | | | | | | |
| Assessments | | administration 0 | | 3h | 4h | 6h | 8h ( | TOh | 12h | 24h | 27h | 34h | 36h | 48h |
| (Assessment window) | - | - | - | (±15min) | | • | 15 | | (±3 | 30min) | | | • | • |

<sup>&</sup>lt;sup>h</sup> For Screening and determination of eligibility, use of laboratory data acquired prior to Screening per standard of care inside or outside the study site within 36 hours prior to the start of the Evaluation Period is allowed.

Table 5–2: Schedule of study assessments – Screening and Evaluation Periods (Confirmatory Cohorts)

| | Pei | ening<br>iod <sup>a</sup> | | | | | < | 500 | 30 | | Evalu | uation | Period | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -36h | Base-<br>line<br>Period <sup>b</sup> | | | | ~4 | nait | etino | | | | | | | | | | | | | |
| Assessments | to up<br>to -1 h | up<br>to -1h<br>to 0h | 0h | 3h | 6h | 8h | 9h | 10h | 12h | 15h | 18h | 21h | 24h | 27h | 34h | 36h | 48h | 60h | 72h | 84h | 96h <sup>c</sup> |
| (Assessment window) | - | - | - | (±15min) | | • | • | | | | | | (±30r | nin) | | | | | | | |
| Informed consent <sup>d</sup> | X | X | S | 30, | | | | | | | | -X- | | | | | | | | | |
| Subject identification card dispensing | X | 0,00 | 2 | | | | | | | | | | | | | | | | | | |
| Inclusion/ex-<br>clusion criteria | X | A Xe | | | | | | | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Thompson score will be used to measure the severity of HIE for subjects with HIE.

The recording of AEDs will include BZDs and opiates taken by the mother at the time of delivery. In addition, details regarding COVID-19 vaccination will be recorded as concomitant medication if the mother was pregnant or breastfeeding when vaccinated.

k Monitoring for BRV infusion site reactions should take place during and 30 minutes after the end of the infusion.

The BRV dosing diary will be dispensed only if the subject enters the BRV Extension Period.

<sup>&</sup>lt;sup>m</sup>Dispensing of BRV is only applicable if the subject enters the BRV Extension Period.

Table 5–2: Schedule of study assessments – Screening and Evaluation Periods (Confirmatory Cohorts)

| | | | | | | | | | | | | | | | | | | <del>\8\</del> . | | <u> </u> | <del></del> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | ening<br>riod <sup>a</sup> | | | | | | | | | Eval | uation ] | Period | | | | of ) | 7 | | | |
| | | o 36h | | | | | | | | | | | | | | | 5 | | | | |
| | СРС | Base- | | | | | | | | | | | | | | SIO | | 10C | | | |
| | | line | | | | | | | | | | | | | × | | | | | | |
| | -36h<br>to up | Period <sup>b</sup> | 01 | 21 | | 01 | 01 | 101 | 101 | 151 | 101 | 211 | 241 | 251 | 34h | | | | 501 | 0.41 | 0616 |
| | to up | up<br>to -1h | 0h | 3h | 6h | 8h | 9h | 10h | 12h | 15h | 18h | 21h | 24h | 27h | 334n | 36h | 48h | 60h | 72h | 84h | 96h <sup>c</sup> |
| Assessments | | to 0h | | | | | | | | | | | | 931 | | | | | | | |
| (Assessment window) | - | - | - | (±15min) | | | | | | | | | (±30r | nin) | | | | | | | |
| Demographic data | | X | | | | | | | | | | 1100 | | | | | | | | | |
| Medical history<br>including Apgar<br>score and HIE | | X | | | | | | | - ( | RT | ी अं | 8, | | | | | | | | | |
| Vital signs | | X | X | X | X | | X | | X | X | X | X | X | | | | X | | X | | X |
| Physical and<br>neurological<br>examination:<br>Sarnat scale for<br>subjects with<br>HIE | | X | | | | | × × | | N NIKO | | | | X | | | | X | | X | | X |
| Length | | X | | | | | SI | | | | | | | | | | | | | | |
| Body weight <sup>f</sup> | X | X | | | | Kn, | | | | | | | X | | | | X | | X | | X |
| Head circumference | | Xg | | | OK | 0 | | | | | | | | | | | | | | | |
| Primary cause of seizure | | X | | SUR | X | | | | | | | | | | | | | | | | X |
| Psychometric<br>parameters:<br>N-PASS and<br>EEG-parameters | | X | 2 15 | 9,0 | | | | | | | | | | | | | | | | | X |
| AED treatment<br>(PB, MDZ, PHT,<br>LEV | X <sup>n</sup> | XX | | | | _ | _ | | | | | | (X | | | | | | | | |

Table 5–2: Schedule of study assessments – Screening and Evaluation Periods (Confirmatory Cohorts)

| | Sere | ening<br>riod <sup>a</sup> | | <i>y</i> 400000 | | | | | | | Evalu | uation | Period | | | | or | 70, | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | Base-<br>line<br>Period <sup>b</sup> | | | | | | | | | | | | | × | ansio | SOT | | | | |
| Assessments | -36h<br>to up<br>to -1h | up<br>to -1h<br>to 0h | 0h | 3h | 6h | 8h | 9h | 10h | 12h | 15h | 18h | 21h | 24h | 27h | 34h | 36h | 48h | 60h | 72h | 84h | 96h <sup>c</sup> |
| (Assessment window) | - | - | - | (±15min) | | | | | | | | 4 | (±30) | nin) | | | | | | | |
| [≤60mg/kg/day],<br>or LDC) | | | | | | | | | | | | 1100 | illo | | | | | | | | |
| Cohort<br>Assignment | | | X | | | | | | | 7 | Si | 2 | | | | | | | | | |
| BRV infusionh | | | X | | | | | | Х_( | D | 0/ | | X | | | X | X | X | X | X | X |
| VEEGi | | | ı | l | ı | | | 1 | .0 | :10 | X- | I | I | I | | ı | | | | | |
| Heart rate<br>monitoring | | X | X | X | X | X | X | B | XU | X | X | X | X | X | X | X | X | X | X | X | X |
| BRV PK samples <sup>j</sup> | | | $\mathbf{X}^{\mathrm{j}}$ | X | | | | X | ) | | | | $(X)^{j}$ | | | | $(X)^{j}$ | | (X) <sup>k</sup> | | |
| AED PK sample<br>(only when PB<br>and PHT are<br>used) | | | | X | | 7 | rail | | | | | | | | | | | | | | |
| Laboratory<br>assessments<br>(safety) <sup>l</sup> | | X | | .0 | POK | 0. | | | | | | | X | | | | | | | | X |
| Thompson score <sup>m</sup> | | X | | SUL | | | | | | | | | | | | | | | | | X |
| Mechanical ventilation | | | c ( | 20,20 | | | | | | | -X | - | | | • | | • | | • | • | |
| AEs | | | 13 | | | | | | | | X- | • | | | | • | | | | | |
| Concomitant medications | | o't'o | | | | | | | | | X- | | | | | | | | | | |
| Medical procedures | | Sallin | | | | | | | | -] | X- | | | | | | | | | | |

Table 5–2: Schedule of study assessments – Screening and Evaluation Periods (Confirmatory Cohorts)

| | C | • | 1 | | | | | | | | | | | | | | _ | 19, | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | ening<br>iod <sup>a</sup> | | | | | | | | | Evalu | uation | Period | | | | Or | 7 | | | |
| | Up t | o 36h | | | | | | | | | | | | | | | 19 | | | | |
| | -36h | Base-<br>line<br>Period <sup>b</sup> | | | | | | | | | | | | | | insilo | SOT | | | | |
| Assessments | to up<br>to -1h | up<br>to -1h<br>to 0h | 0h | 3h | 6h | 8h | 9h | 10h | 12h | 15h | 18h | 21h | 24h | 27h . | 34h | 36h | 48h | 60h | 72h | 84h | 96h <sup>c</sup> |
| (Assessment | - | - | - | (±15min) | | | | | | | | | (±301 | nin) | | | | | | | |
| window) | | | | | | | | | | | | | 20 | | | | | | | | |
| AEDs <sup>n</sup> | | | | | | | | | | -, | X- | - À | | | | | | | | | |
| Infusion site<br>reaction<br>monitoring <sup>o</sup> | | | X | X | X | | | | X | 7 | 015 | Pilice | X | | | X | X | X | X | X | X |
| Neurodevelop-<br>mental testing<br>(Bayley-III<br>score) | | | | | | | | .0 | \<br>\ | 5 12 3 i | , | | | | | | | | | | Xp |
| Dispense BRV dosing diary | | | | | | | < | 3// | Silli | | | | | | | | | | | | Xq |
| Dispense BRV<br>for the BRV<br>Extension Period <sup>r</sup> | | | | | | | 2ix | Sille | | | | | | | | | | | | | X |

AE(s)=adverse events(s); AED(s)=antiepileptic drug(s); bid=twice daily; BRV=brivaracetam; BZD(s)=benzodiazepine(s); EEG=electroencephalography; ENS=electroencephalographic neonatal seizures; HIE=hypoxic-ischemic encephalopathy; ICF=Informed Consent form; iv=intravenous; LDC=lidocaine; LEV=levetiracetam; MDZ=midazolam; N-PASS=neonatal pain, agitation and sedation scale; PB=phenobarbital; PHT=phenytoin; PK=pharmacokinetic(s); VEEG=(multichannel) video-electroencephalography; (X)=optional for that day

- <sup>a</sup> Screening Period is from signing and dating of the written ICF up to initiation of the first BRV dose.
- b The duration of the Baseline EEG depends on seizure activity. Subjects with intermittent seizures will enter the Evaluation Period based on at least 1 hour of EEG recording. Subjects in status epilepticus will enter the Evaluation Period based on up to 30 minutes of EEG recording, ie, as soon as 15 minutes of continuous seizures or 50% of cumulative seizure activity is confirmed on EEG.
- <sup>c</sup> If subjects do not benefit from BRV treatment after 96 hours of BRV administration, BRV administration will be stopped and replaced by another AED; however, the subject's participation in the study will continue. Subjects discontinuing BRV treatment during the Evaluation Period should start the Down-Titration Period while completing the Evaluation Period in parallel for the full 96 hours.
- <sup>d</sup> Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the informed consent after the occurrence of seizures is confirmed on VEEG. Continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s), during the conduct of the study.

## Table 5–2: Schedule of study assessments – Screening and Evaluation Periods (Confirmatory Cohorts)

| | Per | ening<br>iod <sup>a</sup><br>o 36h | | | | | | | | | Evalı | uation | Period | | | ~~ | SOT | 7.0 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -36h | Base-<br>line<br>Period <sup>b</sup> | | | | | | | | | | | | | te | isio. | | | | | |
| Assessments | to up<br>to -1h | up<br>to -1h<br>to 0h | 0h | 3h | 6h | 8h | 9h | 10h | 12h | 15h | 18h | 21h | 24h | 27h | 34h | 36h | 48h | 60h | 72h | 84h | 96h <sup>c</sup> |
| (Assessment window) | - | - | - | (±15min) | in) (±30min) | | | | | | | | | | | | | | | | |

- <sup>c</sup> The occurrence of ENS during the Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS.
- f Measurement of body weight is optional at 24, 48, 72, and 96 hours. Dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the Evaluation Period.
- g Head circumference Baseline measurement should be taken within 7 days prior to drug administration, or at birth for subjects ≤7 days old.
- h Subjects will receive iv BRV 1mg/kg bid (2mg/kg/day), as recommended by the DMC on 05 Nov 2020 based on the results of the PK analysis of the Exploratory Cohort as well as an existing PK model from N01263.
- <sup>1</sup> Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements can be used as part of the Baseline assessment VEEG.
- <sup>j</sup> Following the first BRV infusion, 6 blood microsamples (60μL/sample) will be collected during the Evaluation Period from each subject.
- <sup>k</sup> The schedule of PK sampling for the Confirmatory Cohorts is also provided in Table 5–5.
- <sup>1</sup> For Screening and determination of eligibility, use of laboratory data acquired prior to Screening per standard of care inside or outside the study site within 36 hours prior to the start of the Evaluation Period is allowed.
- <sup>m</sup> Thompson score will be used to measure the severity of HIE for subjects with HIE.
- <sup>n</sup> The recording of AEDs will include BZDs and opiates taken by the mother at the time of delivery. In addition, details regarding COVID-19 vaccination will be recorded as concomitant medication if mother was pregnant or breastfeeding when vaccinated.
- <sup>o</sup> Monitoring for BRV infusion site reactions should take place during and 30 minutes after the end of the infusion. The assessment will be conducted hourly from 0h to 3h of the BRV Evaluation Period.
- <sup>p</sup> The assessment of the Bayley-III score at 96-hour time point only applies to subjects who directly roll-over from the Evaluation Period to the long-term study due to their age at enrollment into N01349.
- <sup>q</sup> The BRV dosing diary will be dispensed only if the subject enters the BRV Extension Period.
- <sup>r</sup> Dispensing of BRV is only applicable if the subject enters the BRV Extension Period.
Table 5-3: Schedule of study assessments - BRV Extension Period and Safety Follow-Up Period (Exploratory and Confirmatory Cohorts)

| Assessments | | BR | Down-<br>Titration<br>Period <sup>a</sup> | Safety<br>Follow-Up<br>Period <sup>b</sup> | | |
|---|---|---|---|---|---|---|
| | EPV1 <sup>c</sup> | EPV2 <sup>d</sup> | Unscheduled<br>Visit | Telephone<br>Contact | Up to 1<br>week | 30 days |
| (Assessment window) | (±2<br>days) | - | | | - | (±3 days) |
| Informed consent <sup>e</sup> | X | X | | | X | 601 |
| Vital signs | | X | X | | X . | X |
| Physical and neurological examination: Sarnat scale for subjects with HIE | | X | X | | XfS | X |
| Biometric parameters: length,<br>body weight and head<br>circumference | | | | andar | 7 | X |
| Primary cause of seizure | | | | 100 | Xf | X |
| Psychometric parameters: N-PASS | | | | dicatile | X | X |
| BRV administration or dispense | X | X <sup>g</sup> | 28× 202 | 97 | $X^h$ | |
| BRV return | | X | CO dilo. | | | |
| 1-hour VEEG | | | City | | Xi | |
| Laboratory assessments (safety) | | XB | Nillo Xº | | | X |
| Neurodevelopmental testing (Bayley-III score) | | Xi | | | | |
| AE(s) | | aike | | -X- | | |
| Concomitant medications | , 4 | 10 | | -X- | | |
| Medical procedures | Kno | | | -X- | | |
| AEDs <sup>k</sup> | N. C. | | | -X- | | |
| Infusion site reaction monitoring <sup>1</sup> | X | X | X | | X | |
| Confirmation/diagnosis of epilepsy | | X | | | | |
| Update on Medical History | | X <sup>m</sup> | | | | X <sup>n</sup> |
| Review BRV dosing diary | X | X | X | X | _ | |

AE(s)=adverse event(s); AED(s)=antiepileptic drug(s); BRV=brivaracetam; BZD(s)=benzodiazepine(s); EEG=electroencephalography; EPV=Extension Period Visit; HIE=hypoxic-ischemic encephalopathy; iv=intravenously; N-PASS=neonatal pain, agitation, and sedation scale; VEEG=(multichannel) video-electroencephalography

Note: An Unscheduled Visit and a Telephone Contact are only applicable to subjects receiving oral BRV at home.

<sup>a</sup> A Down-Titration Period of up to 1 week applies only to subjects in the Confirmatory Cohorts. The Down-Titration Period is recommended for subjects who discontinue BRV treatment prior to completion of the Evaluation Period, who do not proceed to the BRV Extension Period, or start the BRV Extension Period but do not enter the long-term study. Subjects discontinuing BRV treatment during the Evaluation Period can continue assessments pertaining to the Evaluation Period, except the collection of blood microsamples for the determination of BRV plasma


**UCB** N01349 Clinical Study Protocol Brivaracetam

### Schedule of study assessments - BRV Extension Period and Safety **Table 5-3:** Follow-Up Period (Exploratory and Confirmatory Cohorts)

| Assessments | | BR | Down-<br>Titration<br>Period <sup>a</sup> | Safety<br>Follow-Up<br>Period <sup>b</sup> | | |
|---|---|---|---|---|---|---|
| | EPV1 <sup>c</sup> | EPV2 <sup>d</sup> | Unscheduled<br>Visit | Telephone<br>Contact | Up to 1<br>week | 30 days |
| (Assessment window) | (±2<br>days) | - | | | - | (±3 days) |

concentrations. Those subjects should start the Down-Titration Period in parallel to completing the Evaluation Period.

- Subjects will enter the Safety Follow-Up Period if they withdraw from the study at any time, or do not proceed to the BRV Extension Period, or complete the Down-Titration Period. This visit will occur 30±3 days after the last administration of BRV. For subjects unable to return to the hospital due to COVID-19, the Safety Follow-up Visit can be performed remotely. In this case vital signs, the physical and neurological examination, biometric and psychometric parameters, and the laboratory assessment may not be performed.
- <sup>c</sup> Subjects will attend EPV1 at 7±2 days after completion of the Evaluation Period. For subjects unable to return to the hospital due to COVID-19, EPV1 can be performed remotely if BRV oral solution was dispensed at the time when the subject completed the Evaluation Period.
- d Subjects will attend EPV2 when they enter the long-term study. Before entering the long-term study, subjects must have been switched to BRV oral solution and be able to tolerate it. Subjects who have not been switched to BRV oral solution will not be permitted to continue into the long-term study. The timing of switching from iv to oral solution will be at the discretion of the Investigator. Subjects will continue to receive the same BRV dose administered at the end of the Evaluation Period.
- e Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the informed consent after the occurrence of seizures is confirmed on VEEG. Continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s), during the conduct of the study.
- f To be performed on the first day of the Down-Titration Period only.
- g If the subject enters the long-term study, no study drug from N01349 will be dispensed in EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration (only applicable to subjects from the Confirmatory Cohorts).

  h The Down-Titration steps and duration may be adjusted at the Investigator's discretion.
- <sup>i</sup> Video-EEG will only apply to subjects of the Confirmatory Cohorts who complete the study after the Evaluation Period. The VEEG will be recorded for at least 1 hour on the final day of the Down-Titration Period. Additional VEEGs can be performed at any time during the Down-Titration Period at the Investigator's discretion.
- <sup>j</sup> Bayley-III assessment will be assessed for subjects continuing into the long-term study, in countries where a validated translation is available.
- k The recording of AEDs will include AEDs (BZDs and opiates) taken by the mother at the time of delivery. In addition, details regarding COVID-19 vaccination will be recorded as concomitant medication if mother was pregnant or breastfeeding when vaccinated.
- <sup>1</sup> Infusion site reactions will only be monitored for subjects receiving iv BRV. Monitoring for BRV infusion site reactions should take place during and 30 minutes after the end of the infusion.
- <sup>m</sup> Updated Medical History should be recorded at EPV2 for subjects entering the long-term study.
- <sup>n</sup> Updated Medical History should be recorded for subjects not entering the long-term study.
- Laboratory assessment (safety) only required for Unscheduled Visits performed during the BRV Extension Period.


#### Table 5-4: Schedule for PK Sampling (Exploratory Cohort)

| Assessment | 48-hour Evaluation Period Time relative to the start of the most recent BRV infusion | | | | | |
|---|---|---|---|---|---|---|
| | | Day 1 | | Day 2 <sup>a</sup> | | |
| | 30-60min <sup>b</sup> | 30-60min <sup>b</sup> 2-4h 8-12h | | 30-60min | 30-60min 2-4h | |
| BRV PK samples <sup>c</sup> | X | X | X | X | X | X |
| AED PK sample | | X <sup>d</sup> | | | | ċ |
| AED=antiepileptic dru | ıg; BRV=brivarace | tam; h=hours; | min=minutes | s; PK=pharmacokir | netic(s) | 18, |
| Note: Blood for PK sa | imples should be dr | awn from a li | ne different to | that of the BRV ir | ifusion. | d |
| a Blood sampling is or | nly needed on Day | 2 if subjects a | re dosed with | BRV on Day 2. | | 35 |
| b The first PK sample | should be collected | 1 30 to 60 min | utes after the | start of the BRV in | fusion. | ,011 |
| <sup>c</sup> The BRV PK sampli | ing timepoints for t | he first 3 sam | ples of the Ex | ploratory Cohorts a | re as follows: | 30 to |


<sup>&</sup>lt;sup>a</sup> Blood sampling is only needed on Day 2 if subjects are dosed with BRV on Day 2.

<sup>&</sup>lt;sup>b</sup> The first PK sample should be collected 30 to 60 minutes after the start of the BRV infusion.

in acrts an AV infusic at 48-hour Eval attraction and application and a superior <sup>c</sup> The BRV PK sampling timepoints for the first 3 samples of the Exploratory Cohorts are as follows: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. The second set of 3 samples will be collected at the same timepoints on the second day of the 48-hour Evaluation Period.

<sup>&</sup>lt;sup>d</sup> The AED PK sample should be collected 3 hours after the start of the initial BRV administration.

**UCB** 

Schedule for PK Sampling (Confirmatory Cohorts) Table 5-5:

| Assessment | 96-hour Evaluation Period | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Time relative to the start of the most recent BRV infusion | | | | | | | | | | |
| | Day 1 Day 2 | | | | | | Day 3 | | | Day 4 | | |
| | 30-60mi<br>n <sup>a</sup> | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h |
| BRV PK samp<br>les <sup>b</sup> | X | X | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| AED PK sample | | Xc | | | | | | | | | JONS | |

AED=antiepileptic drug; BRV=brivaracetam; h=hours; PK=pharmacokinetic(s); min=minutes; (X)=optional for that day

Note: Blood for PK samples should be drawn from a line different to that of the BRV infusion.

#### 5.3 Schematic diagrams

Figure 5–1 displays a schematic overview of the study for the Exploratory Cohort and the Screening and Evaluation Periods of this Cohort are presented in detail in Figure 5–2. Figure 5–3 displays a schematic overview of the study for the Confirmatory Cohorts and the Screening and This document cannot be used to support any marke Evaluation Periods of these Cohorts are presented in detail in Figure 5–4.

<sup>&</sup>lt;sup>a</sup> The first PK sample will be collected 30 to 60 minutes after the start of the BRV infusion.

<sup>&</sup>lt;sup>b</sup> The BRV PK sampling timepoints for the first 3 samples of the Confirmatory Cohorts are as follows: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. The second set of 3 PK samples will be collected within the same timeframes as the first set on one of the following days: either Day 2 (post-24 hours), OR Day 3 (post-48 hours) OR Day 4 (post-72 hours), It is acceptable if these samples are drawn on different days.

<sup>&</sup>lt;sup>c</sup> The AED PK sample should be collected 3 hours after the start of the initial BRV administration.

Figure 5–1: Schematic overview of the study (Exploratory Cohort)



Figure 5–2: Screening and Evaluation Periods (Exploratory Cohort)



AED=antiepileptic drug; bid=twice daily; BRV=brivaracetam; EEG=electroencephalogram; ENS=electroencephalographic neonatal seizures; ICF=Informed Consent form; iv=intravenous; LEV=levetiracetam; LDC=lidocaine; MDZ=midazolam; PB=phenobarbital; PHT=phenytoin Note: The Screening Period is from signing and dating of the written ICF up to initiation of the first BRV dose.

<sup>a</sup> BRV to be administered in addition to another AED.

Figure 5–3: Schematic overview of the study (Confirmatory Cohorts)





AED=antiepileptic drug; BRV=brivaracetam; EEG=electroencephalogram; ENS=electroencephalographic neonatal seizure; LEV=levetiracetam; LDC=lidocaine; MDZ=midazolam; PB=phenobarbital; PHT=phenytoin

<sup>b</sup> Duration of the Baseline EEG depending on seizure activity:

- for subjects with intermittent ENS: 1 hour
- for subjects in status epilepticus: up to 30 minutes

<sup>&</sup>lt;sup>a</sup> Concomitant treatment with AEDs is permitted to continue in parallel with BRV treatment if subjects are on a stable dose from 1 hour prior to initiation of BRV treatment. Changes to concomitant AEDs are permitted from 3 hours onward following first BRV administration).

### 5.4 Rationale for study design and selection of dose

### 5.4.1 Rationale for study design

The current accepted medical practice (ie, standard of care) for neonatal seizures is initial treatment with PB with rapid progression to treatment with MDZ for patients without adequate seizure control after 2 doses of PB. In more than 50% of subjects, seizures are not controlled after first-line treatment with PB or other AEDs, and subsequent treatment with additional AEDs does not significantly improve seizure control (van Rooij et al, 2013b; Castro Conde et al, 2005; Boylan et al, 2004; Painter et al, 1999). Thus, study N01349 was designed for a flexible treatment of ENS, and only those subjects who do not have adequate seizure control with previous AED treatment will be permitted to continue in the study.

As the patient population of neonates with ENS is limited, the 2-step design of this study will allow confirmation (or adjustment) of dosing based on results from the first step (Exploratory Cohort) and evaluation of BRV efficacy in the second step (Confirmatory Cohorts). This adaptive design allows confirmation of dose and collection of PK, safety, and efficacy data, thereby potentially providing rapid access to alternative treatment in neonates.

The frequency, voltage, and morphology of the discharges may change within an individual seizure and between seizures in an individual neonate. At enrollment, subjects must be at least 34 weeks of CGA. In addition, term neonates up to 27 days of PNA and preterm neonates up to 40 weeks of CGA and 27 days of PNA can be enrolled. Neonates undergoing hypothermia treatment (eg, for the treatment of HIE) will also be enrolled.

Although newer AEDs are efficacious for the treatment of seizures in adults and older children, limited progress has been made in the treatment of neonatal seizures (Pressler et al, 2015; Pressler and Mangum 2013; Tulloch et al, 2012). Thus, clinical studies to assess the efficacy and safety of new treatment options in neonates are warranted.

### 5.4.2 Rationale for dose selection

The doses planned to be applied in this study are based on pediatric data collected in N01263 subjects (overall 96 subjects in the age range of 1 month to 17 years with the following number of subjects per pediatric age group: 1 month to <2 years of age, 29 subjects; 2 years to <6 years of age, 26 subjects; 6 years to <12 years of age, 24 subjects; 12 years to <16 years of age, 17 subjects). A physiological-based PK model was used to extrapolate the PK of BRV from older children. It is estimated that a dose of BRV 0.5mg/kg bid, administered to neonatal subjects, should yield the same BRV exposure range in plasma as observed in older children receiving the same dose on a mg/kg body weight basis. In adults, a similar exposure is achieved with a dose of 25mg bid, which represents the lowest dose approved for adults. A dose of 2mg/kg bid should result in similar exposure in neonates as compared to adults receiving 100mg bid (the highest approved dose in adults). Given the uncertainties of the extrapolation, as well as the variability and rapid changes in neonatal physiology, these predictions may or may not be precise; however, large discrepancies are not expected.

Based on the extrapolation explained above, subjects who enter the Exploratory Cohort will receive an initial low dose of BRV (0.5mg/kg [bid]). A starting dose of BRV 0.5mg/kg was selected because this dose offers a wide safety margin (4-fold) with respect to the highest BRV dose administered and tolerated in older children and adults with epilepsy. Simultaneously, a


dose of BRV 0.5mg/kg is potentially therapeutically beneficial to subjects in this study. In adjunctive treatment studies, a dosage of BRV 25mg bid is effective for POS in adult subjects with epilepsy.

For subjects who enter the Confirmatory Cohorts, the dosing frequency of BRV will be determined based on the PK findings of the Exploratory Cohort (see Section 5.1). The dose of BRV to be administered in the Confirmatory Cohorts will be determined by the evaluation of plasma samples collected in the Exploratory Cohort, as well as by the PK modeling of N01263 data described above, and should not exceed the range of plasma concentrations observed in children ≥1 month old who received BRV 4mg/kg/day. The plasma concentration of BRV 4mg/kg/day for neonates is predicted to be approximately equivalent to the plasma concentrations observed in adults who receive BRV 200mg/day. The dose in neonates to reach the same plasma concentrations will be confirmed or adapted upon completion of enrollment and analysis of PK and safety data from the Exploratory Cohort involving the DMC.

The BRV dose used in the Confirmatory Cohorts will be based on recommendations made by the DMC. Based on the DMC meeting held on 05 Nov 2020, the BRV dose and frequency selected for the Confirmatory Cohorts is 1mg/kg bid (2mg/kg/day). Based on data from the Confirmatory Cohorts, the BRV dose may be further adjusted in a staggered approach as determined by the DMC.

Furthermore, the posology of BRV for the Confirmatory Cohorts is proposed as an approximately 15-minute iv infusion in consideration of the following and is based on PK and safety data available from subjects ≥1 month old in N01263 and N01266:

BRV is well-tolerated orally up to 200mg/day in adult subjects with epilepsy and in children 1 month old to 16 years of age receiving up to 4mg/kg/day. In adults, a single iv infusion over 15 minutes or a bolus of BRV up to 150mg/day is well-tolerated. A dose of BRV 4mg/kg/day is predicted to be approximately equivalent to the highest BRV dosage (200mg/day) received by adults. In addition, iv BRV is bioequivalent to the same dose given orally in healthy adults when given as a bolus or as a 15-minute infusion.

Dose adjustment of BRV for the change in the formulation (switching from iv to oral solution) used during this study is not required as the AUC of BRV is bioequivalent between the following formulations: a tablet, a 15-minute iv infusion, and a bolus iv injection. In adults, iv BRV was administered to healthy volunteers, as well as subjects with epilepsy. Results showed that iv BRV was well-tolerated at all doses, up to 150mg per iv injection. Furthermore, the dose of BRV oral solution is bioequivalent to BRV tablets; therefore, dose adjustment is not required when switching between these formulations.

#### SELECTION AND WITHDRAWAL OF SUBJECTS 6

#### 6.1 Inclusion criteria

To be eligible to participate in this study, all of the following criteria must be met:

- 1. An Independent Ethics Committee (IEC)-approved written ICF is signed and dated by the parent(s) or legal representative(s).
- 2a. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite receiving previous AED treatment for the treatment of electroencephalographic seizures.
  - The occurrence of ENS during an up to 1-hour period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS.
- 3. Subject is male or female and must be at least 34 weeks of CGA. In addition, term neonates up to 27 days of PNA and preterm neonates up to 40 weeks of CGA and 27 days of PNA can be enrolled.
- 4. Subject weighs at least 2.3kg at the time of enrollment.
- 5. Subjects with or without concomitant hypothermia treatment.

#### 6.2 **Exclusion criteria**

Subjects are not permitted to be enrolled in the study if any of the following criteria are met:

- 1a. Subject receiving AED treatment other than PB, MDZ, PHT, LEV (≤60mg/kg/day), or LDC for the treatment of seizures prior to or at the time of enrollment (Confirmatory Cohorts only).
- 2. Subject with seizures responding to any of the following: previous AED treatment immediately prior to BRV treatment, pyridoxine treatment, or correction of metabolic disturbances (hypoglycemia, hypomagnesemia, or hypocalcemia).
- 3. Subject requires extra corporeal membrane oxygenation.
- 4. Subject has seizures related to prenatal maternal drug use or drug withdrawal.
- 5. Subject has known severe disturbance of hemostasis, as assessed by the Investigator.
- 6. Subject has a poor prognosis for survival, as judged by the Investigator.
- aminotransferase (AST), alam with the following exception:

  For subjects with period if initial and rether 7a. Subject has 2x upper limit of normal (ULN) of any of the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP),

For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable, if initial and peak elevation of liver function tests (LFTs) occurs within 5 days after birth, and the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia.

The determination of ULN will be based on the subject's gestational age (GA) and the site's normal range values for the respective GA.8a. Subject has direct (conjugated) bilirubin levels >2mg/dL.

- I Subject with a severe cardiac condition, including subject with a diagnosis or signs of long QT syndrome (LQTS), and subject with a family history of LQTS.

  6.3 Withdrawal criteria

  Parent(s) or legal representative(s) are forwithout prejudice to a without prejudice to a subject with a family history of LQTS.

Subjects **must** be withdrawn from the study if any of the following occur;

- 1. The Sponsor or a regulatory agency requests withdrawal of the subject.
- 2. Parent(s) or legal representative(s) withdraw their consent for the subject to participate.
- 3. Subject is treated with prohibited concomitant medications as defined in this protocol.
- 4a. Subject has direct (conjugated) bilirubin levels >2mg/dL.
- 5. Subject requires phototherapy or exchange transfusion due to elevation of total bilirubin.
- 6a. Subject has AST, ALT or ALP values 3x ULN, with the following exception:

For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable for continuation in the study, if initial and peak elevation of LFTs occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within a few days after birth, and subsequent normalization until up to day 14 after birth).

In case AST, ALT or ALP elevation ≥5x ULN occurs within 5 days after birth, study drug must be discontinued and LFTs retested within 24 hours. If AST, ALT and ALP are confirmed to be <5x ULN, the subject may restart study drug after consultation with and approval by the Medical Monitor.

The determination of ULN will be based on the subject's GA and the site's normal range values for the respective GA.

Subjects may be withdrawn from the study if any of the following events occur:

- 7a. Subject experiences prolongation of seizure duration, a worsening of seizure burden, or emergence of new seizure type considered by the Investigator to require intervention.
- Investigator may withdraw subject due to any medical condition, based on clinical judgment and discretion.
- 9a. Subject has AST, ALT or ALP values between >2x and  $\le 3x$  ULN, with the following exception:

For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable for continuation in the study, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within a few days after birth, and subsequent normalization until up to day 14 after birth).

The determinations of ULN will be based on the subject's GA and the site's normal range values for the respective GA.

10. Subject has rapidly increasing total bilirubin without requiring or being expected to require phototherapy or exchange transfusion; the subject's withdrawal will be at the discretion of the Investigator.

Investigators should attempt to obtain information on subjects in the case of withdrawal. The Investigator should document his/her effort (date and summary of the phone call and copy of the written message in the source documents) to complete the final evaluation. All results of these evaluations and observations, together with a narrative description of the reason(s) for removing the subject, must be recorded in the source documents. The eCRF must document the primary reason for withdrawal.

Investigators should contact the Medical Monitor, whenever possible, to discuss the withdrawal of a subject in advance.

### 6.3.1 Potential drug-induced liver injury IMP discontinuation criteria

Subjects with potential drug-induced liver injury (PDIM) must be assessed to determine if the investigational medicinal product (IMP) must be discontinued. In addition, all concomitant medications that are not medically necessary should also be discontinued.

The PDILI criteria below require immediate and permanent discontinuation of IMP:

- Subject has direct (conjugated) bilirubin >2mg/dL.
- Subject has AST, ALT or ALP values >3x ULN, with the following exception:

For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable for continuation in the study, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within few days after birth, and subsequent normalization until up to day 14 after birth).

In case AST, ALT or ALP elevation ≥5x ULN occurs within 5 days after birth, study drug must be discontinued and LFTs retested within 24 hours. If AST, ALT and ALP are confirmed to be <5x ULN, the subject may restart study drug after consultation with and approval by the Medical Monitor.

The determination of ULN will be based on the subject's GA and the site's normal range values for the respective GA.

• Subject requires or is expected to require phototherapy or exchange transfusion due to elevation of total bilirubin values.

Investigators should attempt to obtain information on subjects in the case of IMP discontinuation to complete the final evaluation. Subjects with PDILI should not be withdrawn from the study


until investigation and monitoring are complete. All results of these evaluations and observations, as well as the reason(s) for IMP discontinuation and subject withdrawal (if applicable), must be recorded in the source documents. The eCRF must document the primary reason for IMP discontinuation.

### 7 STUDY TREATMENTS

### 7.1 Description of investigational medicinal products

Only the following study drug will be supplied by UCB for N01349:

• BRV 10mg/mL iv solution in a 5mL vial.

For subjects who are switched to BRV oral solution in the BRV Extension Period, the following will be supplied by UCB:

• BRV oral solution, at concentrations of 10mg/mL, will be supplied in 300mL glass bottles.

Refer to the IMP Handling Manual for further details on the handling of BRV.

There is no placebo or reference product.

After the completion of the study, BRV treatment per SOC may be continued as prescribed but will not be provided by the Sponsor.

### 7.2 Treatments to be administered

Subjects in the Exploratory Cohort will be dosed during the Evaluation Period with BRV (0.5mg/kg bid) according to the sites standard procedures. Treatment with AEDs per SOC (first-line, second-line, or subsequent treatment) will continue in parallel with BRV treatment.

For subjects who enter the Confirmatory Cohorts, the dosing of BRV (1mg/kg bid [2mg/kg/day]) has been determined based on the PK findings of the Exploratory Cohort. The DMC will continue to monitor the PK and safety of the subjects and dosing may be adjusted as new data are available. Administration of BRV is proposed as approximately 15-minute iv infusions. Treatment with previous AEDs (PB, MDZ, PHT, LEV [≤60mg/kg/day], or LDC) during the Evaluation Period is permitted to continue if the subject is on a stable dose from 1 hour prior to initiation of the BRV treatment.

Subjects can switch from iv to oral BRV at any time during the BRV Extension Period.

For subjects who are switched to BRV oral solution, the dose will be measured using the appropriate syringes (1mL, 3mL or 10mL) with an adaptor able to fit all the bottle sizes. Oral solution should not be mixed with other liquids prior to administration.

### 7.3 Packaging

Brivaracetam (sterile solution for iv infusion and oral solution) is manufactured, packaged, and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. Brivaracetam is suitably packaged in such a way as to be protected from deterioration during transport and storage.

Brivaracetam sterile solution for iv infusion 10mg/mL will be packaged in 5ml vials.

Brivaracetam 10mg/mL oral solution will be packaged in 300mL type-III amber glass bottles with child-resistant tamper evident polypropylene screw closures. Syringes of 1mL, 3mL or 10mL will be provided with an adaptor able to fit all the bottle sizes.

Other AED treatments will be used for this study and will not be provided or covered by the Sponsor.

### 7.4 Labeling

Clinical drug supplies will be labeled in accordance with the current International Council on Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and GMP and will include any locally required statements. If necessary, labels will be translated into the local language.

### 7.5 Handling and storage requirements

The Investigator (or pharmacist/designee) is responsible for the safe and proper storage of BRV at the site. Brivaracetam stored by the Investigator is to be kept in a secured area with limited access according to the storage conditions mentioned on the label.

Appropriate storage conditions must be ensured either by controlling the temperature (eg, room, refrigeration unit) or by completing a temperature log in accordance with local requirements on a regular basis (eg, once per working day), showing actual minimum/maximum temperatures reached over the time interval.

Additional information pertaining to the handling of BRV, a Schedule V drug, is provided in the IMP Handling Manual.

In case an out-of-range temperature is noted, it must be immediately reported as per instructions contained in the IMP Handling Manual.

The Investigator (or designee) will instruct the subject to store the IMP following the instructions on the label.

## 7.6 Drug accountability

A Drug Accountability form will be used to record BRV dispensing and return information on a by-subject basis and will serve as source documentation during the course of the study. Details of any BRV lost, damaged (due to breakage or wastage), not used, partially used, disposed of at the study site, or returned to the Sponsor or designee must also be recorded on the appropriate forms. All supplies and pharmacy documentation must be made available throughout the study for UCB (or designee) to review.

The Investigator (or designee) is responsible for retaining all used, unused, and partially used containers/ bottles of BRV until returned or destroyed.


The Investigator may assign some of the Investigator's duties for drug accountability at the study site to an appropriate pharmacist/designee.

The Investigator must ensure that BRV is used only in accordance with the protocol.

tensions of variations thereof. Periodically, and/or after completion of the clinical phase of the study, all used (including empty containers)/partially used, unused, damaged and/or expired IMP containers/ bottles must be reconciled and either destroyed at the site according to local laws, regulations, and UCB Standard Operating Procedures (SOPs), or returned to UCB (or designee). Investigational medicinal product intended for the study cannot be used for any other purpose than that described in this protocol.

### 7.7 Procedures for monitoring subject compliance

After each iv BRV administration, empty/used BRV containers must be kept.

All unused IMP and empty IMP containers/bottles must be accounted for or returned to the site. For subjects treated at home during the BRV Extension Period, parent(s) or legal representative(s) should be advised to return all unused IMP and empty IMP bottles to the site. Drug accountability must be done in the presence of the subject's parent(s) or legal representative(s) and site staff to obtain explanations regarding discrepancies in compliance with the dosing regimen. Drug accountability must be recorded on the Drug Accountability form.

Site personnel who are administering iv BRV will record information about all doses administered, including the target dose, actual dose administered, and the dates and times of initiation and completion of each iv administration. If the actual dose is less or more than the target dose, the reason a partial or excessive dose was administered will be recorded.

Intravenous BRV solution will be administered under supervision of the Investigator or his/her designee. The noninjected volume will be recorded in the eCRF. Compliance with the recommended duration of the iv administration will also be assessed by recording the start time and the stop time in the eCRF.

Noncompliance will be recorded for subjects who are administered <75% or >125% of the planned BRV dose. If, in the Investigator's opinion, there is persistent noncompliance with the subject's BRV administration, the Sponsor, in conjunction with the Investigator, will make a decision as to whether the subject should be withdrawn from the study.

### **Concomitant treatments and medications** 7.8

#### 7.8.1 Permitted concomitant treatments (medications and therapies)

Concomitant freatment with non-AEDs is permitted for the Exploratory and Confirmatory Cohort(s) at any time throughout the study.

parallel with BRV treatment if subjects are on a stable dose from 1 hour prior to initiation of BRV treatment. Changes to concomitant AEDs are permitted from 3 hours onwerd 6.11 first BRV administration. BRV treatment. Changes to concomitant AEDs are permitted from 3 hours onward following


#### 7.8.2 Prohibited concomitant treatments (medications and therapies)

For the Confirmatory Cohorts, subjects will not be permitted to change concomitant treatment for neonatal seizures for the first 3 hours after the first BRV administration.

Rescue medication

Any treatment initiation with a new AED, or any increase of dose or frequency of an existing concomitant AED for the treatment of seizures during the Evaluation Period is considered recent treatment. Rescue medication can be given at any time if considered necessary livestigator.

However, during the T

However, during the Evaluation Period rescue medication should not be administered – if possible – in the following time frames:

During the first 3 hours after the initial dose of BRV for the Confirmatory Cohorts. If this occurs, subjects will be considered BRV nonresponders for the evaluation of the main efficacy variable.

### 7.9 Blinding

This is an open-label study and, therefore, no blinding is required.

#### Randomization and numbering of subjects 7.10

Because N01349 is an open-label, single-arm study, subjects will not be randomized to any treatment groups. The first 6 subjects meeting the eligibility criteria will be assigned to the Exploratory Cohort. Subsequent subjects will be assigned to the Confirmatory Cohorts.

An IRT system will be used to assign eligible subjects to a treatment regimen based on a predetermined packaging schedule provided by the Sponsor. The IRT will generate individual assignments for subject kits of BRV as appropriate, according to the cohort assignment and dosing schedule.

After the ICF has been signed and dated, the subject will be enrolled in the study. The Investigator or designee will contact the IRT and provide brief details about the subject enrolled. Each subject will be assigned a 5-digit number that serves as the subject identifier throughout the study. The IRT will allocate kit numbers to the subject based on the subject number during the course of the study. The subject number will be required in all communications between the Investigator or designee and the IRT on a particular subject. Subject numbers and kit numbers will be tracked via the IRT.

## STUDY PROCEDURES BY VISIT

A continuous consent process will be followed. Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the ICF after the occurrence of seizures has been confirmed by VEEG. During the course of the study, parent(s) or legal representative(s) will be updated about the care of their neonate, and continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal

 representative(s). Continuous consent will be documented in the subjects' medical charts and eCRF.

### 8.1 Exploratory Cohort

### 8.1.1 Screening Period

The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal representative(s) up to initiation of the first BRV dose. Any AEs, AEDs, concomitant medications, and medical procedures will be collected after the ICF is signed. The subject's eligibility to participate in this study will be assessed. The subject identification card will be dispensed.

The Screening Period starts up to 36 hours prior to the first administration of BRV. Phenobarbital, MDZ, PHT, LEV, or LDC may have been administered prior to the subject's enrollment into the study and/or at a location other than the study site.

Subjects will enter the Evaluation Period and start BRV treatment as soon as the occurrence of ENS per inclusion criterion 2a is confirmed by the Investigator based on local EEG. If preferred by the Investigator, the central VEEG reader can be consulted to confirm the required ENS.

The following assessments will be performed immediately before the first administration of BRV is initiated:

- Verification of inclusion/exclusion criteria. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite treatment with 1 or more AEDs administered per SOC
- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- Length
- Body weight
- Head circumference (to be taken within 7 days prior to drug administration, or at birth for subjects ≤7 days old)
- Heart rate monitoring
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology)
- Thompson score (for subjects with HIE)
- Mechanical ventilation
- AEs as reported by the Investigator
- Recording of AEDs, concomitant medications, and medical procedures

Laboratory measurements will be performed by local laboratories unless historical data is available. Historical safety laboratory assessments, previously collected as standard of care, may

be accepted from referring hospitals as measurement prior to first use of BRV if performed 36 hours prior to the start of the Evaluation Period. In this case, test results will be considered medical history. Prior laboratory assessment results should be available and verified prior to initiation of the first BRV infusion.

At the determination of the Investigator, subjects achieving adequate seizure control following AED treatment per SOC will be considered AED responders. Those subjects will be classified as screen failures and will not be assigned to BRV treatment.

### 8.1.2 Evaluation Period

The first BRV infusion marks the starting point of the 48-hour Evaluation Period.

An initial iv dose of BRV (0.5mg/kg) will be administered as an approximately 15-minute infusion. At the discretion of the Investigator, 3 additional iv BRV doses can be administered, up to a total of 4 iv BRV doses (0.5mg/kg bid) during the 48-hour BRV Evaluation Period.

The following assessments will be performed after the end of the first BRV infusion:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature; at 0, 3, 6, 12, 24, and 48 hours)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity; at 24 hours and 48 hours)
- Body weight (optional [at 24 and 48 hours]; dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the Evaluation Period)
- Confirmation of the primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes [at 48 hours])
- N-PASS and EEG parameters for the assessment of sedation (at 48 hours)
- Video-EEG
- Heart rate monitoring (1, 2, 3, 6, 10, 12, 24, 27, 34, 36, and 48 hours)
- Three to 6 PK samples (30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion; the same timepoints apply to the first and second day of the 48-hour Evaluation Period)
- Collection of AED PK sample 3 hours after the start of the initial BRV administration
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology [at 48 hours])
- Thompson score (for subjects with HIE [at 48 hours])
- Mechanical ventilation
- AEs as reported by the Investigator

- AEDs, concomitant medications, and medical procedures
- Infusion site reaction monitoring

### 8.1.3 BRV Extension Period

The BRV Extension Period is intended to bridge the time until subjects are old enough to participate in the long-term study. Subjects completing the Evaluation Period at a PNA of at least 28 days may directly roll over to the long-term study, if they meet the eligibility criteria. Those patients are not required to enter the BRV Extension Period.

Brivaracetam

At the end of the Evaluation Period, subjects who benefit from BRV treatment may enter the BRV Extension Period in accordance with the Investigator's opinion. Subjects participating in the BRV Extension Period will need to remain at the study site as long as BRV is administered iv or via the enteral route. Only subjects able to swallow oral BRV should be allowed to be treated at home during the BRV Extension Period. In this case the parent(s) or legal representative(s) will receive a dosing diary to record the home administration of oral BRV. If oral BRV administration is not possible, the subjects will be invited to return to the study site and receive iv BRV as indicated below. It will not be possible for subjects to receive iv BRV at any institutions other than the study site.

All subjects who participate in the BRV Extension Period must be offered entry into the long-term study, if they meet the eligibility criteria. Subjects will participate in the BRV Extension Period until they reach a stable condition that will allow them to enter the long-term study, if epilepsy is confirmed. The maximum anticipated duration of the BRV Extension Period per subject is up to 28 days of PNA (+7 days). For subjects entering the BRV Extension Period, study drug will be dispensed at the end of the Evaluation Period. Subjects not continuing the BRV treatment after they completed the Evaluation Period will not enter the BRV Extension Period but proceed immediately to the Safety Follow-Up Period (see Section 8.1.4).

For subjects treated at home with oral BRV during the BRV Extension Period, a total of 2 on-site visits may take place (Extension Period Visit 1 [EPV1], Extension Period Visit 2 [EPV2]). Extension Period Visit 1 will be performed at 7±2 days after completion of the Evaluation Period (see Section 8.1.3.1). Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study (see Section 8.1.3.2). If the long-term study is performed outside the N01349 hospital, an interval of up to 3 days between the N01349 EPV2 and follow-up study Entry Visit is allowed. In addition, an Unscheduled Visit or Telephone Contact can be performed, as needed. For subjects treated during the BRV Extension Period at the study site with iv BRV assessments will be performed at timepoints described for EPV1 and EPV2.

During the BRV Extension Period, subjects may continue receiving iv BRV but must switch to BRV oral solution before entering the long-term study. The timepoint of the switch from iv to oral solution will be at the discretion of the Investigator. Subjects who are not able to be dosed with BRV oral solution when they reach 28 days of postnatal age may continue in the BRV Extension Period for an additional 7 days; subjects who are not able to be switched to BRV oral solution by the end of the additional 7 days of the BRV Extension Period will not be eligible for enrollment in the long-term study.

Subjects who participate in the BRV Extension Period will continue to receive the same BRV dosage administered at the end of the Evaluation Period (ie, BRV 0.5mg/kg bid). The BRV dose extensions or variations thereof. should not be increased, but may be decreased at the discretion of the Investigator.

#### 8.1.3.1 **Extension Period Visit 1**

The EPV1 will be performed at 7±2 days after completion of the Evaluation Period. The following assessments will be performed:

- BRV dispense
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Review of BRV dosing diary (only if oral BRV is administered at home)
- Infusion site reaction monitoring (for subjects treated with iv BRV)

For subjects unable to return to the hospital due to COVID-19, EPV1 can be performed remotely if BRV oral solution was dispensed at the time when the subject completed the Evaluation Period.

#### 8.1.3.2 **Extension Period Visit 2**

The EPV2 should be performed on the same day when the subject enters the long-term study. The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- BRV administration/dispense. If the subject enters the long-term study, no study drug from N01349 will be dispensed at EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration (only applicable to subjects from the Confirmatory Cohorts).
- BRV return
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology)
- Bayley-III (for subjects continuing into the long-term study only and only for subjects enrolled in countries where a validated translation is available)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Review of BRV dosing diary (only if oral BRV is administered at home)
- Infusion site reaction monitoring
- Confirmation/diagnosis of epilepsy
- Medical History (for subjects entering the long-term study)

### 8.1.3.3 Unscheduled Visit

An Unscheduled Visit can take place at any time during the BRV Extension Period. The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Review of BRV dosing diary Infusion site reaction monitoring

### 8.1.3.4 Telephone Contact

For subjects receiving oral BRV at home, a Telephone Contact can be performed at any time during the BRV Extension Period. The following information will be collected by the Investigator:

- AEs
- AEDs, concomitant medications, and medical procedures
- Discussion of BRV dosing diary

### 8.1.4 Safety Follow-Up Period

Subjects will proceed to the Safety Follow-Up Period if they do not enter the BRV Extension Period. The visit will occur 30±3 days after the final administration of BRV. The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- Body weight and length and head circumference
- Primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes)
- N-PASS
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Medical history (for subjects not entering the long-term study)

For subjects unable to return to the hospital due to COVID-19, the Safety Follow-Up Visit can be performed remotely. In this case vital signs, the physical and neurological examination, biometric and psychometric parameters, and the laboratory assessment may not be performed.

### 8.2 **Confirmatory Cohorts**

Based on the PK and safety data review of the Exploratory Cohort by the DMC, enrollment and BRV dosing for the Confirmatory Cohorts will begin. Three consecutive Confirmatory Cohorts (n=12 each) are planned. A PK and safety data review will be performed after completion of each of the 3 Confirmatory Cohorts. During the PK and safety data review, the recruitment of ionsor subjects will continue.

#### 8.2.1 Screening Period

The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal representative(s) of the subject up to initiation of the first BRV dose. Any AEs, AEDs, concomitant medications, and medical procedures will be collected after the ICF is signed. The subject's eligibility to participate in this study will be assessed. The subject identification card will be dispensed.

The Screening Period starts up to 36 hours prior to the first administration of BRV. The treatment with one or more of the following AEDs prior to or at the time of enrollment: PB, MDZ, PHT, LEV (<60mg/kg/day), or LDC (first-line, second-line, or subsequent treatment; choice of treatment, dose, and dosing regimen at the Investigator's discretion) may have started prior to the subject's enrollment in the study and/or at a location other than the study site.

At the determination of the Investigator, subjects achieving adequate seizure control following any of the following AEDs: PB, MDZ, PHT, LEV ( $\leq 60 \text{mg/kg/day}$ ), or LDC will be considered AED responders. Those subjects will be classified as screen failures and will not be assigned to BRV treatment.

#### 8.2.1.1 **Baseline Period**

The Baseline Period will be up to 1 hour immediately prior to the start of initial BRV infusion and depend on seizure activity:

- For subjects with intermittent ENS: at least 1 hour prior to entering the Evaluation Period
- For subjects in status epilepticus: up to 30 minutes prior to entering the Evaluation Period. At least 15 minutes of continuous seizures, or 50% of cumulative seizure activity during a 30-minute interval are to be confirmed on EEG before the administration of BRV can start.

As soon as subjects are considered to be in status epilepticus, steps required for the preparation of the initial BRV infusion can be initiated (eg, assignment of BRV kits through interactive IRT and the dilution of BRV solution for iv infusion), even if the required EEG recording is not completed by that time.

The occurrence of ENS during the Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements (eg., ability for immediate cloudbased central review) can be used as part of the Baseline assessment VEEG.

The following assessments will be performed during the Baseline Period:

- Verification of inclusion/exclusion criteria. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the up to 1 hour prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite treatment with one or more AEDs per SOC
- Demographic data
- Medical history (including Apgar score)
- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- Length
- Body weight
- Head circumference (Baseline measurement should be taken within 7 days prior to drug administration, or at birth for subjects ≤7 days old)
- Primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes)
- N-PASS and EEG parameters for the assessment of sedation
- Video-EEG
- Heart rate monitoring
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology)
- Thompson score (for subjects with HIE)
- Mechanical ventilation
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures

Baseline laboratory measurements will be performed by local laboratories unless historical data is available. Historical safety laboratory assessments, previously collected as standard of care, may be accepted from referring hospitals as Baseline measurement if performed 36 hours prior to the start of the Evaluation Period. In this case, test results will be considered medical history. Prior laboratory assessment results should already be available at Baseline and verified prior to initiation of BRV administration.

### 8.2.2 Evaluation Period

The first administration of BRV marks the starting point of the Evaluation Period.

Up to 8 iv doses of BRV (1mg/kg bid) will be administered as an approximately 15-minute infusion during the 96-hour BRV Evaluation Period. The AED treatment initiated prior to first

administration of BRV can be continued if the subject is on a stable dose for at least 1 hour at the time the first BRV infusion is initiated.

If subjects do not benefit from BRV treatment after 96 hours of BRV administration, BRV

It subjects in the Confirmatory Cohort receive <8 BRV doses, those subjects are allowed to continue study participation and complete study assessments per Table 5–2 with the exception of PK blood sampling. Those subjects should start the Down-Titration Period while completing the Evaluation Period in parallel for the full 96 hours.

After the enrollment of subject

given.

The following assessments will be performed after BRV administration:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature; at 0, 3, 6, 9, 12, 15, 18, 21, 24, 48, 72, and 96 hours)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity [at 24, 48, 72, and 96 hours])
- Primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes [at 96 hours])
- N-PASS and EEG parameters for the assessment of sedation (at 96 hours)
- Body weight (optional [at 24, 48, 72 and 96 hours]; dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the **Evaluation Period**)
- Video-EEG
- Heart rate monitoring
- Up to 6 PK samples (30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion; the same timepoints apply to the first day and 1 of the 3 following days of the 96-hour Evaluation Period).
- Collection of AED PK sample 3 hours after the start of the initial BRV administration
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology [at 24 and 96 hours])
- Thompson score (for subjects with HIE [at 96 hours])
- Mechanical ventilation

- Bayley-III (for subjects continuing into the long-term study only and only for subjects enrolled in countries where a validated translation is available)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Infusion site reaction monitoring

#### 8.2.3 **BRV Extension Period**

Valiations the reof The BRV Extension Period is intended to bridge the period until subjects are old enough to participate in the long-term study. Subjects completing the Evaluation Period at a PNA of at least 28 days may directly roll over to the long-term study, if they meet the eligibility criteria. Those patients are not required to enter the BRV Extension Period.

At the end of the Evaluation Period, subjects who benefit from BRV treatment may enter the BRV Extension Period in accordance with the Investigator's opinion. Subjects participating in the BRV Extension Period will need to remain at the study site as long as BRV is administered iv. Only subjects able to swallow oral BRV should be allowed to be treated at home during the BRV Extension Period. If oral BRV administration is not possible, the subjects will be invited to return to the study site and receive iv BRV as indicated below. It will not be possible for subjects to receive iv BRV at any institutions other than the study site. All subjects who participate in the BRV Extension Period must be offered entry into the long-term study, if they meet the eligibility criteria. Subjects will participate in the BRV Extension Period until they reach a stable condition that will allow them to enter the long-term study, if epilepsy is confirmed. The maximum anticipated duration of the BRV Extension Period per subject is up to 90 days of PNA. For subjects entering the BRV Extension Period, study drug will be dispensed at the end of the Evaluation Period. Subjects not continuing the BRV treatment after they completed the Evaluation Period will not enter the BRV Extension Period but proceed immediately to the Down-Titration Period (see Section 8.2.4).

For subjects treated at home with oral BRV during the BRV Extension Period, a total of 2 on-site visits may take place (EPV1 and EPV2). Extension Period Visit 1 will be performed at 7±2 days after completion of the Evaluation Period (see Section 8.2.3.1). Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study (see Section 8.2.3.2). If the long-term study is performed outside the N01349 hospital, an interval of up to 3 days between the N01349 EPV2 and long-term study Entry Visit is allowed. In addition, an Unscheduled Visit or Telephone Contact can be performed, as needed. For subjects treated during the BRV Extension Period at the study site with iv BRV, assessments will be performed at timepoints described for EPV1 and EPV2.

During the BRV Extension Period, subjects may continue receiving iv BRV but must switch to BRV oral solution before entering the long-term study. The timepoint of the switch from iv to oral solution will be at the discretion of the Investigator

Subjects who participate in the BRV Extension Period will continue to receive the same BRV dosage administered at the end of the Evaluation Period (ie, BRV 1mg/kg bid). The BRV dose should not be increased, but may be decreased at the discretion of the Investigator.


In the event that a long-term study is temporarily not available after the planned duration of the BRV Extension Period (28 [+7] days of PNA), subjects are allowed to remain in the BRV Jextensions or variations thereof Extension Period until they reach a PNA of up to 90 days. For those subjects, the assessments planned for Unscheduled Visits (Section 8.2.3.3) will be conducted in intervals of approximately 30 days during the prolonged Extension Period.

#### 8.2.3.1 **Extension Period Visit 1**

This visit will be performed at 7±2 days after completion of the Evaluation Period. The following assessments will be performed:

- BRV dispense
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Review of BRV dosing diary (only if oral BRV is administered at home)
- Infusion site reaction monitoring (for subjects treated with iv BRV)

For subjects unable to return to the hospital due to COVID-19, EPV1 can be performed remotely if BRV oral solution was dispensed at the time when the subject completed the Evaluation Period.

#### 8.2.3.2 **Extension Period Visit 2**

This visit should be performed on the same day when the subject enters the long-term study. The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- BRV administration/dispense. If the subject enters the long-term study, no study drug from N01349 will be dispensed at EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration (only applicable to subjects from the Confirmatory Cohorts).
- BRV return
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology)
- Bayley-III (for subjects continuing into the long-term study only and only for subjects enrolled in countries where a validated translation is available)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Review of BRV dosing diary (only if oral BRV is administered at home)
- Infusion site reaction monitoring (for subjects treated with iv BRV)
- Confirmation/diagnosis of epilepsy

Medical History (for subjects entering the long-term study)

#### **Unscheduled Visit** 8.2.3.3

An Unscheduled Visit can take place at any time during the BRV Extension Period. The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology) and any exten
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Review of BRV dosing diary
- Infusion site reaction monitoring

For subjects who remain in the BRV Extension Period for a prolonged duration (ie, until they reach a PNA of 90 days), these assessments will be conducted at intervals of 30 ( $\pm$ 3 days).

#### 8.2.3.4 **Telephone Contact**

For subjects receiving oral BRV at home, a Telephone Contact can be performed at any time during the BRV Extension Period. The following information will be collected by the Investigator:

- **AEs**
- AEs
  AEDs, concomitant medications, and medical procedures

### **Down-Titration Period** 8.2.4

A Down-Titration Period of up to 1 week is recommended for subjects who complete the Evaluation Period, but do not enter the BRV Extension Period, discontinue BRV during the Evaluation Period, or start the BRV Extension Period but do not continue into the long-term study for any reason. The Down-Titration steps and duration may be adjusted at the Investigator's discretion.

The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity; to be performed on the first day of the Down-Titration Period only)
- Primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes; to be performed on the first day of the Down-Titration Period only)

- **N-PASS**
- **BRV** administration
- lons of variations thereof At least a 1-hour video-EEG on the final day of the Down-Titration Period (during the Down-Titration Period, additional VEEGs can be performed at the Investigator's discretion)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Infusion site reaction monitoring

#### Safety Follow-Up Period 8.2.5

Subjects will proceed to the Safety Follow-Up Period once they complete the Down-Titration Period. This visit will occur 30±3 days after the final administration of BRV. The following assessments will be performed:

- Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)
- Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)
- Body weight and length and head circumference
- Confirmation of the primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes)
- N-PASS
- Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology)
- AEs as reported by the Investigator
- AEDs, concomitant medications, and medical procedures
- Medical History (for subjects not entering the long-term study)

For subjects unable to return to the hospital due to COVID-19, the Safety Follow-Up Visit can be performed remotely. In this case vital signs, the physical and neurological examination, biometric and psychometric parameters, and the laboratory assessment may not be performed.

### **ASSESSMENT OF PHARMACOKINETIC VARIABLES** 9

### Pharmacokinetic sampling and handling 9.1

For the determination of plasma concentrations of BRV and BRV metabolites, up to 6 blood microsamples (60µL/sample) will be collected per subject in the Exploratory (3 to 6 blood microsamples) and Confirmatory Cohorts (up to 6 blood microsamples) at 3 predetermined timepoints per day. An additional microsample (60µL) will be collected per subject for the determination of plasma concentrations of concomitant AEDs (PB and PHT).

Pharmacokinetic samples will be obtained either through a venous or arterial catheter or taken from routinely performed heel-pricks. Blood for PK samples should be drawn from a line different to that of the BRV infusion. Three BRV PK samples of blood will be collected at the following predetermined timepoints at the first day of the Evaluation Period: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. For the Exploratory Cohort the same timepoints apply to the second day of the 48-hour Evaluation Period. For the Confirmatory Cohort(s), the second set of 3 BRV PK samples will be collected at the same timepoints on 1 of the other days of the 96-hour Evaluation Period. It will be acceptable if these samples are drawn on different days. The AED PK sample should be collected 3 hours after the start of the initial BRV administration. The timepoints for the collection of PK samples are described in Table 5–4 for the Exploratory Cohort and in Table 5–5 for the Confirmatory Cohorts.

Additional opportunistic blood samples for the PK analysis (Leroux et al, 2015) may be obtained at the Investigator's discretion at any time during the Evaluation Period. As opportunistic blood samples will be taken from routine laboratory blood samples, they are not considered an additional burden for the neonates. The plan for microsampling in N01349 is consistent with blood sampling schema in other neonatal studies (Allegaert and van den Anker, 2015; Jullien et al, 2015; O'Hara et al, 2015; Zhao and Jacqz-Aigrain, 2015; Zhao et al, 2014).

Exact dosing and sampling times will be recorded in the eCRF. Sampling times of will be shippy cook and marketing authoritation and marketing authoritation. pre-determined PK samples may be subject to change after analysis and review of data from the Exploratory Cohort to complete the PK profile.

The full set of a subject's PK plasma samples will be shipped for analyses after the subject has

### 9.2 Pharmacokinetic sample shipment

Instructions on blood sample collection, processing, storage, and labeling/shipping will be provided in the laboratory manual for this study. On arrival, the samples will be stored at -20°C, until analysis.

Shipments due to arrive over the weekend or holidays must be avoided. For PK samples collected over a weekend in the site, these should be stored at -20°C and must be shipped under frozen conditions (packaged with dry ice) to the central laboratory on the following Monday. Prior to any shipment, an agreement must be made with the analytical laboratory for receipt of the samples.

### 10 ASSESSMENT OF EFFICACY

# 10.1 Assessment of the secondary efficacy variables (Confirmatory Cohort[s] only)

The main secondary efficacy variable is:

Proportion of responders to BRV treatment from Baseline to 3 hours after the initial BRV dose

A BRV responder is defined as a subject who achieved the following reduction in seizure burden (ENS in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment:

At least 80% reduction in nonsevere seizure burden
 (Nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in all 30-minute timespans)

OR

- At least 50% reduction in severe seizure burden

A severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan. Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to  $\leq$ 30 minutes, >30 to  $\leq$ 60 minutes, >60 to  $\leq$ 90 minutes, and >90 to  $\leq$ 120 minutes

For this study, an ENS is defined as EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug.

For the analysis of the main secondary efficacy variable (Section 4.2.1), subjects who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS during the first 3 hours after initiation of BRV treatment will be considered BRV nonresponders.


For the analysis of the following secondary efficacy variables, subjects who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS following the first 3 hours after initiation of BRV treatment will be considered BRV responders:

- Proportion of subjects with at least 80% reduction in nonsevere seizure burden from Baseline to 3 hours after the initial BRV treatment
- Proportion of subjects with at least 50% reduction in severe seizure burden from Baseline to 3 hours after the initial BRV treatment
- Absolute reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period
- Percent reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period
- Proportion of BRV responders at the end of the 96-hour Evaluation Period
- Proportion of subjects who are seizure-free (100% reduction in seizure burden from Baseline) at 24 hours following the start of initial BRV treatment, categorized by subjects with nonsevere or severe seizure burden at Baseline
- Time to reduction in seizure burden for BRV responders (defined as the first timepoint when BRV responder criteria were met)
- Seizure freedom at the end of the Down-Titration Period
- Rate of at least 50% reduction in ENS frequency per hour from Baseline to the end of the 96-hour Evaluation Period
- Proportion of subjects who are seizure-free by time interval at 3 hours, at 3-hour intervals thereafter through 24 hours, and every 12 hours to 24 hours following the start of the initial BRV treatment
- Absolute difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion
- Percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion

# 10.2 Assessment of other efficacy variables

Other efficacy variables will include:

- Absolute and percentage reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
- Categorized percentage reduction from Baseline to the end of the 96-hour Evaluation Period in seizure burden (<-25% [worsening], -25% to <25% [no change], 25% to <50%, 50% to <80%, and ≥80%)

- Proportion of BRV responders by time interval at evaluation periods of 0 to 3 hours, >3 to 6 hours, >6 to 12 hours, >12 to 24 hours, >24 to 36 hours, >36 to 48 hours, >48 to 72 hours, and >72 to 96 hours after the start of initial BRV treatment
- Proportion of subjects who switch over from BRV to another AED during the 96-hour **Evaluation Period**
- Proportion of responders to other treatment during the 96-hour Evaluation Period (including at the end of the 96-hour Evaluation Period, and by time intervals: 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment)

(A responder to other treatment is defined as at least 80% reduction in nonsevere seizure burden from start of other treatment to end of other treatment or at least 50% reduction in severe seizure burden from the initiation of other treatment to end of other treatment during the 96-hour Evaluation Period).

To further evaluate BRV efficacy, a descriptive comparison will be conducted of the main efficacy variable data from N01349 with published responder rates for one or more AED treatments from literature (historical control group matched in age and condition) effective for the treatment of neonatal seizures in subjects of similar age (<29 days of PNA) and condition (neonatal seizures as noted in N01349 eligibility criteria). A recent study (Weeke et al, 2016) provides response rates for second line AED treatment of neonatal seizures in a similar population and with primary endpoints comparable to N01349. Results from this study, as well as results from other studies available in the literature at the time of N01349 completion and with populations and efficacy endpoints comparable to N01349, will be used for these comparisons.

#### Seizure burden 10.3

Seizure burden is defined as the total minutes of ENS per hour. Seizure burden information will be recorded for the Confirmatory Cohorts via a continuous VEEG. Seizure burden at Baseline will be evaluated over a period of at least 1 hour (subjects with intermittent seizures) or up to 30 minutes (subjects in status epilepticus).

Electroencephalographic neonatal seizures are defined as EEG seizures occurring for at least 10 seconds.

Seizure counts/seizure burden will be based on data collected using continuous VEEG. The VEEG recording will be evaluated by the local physician or central reader to evaluate eligibility of the subject. The VEEG recordings will subsequently be confirmed and quantified by the central reader at the end of the study.

### **ASSESSMENT OF SAFETY**

# Adverse events is document

### **Definitions**

#### 11.1.1.1 Adverse event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In order to ensure complete safety data collection, all AEs occurring during the study (ie, after the signing of the ICF), including any pretreatment and posttreatment periods required by the protocol, must be recorded even if no IMP was taken but specific study procedures were conducted. This includes all AEs not present prior to the signing of the ICF and all AEs that recurred or worsened after the signing of the ICF.

Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the Investigator from the subject's history or based on assessments performed prior to the first administration of BRV.

#### 11.1.1.2 Serious adverse event

Once it is determined that a subject experienced an AE, the seriousness of the AE must be determined. An SAE must meet 1 or more of the following criteria:

- Death
- Life-threatening

(Life-threatening does not include a reaction that might have caused death had it occurred in Significant or persistent disability/incapacity

Congenital and 1. 7.

- Congenital anomaly/birth defect (including that occurring in a fetus)
- Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious

(Important medical events may include, but are not limited to, allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse).

Initial inpatient hospitalization or prolongation of hospitalization

(A patient admitted to a hospital, even if he/she is released on the same day, meets the criteria for the initial inpatient hospitalization. An emergency room visit that results in admission to the hospital would also qualify for the initial inpatient hospitalization criteria. However, emergency room visits that do not result in admission to the hospital would not qualify for this criteria and, instead, should be evaluated for 1 of the other criteria in the definition of serious [eg, life-threatening adverse experience, important medical event].

Hospitalizations for reasons not associated with the occurrence of an AE [eg, preplanned surgery or elective surgery for a pre-existing condition that has not worsened or manifested in an unusual or uncharacteristic manner do not qualify for reporting. For example, if a subject has a condition recorded on his/her medical history and later has a preplanned surgery for this condition, it is not appropriate to record the surgery or hospitalization as an SAE, since there is no AE upon which to assess the serious criteria. Please note that, if the pre-existing condition has worsened or manifested in an unusual or uncharacteristic manner.

This communication and the serious adverse events

The following list of anticipated SAEs has been identified, as these events are anticipated to occur in the population studied in this protocol at some frequency that is independent of drug exposure:

Respiratory distress syndrome

Convulsion 

This original list will remain in effect for the duration of the protocol.

In addition, the following are anticipated SAEs in babies with HIE:

### Acute

- Lany
  Lipratory failure

  Multiorgan failure

  Severe encephalopathy with coma
  Status epilepticus
  Cerebral oedema
  Death

  nic
  rebral palsy

  ual Imparis

### Chronic

- Visual Impairment
- **Epilepsy**
- Learning Difficulties
- Behavioural Difficulties

These lists do not change the Investigator's obligation to report all SAEs (including anticipated SAEs) as detailed in Section 11.1.2.3.

#### 11.1.1.3 Adverse events of special interest

and any extensions or variations thereoft. An AE of special interest is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.

The following will be considered AEs of special interest for the study population:

- Autoimmune nephritis
- **Nephritis**
- Nephritis allergic
- Tubulointerstitial nephritis
- Tubulointerstitial nephritis and uveitis syndrome
- Potential drug-induced liver injury as indicated by:
  - Direct (conjugated) bilirubin >2mg/dL
  - Condition requiring phototherapy or exchange transfusion due to elevation total of bilirubin values
  - AST, ALT or ALP values ≥3x ULN according to the subject's GA and the site's normal values for that GA, with the following exception:

For subjects with perinatal asphyxia, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of the elevation of LFT is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within few days after birth, and subsequent normalization until up to day 14 after birth) only AST, ALT or ALP elevation  $\geq 5x$  ULN must be reported as an AE of special interest.

### Procedures for reporting and recording adverse events 11.1.2

The subject's parent(s) or legal representative(s) will be given the opportunity to report AEs spontaneously. A general prompt will also be given at each study visit to detect AEs. For example:

"Did you notice anything unusual about your child's health (since your last visit)?"

The requirements for recording AEs are detailed in Articles 16 and 17 of the Clinical Trials Directive (CTD) 2001/20/EC1 published in 2001, which establishes specific provisions regarding the conduct of clinical trials, in particular relating to the implementation of GCP. Articles 16 and 17 of the CTD outline the legal obligations for both the Investigator and Sponsor for the recording and reporting of all AEs and reactions.

In line with GCP, from the signing of the ICF, the Investigator will evaluate the subject for occurrence of any AEs based on continued observation and medical notes throughout the study. Serious AEs, AEs that are considered related to the medicinal (investigational) product, AEs leading to discontinuation, BRV infusion site reactions, or AEs considered by the Investigator to be critical to the safety evaluation of the protocol will also be recorded on the Adverse Event eCRF. Further guidance on the reporting requirements for AEs is provided in Figure 11–1. The
The deciment denerate beautre appearant with the property of t

Figure 11–1: Adverse event reporting flowchart



AE=adverse event; BRV=brivaracetam; eCRF=electronic case report form; SAE=serious adverse event This AE reporting flowchart details the decision-making process for recording AEs in the eCRF. Serious AEs and nonserious AEs (that are potentially related to the study drug, result in discontinuation, are considered BRV infusion site reactions, or are considered by the Investigator to be critical to the safety evaluation) are to be recorded in the eCRF. All AEs will be recorded in the subject's medical notes.

Examples of AEs critical to the safety evaluation of the protocol include:

- AEs that might alter the current benefit-risk assessment of BRV use in neonatal seizures
- AEs that would be sufficient to consider changes in the study protocol
- AEs that would be sufficient to consider changes in the overall conduct of the study

#### 11.1.2.1 **Description of adverse events**

When recording an AE, the Investigator should use the overall diagnosis or syndrome using Details for completion of the Adverse Event eCRF (including judgment of relationship to IMP) are described in the eCRF Completion Guidelines.

11.1.2.2 Rule of repetition of an adverse event

An increase in the intensity of an AE should lead to the repetition of the AE L.

• The outcome date of the first AE AL.

the second standard medical terminology, rather than recording individual symptoms or signs. The eCRF

- the same as the start date of the repeated AE, and the outcome of "worsening"
- The AE verbatim term being the same for the first and repeated AE, so that the repeated AE can be easily identified as the worsening of the first one

### Additional procedures for reporting serious adverse events 11.1.2.3

If an SAE is reported, UCB must be informed within 24 hours of receipt of this information by the site (see contact information for SAE reporting listed in the Serious Adverse Event Reporting section at the front of the protocol). The Investigator must forward to UCB (or its representative) a duly completed "Investigator SAE Report Form for Development Drug" (SAE Report form) provided by UCB, even if the data are incomplete, or if it is obvious that more data will be needed in order to draw any conclusions. Information recorded on this form will be entered into the global safety database.

An Investigator SAE Report form will be provided to the Investigator. The Investigator SAE Report form must be completed in English.

It is important for the Investigator, when completing the SAE Report form, to include the assessment as to a causal relationship between the SAE and the IMP administration. This insight from the Investigator is very important for UCB to consider in assessing the safety of the IMP and in determining whether the SAE requires reporting to the regulatory authorities in an expedited manner.

Additional information (eg, autopsy or laboratory reports) received by the Investigator must be provided within 24 hours. All documents in the local language must be accompanied by a translation in English, or the relevant information included in the same document must be summarized in the Investigator SAE Report form.

The Investigator is specifically requested to collect and report to UCB (or its representative) any SAEs (even if the Investigator is certain that they are in no way associated with the IMP), up to 30 days from the end of the study for each subject, and to also inform participating subjects parent(s) or legal representative(s) of the need to inform the Investigator of any SAE within this period. Serious AEs that the Investigator thinks may be associated with the IMP must be reported to UCB regardless of the time between the event and the end of the study.

Upon receipt of the SAE Report form, UCB will perform an assessment of expectedness of the reported SAE. The assessment of the expectedness of the SAE is based on the IB.

#### 11.1.2.4 Immediate reporting of adverse events

The following AEs must be reported immediately (see Section 11.1.2.3):

- Serious adverse event (see Section 11.1.1.2):
  - Adverse event that the Investigator classifies as serious by the above definitions regardless of causality
  - New onset or worsening of status epilepticus after the administration of BRV
- s of variations thereof Suspected transmission of an infectious agent via a medicinal product (see Section 1.1.4) anyetier
- Adverse event of special interest (see Section 11.1.1.3)

### 11.1.3 Follow-up of adverse events

An AE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, and AEs of special interest; further details regarding follow-up of PDILI events are provided in Section 11.2.1.4.

If an AE is ongoing at the end of the study for a subject, follow-up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems that it is clinically significant, or until the subject is lost to follow-up. If no follow-up is provided, the Investigator must provide a justification. The follow-up will usually be continued for 30 days after the subject has discontinued his/her IMP.

Information on SAEs obtained after clinical database lock will be captured through the Patient Safety (PS) database without limitation of time.

#### 11.1.4 Suspected transmission of an infectious agent

A suspected transmission of infectious agent is defined as any infection that is temporally related to the administration of the medicinal product with no other likely cause. The Medical Monitor should be contacted immediately. No further medicinal product from that specific batch should be administered. Infections should be treated according to normal clinical practice.

For the purposes of reporting, any suspected transmission of an infectious agent via a medicinal product should be considered as an SAE; such cases must be reported immediately, recorded in the AE module of the eCRF, and followed as any other SAE. Any organism, virus, or infectious particle (eg, prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

### 11,105 Overdose of investigational medicinal product

Excessive dosing (beyond that prescribed in the protocol and including overdose) should be recorded in the eCRF. Any SAE or nonserious AE associated with excessive dosing must be followed as any other SAE or nonserious AE. These events are only considered AEs or SAEs if there are associated clinical signs and symptoms.

## 11.1.6 Safety signal detection

Selected data from this study will be reviewed periodically to detect as early as possible any safety concern(s) related to BRV so that Investigators, parent(s) or legal representative(s) of the clinical study subject, regulatory authorities, and IECs will be informed appropriately and as early as possible.

The Study Physician or medically qualified designee/equivalent will conduct an ongoing review of SAEs and perform ongoing SAE reconciliations in collaboration with the PS representative.

No formal interim analysis is planned for this study; however, PK and safety data will be presented to and reviewed by a DMC. It was originally planned that the DMC would convene to review the PK and safety data every 6 months; however, due to the low enrollment rate, the interval between DMC meetings may exceed 6-month intervals, at the discretion of the DMC. The DMC will oversee the safety of the study by convening to review the PK and safety data after the 6 subjects from the Exploratory Cohort have completed or withdrawn from the study. The PK and safety data will again be reviewed after each of the 3 Confirmatory Cohorts (12 subjects each) have completed or withdrawn from the study.

The DMC will consist of 3 voting members, none of whom will be involved in the conduct of the study, either by management or participation. As appropriate for the stage of development and accumulated experience with BRV, medically qualified personnel at UCB may identify additional safety measures (eg, AEs, vital signs, laboratory or heart rate results) for which data will be periodically reviewed during the course of the study.

Serious adverse events and AEs of special interest will be monitored and will be triaged by the Study Physician and UCB PS in real time. After this triage, events will be passed on to the DMC as appropriate. The DMC or Sponsor can convene an ad hoc DMC meeting to review the data and make recommendations on the continuation or modification of the study. The objectives and procedures for the DMC will be detailed in the DMC Charter.

A DMC will be in place for the duration of this study (see Section 13.8.3).

# 11.2 Laboratory measurements

Safety laboratory assessments will be performed as shown in Table 5–1, Table 5–2, and Table 5–3. Blood samples will be collected in line with Section 13.2 of the "Ethical Considerations for Clinical Trials on Medicinal Products Conducted with the Paediatric Population" (European Union Commission ad hoc group, 2008). If clinically significant abnormalities are observed, the laboratory measurements may be performed more frequently at the Investigator's discretion.

Laboratory measurements, including laboratory assessments for PDILI, will be performed by local laboratories unless historical data is available. Historical safety laboratory assessments, previously collected as standard of care, may be accepted from referring hospitals as Baseline measurement if performed 36 hours prior to the Evaluation Period.

As part of routine assessments performed by local laboratories, the parameters shown in Table 11–1 and Table 11–2 will be measured.

### Table 11-1: Mandatory laboratory measurements

| Hematology | Biochemistry |
|----------------------|-------------------------------|
| Basophils | Calcium |
| Eosinophils | Chloride |
| Lymphocytes | Potassium |
| Atypical lymphocytes | Sodium |
| Monocytes | Glucose |
| Neutrophils | Urea/BUN <sup>a</sup> |
| Hematocrit | Creatinine <sup>b</sup> 5 |
| Hemoglobin | Creatine kinase |
| МСН | AST |
| MCHC | ALT O |
| MCV | ALP |
| Platelet count | ĢĢT |
| RBC count | LDH |
| WBC count | Total bilirubin |
| | Direct (conjugated) bilirubin |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; GGT=gamma-glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; WBC=white blood cell

Table 11–2: Optional laboratory measurements

| Biochemistry | Urinalysis <sup>b</sup> | <b>Endocrinology</b> <sup>c</sup> |
|---|---|---|
| Total cholesterol <sup>a</sup> | Protein | TSH |
| × 7 | Bacteria | $T_4$ |
| 2018 | Glucose | |
| EN/64 | рН | |
| *0 | RBC | |
| 60 | WBC | |

RBC=red blood cell; T<sub>4</sub>=thyroxine; TSH=thyroid-stimulating hormone; WBC=white blood cell

<sup>&</sup>lt;sup>a</sup> Urea or BUN to be tested depending on the local lab's standard panel for neonates.

<sup>&</sup>lt;sup>b</sup> During the first days of life, creatinine will only be collected if the site assesses this parameter per standard of care.

<sup>&</sup>lt;sup>a</sup> Total cholesterol to be measured if this is part of the local lab's standard panel for neonates.

<sup>&</sup>lt;sup>b</sup> Urinalysis to be performed only if a urine sample was obtained for clinical purposes. A urine dipstick is acceptable.

<sup>&</sup>lt;sup>c</sup> TSH and T<sub>4</sub> to be recorded for the study only if measured for neonatal screening of congenital hypothyroidism prior to or during study participation.

#### 11.2.1 **Evaluation of PDILI**

The PDILI IMP discontinuation criteria (Food and Drug Administration [FDA], Guidance for Industry, Drug-induced liver injury, 2009) for this study are provided in Section 6.3.1, with the accompanying required follow-up investigation and monitoring detailed below. All PDILI events must be reported as an AE and reported to the study site and Sponsor within 24 hours of learning of their occurrence. Any PDILI event that leads to discontinuation must be reported as an AE of special interest (see Section 11.1.1.3) and must also be reported as an SAE see Section 11.1.1.2).

Evaluation of PDILI consists of the diagnostic testing and continued monitoring included in Table 11–3 specific tests dependent on laboratory results and corresponding symptoms) and consultation with a local hepatologist (if applicable; discussed in Section 11.2.1.1). Additional investigation and monitoring may be required and adapted based on the diagnosis after the cause of the liver injury/abnormality is confirmed (details in Section 11.2.1.4).

The results of all monitoring, including laboratory testing and other testing, should be made available to the study site and Sponsor.

waiting is and follow, and fol All initial tests resulting in abnormal hepatic laboratory values need to be repeated, but appropriate medical action must not be delayed while waiting for the repeat result.

Table 11–3 summarizes the required investigations and follow-up for PDILI.

Table 11-3: Required investigations and follow-up for PDILI

| Patient population | Laborato | ory value | Immediate | | Follow-Up | |
|---|---|---|---|---|---|---|
| | ALT/<br>AST/ALP | Direct<br>(conjuga-<br>ted)<br>bilirubin <sup>a</sup> | Consultation requirements | Actions | Testing io | Evaluation |
| Subjects<br>without<br>perinatal<br>asphyxia | ≥3xULN<br>according to<br>the subject's<br>GA and site's<br>normal value | NA | Hepatology<br>consultation<br>(see Section 11.2.1);<br>Medical Monitor<br>must be notified | Immediate, permanent IMP discontinuation. | Essential: Must have repeat liver chemistry values and additional testing completed ASAP (see Section 11.2.1.1); | Monitoring of liver<br>chemistry values at least<br>twice per week until<br>values normalize,<br>stabilize, or return to |
| Subjects<br>with<br>perinatal<br>asphyxia <sup>c</sup> | ≥5xULN<br>according to<br>the subject's<br>GA and site's<br>normal value | NA | within 24 hours (eg, laboratory alert) and subject discussed with Medical Monitor ASAP <sup>b</sup> | CCOP dion appli | recommended to occur at the site with HCP. | within Baseline values. |
| All subjects | NA | ≥2mg/dL | *ejins | | | |

ASAP=as soon as possible; GA=gestational age; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug-induced liver injury; ULN=upper limit of normal

<sup>&</sup>lt;sup>a</sup> Any requirement for phototherapy or exchange transfusion due to elevated bilirubin necessitates withdrawal regardless of laboratory values.

b Details provided in Section 11.2.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist.

<sup>°</sup> For subjects with perinatal asphyxia, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within few days after birth, and subsequent normalization until up to day 14 after birth): in case AST, ALT or ALP elevation ≥5x ULN occurs within 5 days after birth in patients with perinatal asphyxia and suspected hepatic hypoxic injury, study drug must be discontinued and LFTs retested within 24 hours. If AST, ALT and ALP values confirmed <5x ULN, the subject may restart study drug after consultation with and approval by the Medical Monitor.

### 11.2.1.1 **Consultation with Medical Monitor and local hepatologist**

Potential drug-induced liver injury events require notification of the Medical Monitor within ions or variations thereof. 24 hours, and the subject must be discussed with the Medical Monitor as soon as possible. If applicable, the subject may also be discussed with the local hepatologist. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist or neonatologist with relevant expertise. If determined necessary, this discussion should be followed by a full assessment (see Section 11.2.1.3) and SAE report (if applicable).

#### 11.2.1.2 Immediate action: determination of IMP discontinuation

All PDILI events require immediate action, testing, and monitoring.

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.3.1 and Table 11–3 for details).

When IMP is discontinued, all concomitant medications that are not medically necessary should also be discontinued. The Investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

### Testing: identification/exclusion of alternative etiology 11.2.1.3

The measurements and additional information recommended for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are detailed in Table 11–4 (laboratory measurements) and Table 11–5 (additional information). Recommended testing is at the discretion of the Investigator and should be individualized appropriately based on clinical situation.

Results of the laboratory measurements and information collected are to be submitted to the Sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other assessments not included below, these additional assessments should be completed and submitted, as applicable.

All blood samples will be tested locally.

Table 11–4 shows the PDILI laboratory measurements recommended to be assessed. This document cannot be used to

### Table 11–4: Recommended PDILI laboratory measurements<sup>a</sup>

| Virology-related (virology tests dependent on local vaccination | HSV blood PCR (or other testing: HSV IgM, viral culture of blood or CSF, CSF PCR) |
|---|---|
| schedule) | Enterovirus blood PCR (or other testing) |
| | Hepatitis A IgM antibody <sup>b</sup> |
| | Hepatitis E IgM antibody <sup>b</sup> |
| | Hepatitis C IgM <sup>b</sup> |
| | HBsAg <sup>b</sup> |
| | Cytomegalovirus testing (culture or polymerase chain reaction) of saliva/urine |
| | Epstein-Barr viral capsid antigen IgM antibody |
| Hematology | Eosinophil count Toxicology screen |
| Urinalysis | |
| Chemistry | Amylase |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| OUBL I | Lactate, pyruvate (mitochondrial screen) |
| Hejing! | Plasma acylcarnitine profile (fatty acid oxidation defects) |
| any mail | Ferritin (screen for gestational alloimmune liver disease [neonatal hemochromatosis]) |
| "Obolt or | Confirm newborn screening results (galactosemia and tyrosinemia) |
| Additional elised to support any marketing at | Serum amino acid profile (urea cycle and metabolic) |
| Additional | Prothrombin time/INR |

CPK=creatine phosphokinase; CSF=cerebrospinal fluid; HBsAg=hepatitis B virus surface antigen; HSV=herpes Recommended testing on clinical situation
Maternal viral here

Table 11 simplex virus; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PCR=polymerase chain reaction; PDILI=potential drug-induced liver injury

Maternal viral hepatitis status may be considered

Table 11–5 shows the additional PDILI information to be collected:

<sup>&</sup>lt;sup>a</sup> Recommended testing is at the discretion of the Investigator and should be individualized appropriately based

### Table 11–5: PDILI information to be collected

### New or updated information

Concomitant medications prescription with dosages and dates should be included.

Pertinent medical history, including the following:

- Relevant family history or inheritable disorders (eg, Gilbert's syndrome, alpha-1 antitrypsin deficiency)

  Pearance or worsening of clinical symptoms of hepatitis or hypersensitions.

  Slinically significant hypotension or hypersensitions.

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Results of Echocardiogram (for evaluation of potential cardiac dysfunction) and abdominal ultrasound with Doppler (vascular and anatomic), if done

ion of

Any postmortem/pathology reports

PDILI=potential drug-induced liver injury

#### 11.2.1.4 Follow-up evaluation

Potential drug-induced liver injury events require follow-up monitoring as described in Table 11–5. Monitoring should continue until liver chemistry values normalize, stabilize, or return to Baseline. Determination of stabilization is at the discretion of the Investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

### Other safety measurements 11.3

### 11.3.1 Physical and neurological examinations

Physical and neurological examinations will be performed at study timepoints described in Table 5–1 and Table 5–2 for the Exploratory and Confirmatory Cohorts, respectively; and in Table 5-3 during the BRV Extension Period and Safety Follow-Up Period for both the Exploratory and Confirmatory Cohorts. Physical and neurological examinations will be performed by a medically qualified clinician. The physical examinations will include a check for the presence of skin rash and skin hypersensitivity.

Physical and neurological assessments for subjects with HIE will also include the Sarnat scale, a classification scale for HIE with grading based on clinical presentation, EEG findings, the presence of seizures, and the duration of illness. The Sarnat grading scale comprises 6 components: alertness, muscle tone, seizures, pupils, respiration, and duration assessed together to provide 3 stages (Grade I [mild]; Grade II [moderate]; Grade III [severe]) of HIE (Sarnat and Sarnat, 1976).

Clinically significant new or worsened abnormalities must be reported as AEs.

### 11.3.2 Medical history including Apgar score

The Appar score describes the condition of the newborn infant immediately after birth (Papile, 2001) and, when properly applied, is a tool for standardized assessment. It also provides

Ine Apgar score comprises 5 components: heart rate, respiratory effort, muscle tone, reflex irritability, and color, each of which is given a score of 0, 1, or 2. The score is reported at 1 and 5 minutes after birth. The Apgar score continues to provide convenient shorthand for reporting the status of the newborn infant and the response to resuscitation (C). Practice, ACOG; American Academy of B. "
2006). 2006).

### 11.3.3 Vital signs

Vital sign measurements, including systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate (including apneas), oxygen saturation (pulse oximetry), and body temperature, should be measured at the study timepoints as described in Table 5–1 and Table 5–2 for the Exploratory and Confirmatory Cohorts, respectively; and in Table 5-3 during the BRV Extension Period and Safety Follow-Up Period for both the Exploratory and Confirmatory Cohorts.

### 11.3.4 **Biometric parameters**

Biometric parameters, including length, body weight and head circumference, will be measured at the study timepoints as described in Table 5–1 and Table 5–2 for the Exploratory and Confirmatory Cohorts, respectively; and in Table 53 during the Safety Follow-Up Period for both the Exploratory and Confirmatory Cohorts. Head circumference Baseline measurement should be taken within 7 days prior to drug administration, or at birth for subjects  $\leq$ 7 days old.

#### **N-PASS** 11.3.5

The psychometric parameters, including N-PASS, will be measured at the study timepoints as described in Table 5–1 and Table 5–2 for the Exploratory and Confirmatory Cohorts, respectively; and in Table 5-3 during the BRV Extension Period and Safety Follow-Up Period for both the Exploratory and Confirmatory Cohorts.

The N-PASS was developed as a clinically relevant tool to assess ongoing or acute pain in neonates and infants, as well as sedation levels. The 5 indicators are: (1) crying/irritability (silent cry observed in the intubated infant is scored as a cry), (2) behavior/state, (3) facial expression, (4) extremities/tone, and (5) vital signs. Points are added to the preterm infant's pain score to approximate the normal response of a full-term infant. These points were derived from the Premature Infant Pain Profile pain assessment tool (Stevens et al, 1996).

Gestational age groups are <28 weeks (3 points), 28 to 31 weeks (2 points), 32 to 35 weeks (1 point), and >35 weeks (0 points). Scores range from 0 to 13. Behavioral state as a modifier was not included in the development of N-PASS, as it was designed initially for ongoing pain assessment (Hummel et al, 2010).

#### 11.3.6 **Video-EEG Parameters**

Video-EEG monitoring performed during the Evaluation Period will be assessed for the subject's reactivity, in addition to the interpretation of the N-PASS in terms of sedation status.


### 11.3.7 HIE (Thompson score)

The Thompson score will be used to measure the severity of HIE for subjects with HIE at the timepoints described in Table 5–1 and Table 5–2 for the Exploratory and Confirmatory Cohorts, respectively.

The Thompson score is derived from 9 aspects of the neurological examination of infants with HIE: the total score ranges from 0 to 22 and the kappa coefficient is 0.87 (Thompson et al, 1997). This score allows a more precise description of infants than "mild", "moderate" or "severe" and recognizes the prognostic significance of mixed signs within these 3 categories. In normothermic infants, a maximum score >10 during the first 7 days of life predicts an abnormal outcome with 100% sensitivity and 61% specificity (Thompson et al, 1997).

# 11.3.8 Withdrawal and rebound phenomena

Withdrawal and rebound phenomena will be assessed by observing any AEs experienced by subjects following the cessation of BRV administration. These AEs will be reported by the Investigators, and any AEs relating to BRV withdrawal will be used for the analysis of withdrawal and rebound phenomena. Withdrawal and rebound phenomena, if any, will be captured from data collected at the end of BRV exposure for subjects in both the Exploratory and Confirmatory Cohorts.

### 11.3.9 Mechanical ventilation

Numbers and percentage of subjects requiring mechanical ventilation will be recorded from Baseline through the 48-hour Evaluation Period for the Exploratory Cohort and the 96-hour Evaluation Period for the Confirmatory Cohort.

Duration of mechanical ventilation will be recorded over the Evaluation Period.

# 11.3.10 Bayley Scales of Infant and Toddler Development, Third Edition

The Bayley-III scales will be used in this study. The data collected will not be used for analysis, but as the Baseline for subjects who are entering the long-term study.

The Bayley-III scales are recognized internationally as one of the most comprehensive developmental assessment instruments (Sattler and Hoge, 2006) used to examine the major facets of a young child's development (Bayley, 2006). The Bayley-III scales are a standardized, individually administered adaptive assessment that measures the developmental functioning of infants and young children from 1 month to 42 months of age (Bayley, 2006). The Bayley-III scales measure cognitive, language, motor, social-emotional, and adaptive.

The Bayley-III scales are an individually administered adaptive assessment that presents children with situations and tasks designed to produce an observable set of behavioral responses. They consist of a cognitive scale, a language composite scale with receptive and expressive language subscales, a motor composite scale with fine and gross motor subscales to be completed by the Investigator or designee, a social-emotional scale, comprising social-emotional competence, and sensory processing, and an adaptive behavior scale, which assesses the attainment of skills necessary for the development of independence, to be completed by the neonate's parent(s) or caregiver.

The Bayley-III scales will be completed before the subject enters the long-term study (at EPV 2) and again in the long-term study for subjects enrolled in countries where a validated translation of the scale is available in the local language.

The Investigator should not deviate from the protocol. However, the Investigator should take any measure necessary in deviation from or not defined by the protocol to protect clinical study subjects from any immediate hazard to their health and safety. In the taken immediately, without prior potification.

After implementation of such a measure, the Investigator must notify the Clinical Project Manager of the Sponsor within 24 hours and follow any local regulatory requirements.

### 12.2 Monitoring

Monitoring of the study will be delegated by UCB to a CRO. The CRO will monitor the study to meet the CRO's monitoring Standard Operating Procedures (SOPs), ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate.

The Investigator and his/her staff are expected to cooperate with UCB (or designee) and to be available during the monitoring visits to answer questions sufficiently and to provide any missing information. The Investigator(s)/institution(s) will permit direct access to source data/documents for study-related monitoring, audits, IEC review, and regulatory inspection(s).

The Investigator will allow UCB (or designee) to periodically review the eCRF entries against the corresponding source documents (eg, hospital and laboratory records for each study participant). Monitoring visits will provide UCB (or designee) with the opportunity to evaluate the progress of the study, verify the accuracy and completeness of eCRFs, ensure that all protocol requirements, applicable authorities' regulations, and Investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records.

#### 12.2.1 Definition of source data

All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. They should be made using some permanent form of recording (ink, typing, printing, optical disc). They should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Printouts of eCRF screens are not considered acceptable source documents.

Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records or other printouts, completed scales, quality of life questionnaires, or video, for example. Source documents should be kept in a secure, limited access area.

Apart from the VEEG, other source documents that may be computer generated and stored electronically must be printed for review by the monitor. Once printed, these copies should be signed and dated by the Investigator and become a permanent part of the subject's source


documents. The Investigator will facilitate the process for enabling the monitor to compare the content of the printout and the data stored in the computer to ensure all data are consistent.

### 12.2.2 Source data verification

Source data verification ensures accuracy and credibility of the data obtained. During monitoring visits, reported data are reviewed with regard to being accurate, complete, and verifiable from source documents (eg, subject files, recordings from automated instruments, tracings [VEEG], laboratory notes). All data reported on the eCRF should be supported by source documents, unless otherwise specified in Section 12.2.1.

## 12.3 Data handling

# 12.3.1 Case Report form completion

The Investigator is responsible for prompt reporting of accurate, complete, and legible data in the eCRFs and in all required reports.

Any change or correction to the eCRF after saving must be accompanied by a reason for the change.

Corrections made after the Investigator's review and approval (by means of a password/electronic signature) will be reapproved by the Investigator.

The Investigator should maintain a list of personnel authorized to enter data into the electronic eCRF.

Detailed instructions will be provided in the eCRF Completion Guidelines.

# 12.3.2 Database entry and reconciliation

Case Report forms/external electronic data will be entered/loaded into a validated electronic database using a clinical data management system (CDMS). Computerized data cleaning checks will be used in addition to manual review to check for discrepancies and to ensure consistency of the data. This study will be performed using remote data capture. The data are entered into the eCRFs once and are subsequently verified if the study is performed using electronic data capture.

An electronic audit trail system will be maintained within the CDMS to track all data changes in the database once the data have been saved initially into the system or electronically loaded. Regular backups of the electronic data will be performed.

# 12.3.3 Subject Screening and Enrollment log/Subject Identification Code list

The subject's screening and enrollment will be recorded in the Subject Screening and Enrollment Log.

The Investigator will keep a Subject Identification Code list. This list remains with the Investigator and is used for unambiguous identification of each subject.

The subject's consent and enrollment in the study must be recorded in the subject's medical record. These data should identify the study and document the dates of the subject's participation.

## 12.4 Termination of the study

UCB reserves the right to temporarily suspend or prematurely discontinue this study either at a single site, multiple sites, or at all sites at any time for reasons including, but not limited to, safety or ethical issues, inaccurate or incomplete data recording, noncompliance, or unsatisfactory enrollment with respect to quality or quantity.

If the study is prematurely terminated or suspended, UCB (or its representative) will inform the Investigators/institutions and the regulatory authority(ies) of the termination or suspension and the reason(s) for the termination or suspension, in accordance with applicable regulatory requirement(s). The IEC should also be informed and provided with reason(s) for the termination or suspension by the Sponsor or by the Investigator/institution, as specified by the applicable regulatory requirement(s). In addition, arrangements will be made for the return of all unused BRV and other material in accordance with UCB procedures for the study.

# 12.5 Archiving and data retention

The Investigator will maintain adequate records for the study, including eCRFs, medical records, laboratory results, Informed Consent documents, drug dispensing and disposition records, safety reports, information regarding participants who discontinued, and other pertinent data.

All essential documents are to be retained by the Investigator until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the IMP. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or by an agreement with UCB (Committee for Proprietary Medicinal Products [CPMP]/ICH/135/95, 2002 [Section 4.9.5]). The Investigator will contact UCB for authorization prior to the destruction of any study records or in the event of accidental loss or destruction of any study records. The Investigator will also notify UCB should he/she relocate or move the study-related files to a location other than that specified in the Sponsor's trial master file.

# 12.6 Audit and inspection

The Investigator will permit study-related audits mandated by UCB, after reasonable notice, and inspections by domestic or foreign regulatory authorities.

The main purposes of an audit or inspection are to confirm that the rights and well-being of the subjects enrolled have been protected, that enrolled subjects (ie, signing consent and undergoing study procedures) are appropriate for the study, and that all data relevant for the evaluation of the IMP have been processed and reported in compliance with the planned arrangements, the protocol, investigational site, and IEC SOPs, ICH-GCP, and applicable regulatory requirements.

The Investigator will provide direct access to all study documents, source records, and source data. If an inspection by a regulatory authority is announced, the Investigator will immediately inform UCB (or designee).

### 12.7 Good Clinical Practice

Noncompliance with the protocol, ICH-GCP, or local regulatory requirements by the Investigator, institution, institution staff, or designees of the Sponsor will lead to prompt action


by UCB to secure compliance. Continued noncompliance may result in the termination of the site's involvement in the study.

#### 13 **STATISTICS**

SOF Variations thereof A description of statistical methods follows and will be given in more detail in the Statistical Analysis Plan (SAP). In general, descriptive summaries will be used to present the study results overall and by cohorts (Exploratory Cohort and each individual Confirmatory Cohort).

### 13.1 **Definition of analysis sets**

Analysis sets will be defined as follows:

- The Pharmacokinetic Per-Protocol Set will consist of all subjects who provide at least 1 measurable plasma sample (with recorded sampling time) on at least 1 post-Baseline visit with documented study drug intake times. This analysis set will be used for the Exploratory Cohort and the Confirmatory Cohort(s).
- The SS will consist of all enrolled subjects who take at least 1 dose of BRV. All safety analyses will be performed on the SS for the Exploratory Cohort and the Confirmatory Cohort(s).
- The Full Analysis Set will be used for the analysis of seizure data (efficacy) and will consist of all subjects in the SS who have a minimum of 2 hours of interpretable VEEG data from both the Baseline period and the first 3 hours of the post-Baseline period after initial BRV treatment.

### General statistical considerations 13.2

Descriptive statistics, such as the mean, standard deviation, median, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, minimum value, and maximum value will be provided for quantitative variables. Counts and percentages will be provided for categorical variables. Confidence intervals (CIs) (95%) will be provided for efficacy variables, which will be described in the SAP. Key supporting data will be provided in data listings.

### 13.3 Pharmacokinetic variable analysis

The PK data, along with the safety data collected from the Exploratory Cohort and the 3 Confirmatory Cohorts, will be reviewed by the DMC. In addition, plasma concentrations of BRV and its metabolites will be monitored and subjected to interpretation on an ongoing basis. The analysis of the PK parameters for the Exploratory and Confirmatory Cohorts will include a sub-analysis for any concomitant use of hypothermia.

# **Exploratory Cohort**

Based on the plasma samples collected for the Exploratory Cohort, relevant PK parameters including AUC, C<sub>max</sub>, volume of distribution, and clearance, will be estimated using noncompartmental methods, with sub-analysis by concomitant use of hypothermia. Clinical interpretation of the tolerability of BRV, as well as plasma concentration data from the Exploratory Cohort, will be used to confirm, or adjust as needed, the maximum recommended dose for the Confirmatory Cohorts.



### 13.3.2 **Confirmatory Cohorts**

Plasma concentrations of BRV will be used as described for the PK Exploratory Cohort together

Safety analyses

All safety analyses will be presented for the SS. Descriptive summaries will be presented by cohort for AEs, SAEs, physical and neurological examination assessments, laboratory results heart rate, vital signs, body weight, and head circumference. Subject charact safety, such as cooling status variables (target low body) cooling began, duration of cooling Idea cooling in relation 1. [date and start and stop time of rewarming] and timing of rewarming in relation to first dose of BRV), the mother's use of AEDs (including BZD and opiates) at childbirth, N-PASS score, and Thompson score will also be summarized descriptively. The primary cause of seizure (eg, HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes) may also be used to categorize the safety review. EEG parameters for the assessment of sedation will also be summarized.

### Planned efficacy analyses 13.5

All efficacy parameters will be summarized descriptively.

Video-EEGs will be assessed locally by the Investigator for any medical decisions or medical interventions. Video-EEGs may also be assessed by a blinded, central reader to support Investigators if needed. The final analysis of VEEG outputs will be based solely on the assessment of a central reader. Efficacy parameters will be summarized descriptively (overall [with CIs]) by cohort. All efficacy variables will be analyzed by the primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes) and concomitant use of hypothermia, and reported for each subject using data listings.

### 13.5.1 Analysis of the secondary efficacy variables

The main secondary efficacy variable is as follows:

Proportion of responders to BRV treatment from Baseline to 3 hours after the initial BRV dose.

A BRV responder is defined as a subject who achieves the following reduction in seizure burden (ENS in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment:

At least 80% reduction in nonsevere seizure burden

(Nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in all 30-minute timespans)

### OR

At least 50% reduction in severe seizure burden

(Severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan). Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to  $\le 30$  minutes, >30 to  $\le 60$  minutes, >60 to  $\le 90$  minutes, and >90 to  $\le 120$  minutes.

For this study, an ENS is defined as an EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug.

For the Confirmatory Cohorts this means:

- For the analysis of the main secondary efficacy variable, subjects must not have used any rescue medication for the treatment of ENS during the first 3 hours after initiation of BRV treatment to be considered BRV responders.
- For the analysis of the secondary efficacy variables (other than the main secondary efficacy variable) and other efficacy variables, subjects must not have used any rescue medication for the treatment of ENS following the first 3 hours after initiation of BRV treatment to be considered BRV responders.

Additional details will be provided in the SAP.

Descriptive statistics will be presented for the following secondary efficacy variables:

- Proportion of subjects with at least 80% reduction in nonsevere seizure burden from Baseline to 3 hours after the initial BRV treatment
- Proportion of subjects with at least 50% reduction in severe seizure burden from Baseline to 3 hours after the initial BRV treatment
- Absolute reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period
- Percent reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period
- Proportion of BRV responders at the end of the 96-hour Evaluation Period
- Proportion of subjects who are seizure-free (100% reduction in seizure burden from Baseline) at 24 hours following the start of initial BRV treatment, categorized by subjects with nonsevere or severe seizure burden at Baseline
- Time to reduction in seizure burden for BRV responders (defined as the first timepoint when BRV responder criteria are met)
- Seizure freedom at the end of the Down-Titration Period (Confirmatory Cohorts only)

- Rate of at least 50% reduction in ENS frequency per hour from Baseline to the end of the 96-hour Evaluation Period
- Absolute difference in clinical seizures at the end of the 24-hour Evaluation Period from

Percent difference in clinical seizures at the end of the 24-hour Evaluation Period from
Baseline for neonates with motor seizures at the end of the 24-hour Evaluation Period from
Baseline for neonates with motor seizures at the time of inclusion

torical controls will be matched by age and condition, using comparation period from the property of the BRV will be evaluated by the property of the BRV moder rates for the time of the 24-hour Evaluation Period from the property of the BRV moder rates for the BRV moder rates for the time of the 24-hour Evaluation Period from the property of the BRV moder rates for the BRV moder Historical controls will be matched by age and condition, using comparable standard of care and diagnostic methods. The efficacy of BRV will be evaluated for the main efficacy variable by comparing the 95% CI of the BRV responder rate (with all Confirmatory Cohorts combined) to responder rates for the referenced historical control group. If the BRV lower 95% CI limit is higher than the historical control group responder rate, then BRV would be considered efficacious compared to the historical control group. If the BRV upper 95% CI limit is lower than the historical control group responder rate, then BRV will not be considered efficacious compared to the historical control group. If the BRV 95% CI limits contain the historical control group responder rates, then the results will be considered inconclusive.

### 13.5.2 Analysis of the other efficacy variables

Descriptive statistics will be presented for the other efficacy variables:

- Absolute reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
- Percentage reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
- Categorized percentage reduction from Baseline to the end of the 96-hour Evaluation Period in seizure burden <-25% [worsening], -25% to <25% [no change], 25% to <50%, 50% to <80%, and  $\ge 80\%$ )
- Proportion of BRV responders by time interval at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment
  - Proportion of subjects who are switched over from BRV to another AED during the 96-hour **Evaluation Period**
- Proportion of responders to other treatment during the 96-hour Evaluation Period (including at the end of the 96-hour Evaluation Period, and by time intervals: 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours,

>36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment

Variations thereof (A responder to other treatment is defined as at least 80% reduction in nonsevere seizure burden from start of other treatment to end of other treatment or at least 50% reduction in severe seizure burden from the initiation of other treatment to end of other treatment during the 96-hour Evaluation Period).

### 13.6 Handling of protocol deviations

Important protocol deviations are deviations from the protocol that could potentially have a meaningful impact on key PK, efficacy, or safety outcomes for an individual subject. The criteria for identifying important protocol deviations and the classification of important protocol deviations will be documented in a protocol-defined specification document. To the extent feasible, rules for identifying important protocol deviations will be defined without review of the data and without consideration of the frequency of occurrence of such deviations. Whenever possible, criteria for identifying important protocol deviations will be implemented algorithmically to ensure consistency in the classification of important protocol deviations across all subjects.

Important protocol deviations will be reviewed as part of the ongoing data cleaning process prior to database lock to confirm exclusion from analysis sets.

### Handling of dropouts or missing data 13.7

For subjects who dropped out during the Evaluation Period, the number of hours from the start of the Evaluation Period to the time of withdrawal (in hours) will be considered for analysis. Subjects in the Confirmatory Cohorts who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS during the first 3 hours after initiation of BRV treatment will be considered BRV nonresponders.

The impact of missing data on the assessment of the main secondary efficacy variable will be evaluated with sensitivity analyses with further details to be included in the SAP.

No imputation of missing values associated with an individual date or visit is planned for the safety analysis, with the exception of partial date information for AEs and concomitant medications, in order to determine whether they are treatment emergent.

### 13.8 Planned PK data review and safety data monitoring

### Exploratory Cohort 13.8.1

Upon the completion of the Exploratory Cohort, the DMC will be provided with the summaries and the listings of PK and safety data for review to make recommendations concerning the dosing of BRV in the Confirmatory Cohorts (see Section 13.8.3). During the DMC review of PK and safety data, the enrollment of subjects will be on hold.

### 13.8.2 **Confirmatory Cohorts**

At least 36 subjects will be enrolled in 3 consecutive Confirmatory Cohorts, each consisting of 12 subjects. A PK and safety data review will be performed after completion each of the cohorts. Both PK and safety summaries and data listings will be generated first for the DMC to review. In

 addition, plasma concentrations of BRV and its metabolites will be monitored and subjected to interpretation on an ongoing basis.

During the DMC review of the PK and safety data, the recruitment of subjects for the subsequent

DMC and stopping rules

The DMC will consist of 3 voting members, none of whom will be involved in the conduct of the study, either by management or participation.

The DMC will oversee the PK and safety of the study by review periodically, in order to evaluate the study by the study. The DMC study. The DMC will make recommendations regarding subject safety and continuance of the study based on the observed risk-benefit of the emerging data; however, no formal statistical stopping rules will be defined. Details will be provided in a DMC charter.

### 13.9 **Determination of sample size**

At least 42 evaluable subjects will be enrolled in this study. At least 6 subjects will be enrolled in the Exploratory Cohort and at least 36 subjects will be enrolled in 3 successive Confirmatory Cohorts, each consisting of 12 subjects. At least 2 subjects undergoing hypothermia treatment will be included in the Exploratory Cohort and each of the 3 Confirmatory Cohorts.

Subjects in the Exploratory Cohort might be replaced due to lack of data, as deemed necessary following the review of PK and safety data by the DMC.

No formal sample size calculation has been performed as a single treatment BRV arm is planned for descriptive summary of results and for comparison with the 6 subjects from the Exploratory Cohort. The total number of at least 36 subjects in the Confirmatory Cohorts is expected to provide sufficient evidence of tolerability, safety, and efficacy, as well as good precision for the PK profile of BRV in neonates.

Subjects who drop out or are withdrawn from study participation will not be replaced.

### **ETHICS AND REGULATORY REQUIREMENTS** 14

### Informed consent 14.1

The informed consent of the parent(s) or legal representative(s) for the subject must be obtained and documented in accordance with local regulations, ICH-GCP requirements, and the ethical principles that have their origin in the principles of the Declaration of Helsinki.

When a neonate with repeated EEG seizures is identified, the parent(s) or legal representative(s) will be approached and given written information about the underlying disease and a basic description of the study. This information will be discussed with the parent(s) or legal representative(s). If the parent(s) or legal representative(s) of the subject are interested in study participation, the approved ICF will be provided to them, and they will be given time to read the document. Prior to obtaining informed consent, information should be given in both oral and written form in a language and at a level of complexity understandable to the subject's parent(s) or legal representative(s), by the Investigator (or designee). The parent(s) or legal

representative(s) of each subject will have the opportunity to discuss the study and its alternatives with the Investigator.

Prior to participation in the study, the ICF must be signed and personally dated by the subject's parent(s) or legal representative(s), and by the person who conducted the informed consent discussion (Investigator or designee). The subject's parent(s) or legal representative(s) must receive a copy of the signed and dated ICF. As part of the consent process, the parent(s) or legal representative(s) of each subject must consent to direct access to the subject's medical records for study-related monitoring, auditing, IEC review, and regulatory inspection. An informed consenting process managed via telephone is allowed where applicable per local regulations.

During the Screening, Baseline, Evaluation, and BRV Extension Periods, continuous consent will be ensured by meetings between the Investigator and/or designee and the parent(s) or legal representative(s). The purpose of these meetings will be to discuss the ongoing care of the subject, as well as their continued participation in the study. Parent(s) or legal representative(s) will be informed again that they can withdraw the subject from the study at any time and that the decision will not influence the care of the subject. Continuous consent will be documented in the subjects' medical charts and eCRF. Comprehension of the study and its potential risks is enhanced by this continuous process (Allmark and Mason, 2006) and, thus, a more informed consent is obtained.

If the ICF is amended during the study, the Investigator (or the Sponsor, if applicable) must follow all applicable regulatory requirements pertaining to the approval of the amended ICF by the IEC and use of the amended form.

# 14.2 Subject identification cards

Upon signing the ICF, the subject's parent(s) or legal representative(s) will be provided with a subject identification card of his/her neonate in the language of the subject's parent(s) or legal representative(s). The Investigator will full in the subject identifying information and medical emergency contact information. The Investigator will instruct the subject's parent(s) or legal representative(s) to keep the card with him/her at all times.

# 14.3 Independent Ethics Committees

The study will be conducted under the auspices of an IEC, as defined in local regulations, ICH-GCP, and in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

The Investigator/UCB will ensure that an appropriately constituted IEC that complies with the requirements of the current ICH-GCP version or applicable country-specific regulations will be responsible for the initial and continuing review and approval of the clinical study. Prior to initiation of the study, the Investigator/UCB will forward copies of the protocol, ICF, IB, Investigator's curriculum vitae (if applicable), advertisement (if applicable), and all other subject-related documents to be used for the study to the IEC for its review and approval.

Before initiating the study, the Investigator will have written and dated full approval from the IEC responsible for the protocol.

The Investigator will also promptly report to the IEC all changes in the study, all unanticipated problems involving risks to human subjects or others, and any protocol deviations, to eliminate immediate hazards to subjects.

The Investigator will not make any changes in the study or study conduct without IEC approval, except where necessary to eliminate apparent immediate hazards to the subjects. For minor changes to a previously approved protocol during the period covered by the original approval, it may be possible for the Investigator to obtain an expedited review by the IEC as allowed.

As part of the IEC requirements for continuing review of approved studies, the Investigator will be responsible for submitting periodic progress reports to the IEC (based on IEC requirements), at intervals appropriate to the degree of subject risk involved, but no less than once per year. The Investigator should provide a final report to the IEC following study completion.

UCB (or its representative) will communicate safety information to the appropriate regulatory authorities and all active Investigators in accordance with applicable regulatory requirements. The appropriate IEC will also be informed by the Investigator or the Sponsor, as specified by the applicable regulatory requirements in each concerned country. Where applicable, Investigators are to provide the Sponsor (or its representative) with evidence of such IEC notification.

## 14.4 Subject privacy

UCB staff (or designee) will affirm and uphold the subject's confidentiality. Throughout this study, all data forwarded to UCB (or designee) will be identified only by the subject number assigned at Screening.

The Investigator agrees that representatives of UCB, its designee, representatives of the relevant IEC, or representatives of regulatory authorities will be allowed to review that portion of the subject's primary medical records that directly concerns this study (including, but not limited to, laboratory test result reports, ECG reports, admission/discharge summaries for hospital admissions occurring during a subject's study participation, and autopsy reports for deaths occurring during the study).

### 14.5 Protocol amendments

Protocol changes may affect the legal and ethical status of the study and may also affect the statistical evaluations of sample size and the likelihood of the study fulfilling its primary objective.

Significant changes to the protocol will only be made as an amendment to the protocol and must be approved by UCB, the IEC, and the regulatory authorities (if required), prior to being implemented.

# 15 FINANCE, INSURANCE, AND PUBLICATION

Insurance coverage will be handled according to local requirements.

Finance, insurance, and publication rights are addressed in the Investigator and/or CRO agreements, as applicable.

### 16 REFERENCES

Allegaert K, van den Anker J. Neonatal drug therapy: the first frontier of therapeutics for children. Clin Pharmacol Ther. 2015;98:288-97.

Allmark P, Mason S. Should desperate volunteers be included in randomised controlled trials? J Med Ethics. 2006;32:548-53.

Bayley N. Bayley Scales of Infant and Toddler Development. 3rd ed. San Antonio: Pearson Education Inc; 2006.

Boylan GB, Rennie JM, Chorley G, Pressler RM, Fox GF, Farrer K et al. Second-line anticonvulsant treatment of neonatal seizures: a video-EEG monitoring study. Neurology. 2004;62:486-8.

Boylan GB, Rennie JM, Pressler RM, Wilson G, Morton M, Binnie CD. Phenobarbitone, neonatal seizures, and video-EEG. Arch Dis Child Fetal Neonatal Ed. 2002;86:F165-70.

Castro Conde JR, Hernández Borges AA, Doménech Martínez E, González Campo C, Perera Soler R. Midazolam in neonatal seizures with no response to phenobarbital. Neurology. 2005;64:876-9.

Clancy RR, Legido A, Lewis D. Occult neonatal seizures. Epilepsia. 1988;29:256-61.

Committee on Obstetric Practice, ACOG; American Academy of Pediatrics; Committee on Fetus and Newborn, ACOG. ACOG Committee Opinion. Number 333, May 2006 (replaces No. 174, July 1996): The Agpar score. Obstet Gynecol. 2006;107:1209-12.

CPMP/ICH/135/95 Note for guidance on Good Clinical Practice (EMEA) Jul 2002.

European Union Commission ad hoc group. Recommendations of the ad hoc group for the development of implementing guidelines for Directive 2001/20/EC relating to good clinical practice in the conduct of clinical trials on medicinal products for human use. Ethical Considerations for Clinical Trials on Medicinal Products Conducted with the Paediatric Population. 2008; 13.2. https://ec.europa.eu/health/sites/health/files/files/eudralex/vol-10/ethical\_considerations\_en.pdf.

Food and Drug Administration. Guidance for Industry. Drug-induced liver injury: premarketing clinical evaluation. US Dept of Health and Human Services, Center for Drug Evaluation and Research, Center for Biologics Evaluation and Research, 07/2009.

Glass HC, Kan J, Bonifacio SL, Ferriero DM. Neonatal seizures: treatment practices among term and preterm infants. Pediatr Neurol. 2012;46:111-5.

Hummel P, Lawlor-Klean P, Weiss MG. Validity and reliability of the N-PASS assessment tool with acute pain. J Perinatol. 2010;30:474-8.

Jullien V, Pressler RM, Boylan G, Blennow M, Marlow N, Chiron C, et al. Pilot evaluation of the population pharmacokinetics of bumetanide in term newborn infants with seizures. J Clin Pharmacol. 2015;56:284-90

Leroux S, Turner MA, Barin-Le Guellec C, Hills H, van den Ankers JN, Kearns GL, et al. Pharmacokinetic Studies in Neonates: The Utility of an Opportunistic Sampling Design. Clin Pharmacokinet. 2015;54:1273–85.

Mizrahi E, Kellaway P. Characterization and classification of neonatal seizures. Neurology. 1987;37:1837-44.

O'Hara K, Wright IM, Schneider JJ, Jones AL, Martin JH. Pharmacokinetics in neonatal prescribing: evidence base, paradigms and the future. 2015;80:1281-8.

Painter MJ, Scher MS, Stein AD, Armatti S, Wang Z, Gardiner JC, et al. Phenobarbital compared with phenytoin for the treatment of neonatal seizures. N Engl J Med. 1999;341:485-9.

Papile LA. The Apgar score in the 21st century. N Engl J Med. 2001;344:519-20.

Pressler RM, Mangum B. Newly emerging therapies for neonatal seizures. Semin Fetal Neonatal Med. 2013;18:216-23

Pressler RM, Boylan GB, Marlow N, Blennow M, Chiron C, Cross JH. Bumetanide for the treatment of seizures in newborn babies with hypoxic ischaemic encephalopathy (NEMO): an open-label, dose finding, and feasibility phase 1/2 trial. Lancet Neurol. 2015;14:469-77.

Ronen GM, Penney S, Andrews W. The epidemiology of clinical neonatal seizures in Newfoundland: a population-based study. J Pediatr. 1999;134:71-5.

Sarnat HB, Sarnat MS. Neonatal encephalopathy following fetal distress. A clinical and electroencephalographic study. Arch Neurol. 1976;33:696-705.

Sattler JM, Hoge RD. Assessment of children: behavioral, social, and clinical foundations. Fifth ed. La Mesa: Jerome M Sattler; 2006.

Scher MS, Alvin J, Gaus L, Minnigh B, Painter MJ. Uncoupling of EEG-clinical neonatal seizures after antiepileptic drug use. Pediatr Neurol. 2003;28:277-80.

Slaughter L, Patel AD, Slaughter JL. Pharmacological treatment of neonatal seizures: a systematic review. J Child Neurol. 2013;28:351-64.

Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996;12:13-22.

Thompson CM, Puterman AS, Linley LL, Hann FM, van der Elst CW, Molteno CD, et al. The value of a scoring system for hypoxic ischaemic encephalopathy in predicting neurodevelopmental outcome. Acta Paediatr. 1997;86:757-61.

Tulloch JK, Carr RR, Ensom MA. A systematic review of the pharmacokinetics of antiepileptic drugs in neonates with refractory seizures. J Pediatr Pharmacol Ther. 2012;17:31-44.

van Rooij LG, van den Broek MP, Rademaker CM, de Vries LS. Clinical Management of Seizures in Newborns: diagnosis and management. Paediatr Drugs. 2013a;15:9-18.

van Rooij LG, Hellström-Westas L, de Vries LS. Treatment of neonatal seizures. Semin Fetal Neonatal Med. 2013b;18:209-15.

Wolpe J. Neurology of the newborn. Fifth ed. Philadelphia: Saunders Elsevier; 2008.

Weeke LC, Toet MC, van Rooij LG, Groenendaal F, Boylan GB, Pressler RM, et al. Lidocaine response rate in aEEG-confirmed neonatal seizures: Retrospective study of 413 full-term and preterm infants. Epilepsia. 2016;57(2):233-42.

Anates:
Anates


### 17 **APPENDICES**

#### 17.1 **Protocol Amendment 1**

### Rationale for the amendment

The primary purpose of this non-substantial amendment is to make LFT ranges specified in the exclusion and withdrawal criteria, as well as the PDILI criteria, required investigations and laboratory measurements more age specific and appropriate for the target patient population. Changes were also made to take into account feedback from investigators on the practical aspects of conducting a clinical study in the neonatal population. In addition, editorial changes were made to the text in order to clarify different aspects of the study design. Administrative changes may not be included in the summary table of changes since they are considered minor. ind any exter

# Modifications and changes

# Global changes

- Duration of BRV infusion was specified
- Condition under which BRV treatment should be stopped after a subject completed the Evaluation Period was clarified.
- The Schedule of Assessment was adapted to reflect protocol changes
- Drug dosing diary was introduced for subjects treated with oral BRV at home during the **BRV** Extension
- Duration of VEEGs performed during the Down-Titration Period was specified
- Exclusion criterion #7 was modified: AST, ALT and ALP values were specified for subjects with perinatal asphyxia
- Numbering of "may" withdrawal criteria" was changed to a consecutive numbering throughout section 6.3
- Withdrawal criterion #6 was modified: AST, ALT and ALP values were specified for subjects with perinatal asphyxia
- Withdrawal criterion #9a was modified (former "may" withdrawal criterion #3): AST, ALT and ALP values were specified for subjects with perinatal asphyxia
- PDILI criterion was aligned with updated exclusion criterion#7, withdrawal criterion #6 and withdrawal criterion #9a (former "may" withdrawal criterion #3)
- Type of syringes used to administer oral BRV during the BRV Extension Period was aligned with those used in Follow-up study N01266
- Timepoint of EPV2 was specified
- Method of PK blood sample collection was specified
- Description of AESI associated with PDILI was aligned with the updated PDILI criterion
- Reporting requirements for PDILI were clarified
- Number of DMC voting members was increased from 3 to 4 members

- \*DILI'In present of the standard of the standa

# Specific changes

| UCB<br>Clinical Study Pr | otocol | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|---|
| Specific ch | anges | | iation |
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| Sections 2.3, 5.1.1, 5.4.2, 7.2 and 8.1.3 | Intravenously administered BRV is bioequivalent to the same dosage given orally in healthy adults when given as a bolus or as a 15-minute infusion | Intravenously administered BRV is bioequivalent to the same dosage given orally in healthy adults when given as a bolus or as an approximately 15-minute infusion | Based on Investigators' feedback, the duration of infusions was adapted to clinical needs. |
| Sections<br>5.1.2, 8.2.3<br>and Footnote<br>to Table 5-2 | If subjects continue to have seizures after 96 hours of BRV administration, BRV administration will be stopped and replaced by another AED. | If subjects do not benefit from BRV treatment after 96 hours of BRV administration, BRV administration will be stopped and replaced by another AED | Condition clarified under which BRV treatment should be stopped after a subject completed the Evaluation Period. |
| Table 5-1 | MDZ infusion | Removed | MDZ treatment removed as it is not considered a study specific assessment but standard of care. |
| Tables 5-1 and 5-2 | Not applicable | Dispense BRV dosing diary | Dosing diary added to allow parents to document the dosing of BRV during the BRV Extension Period, if oral BRV is administered at home. |
| Footnote to Table 5-1 | Not applicable | The BRV dosing diary will be dispensed only if the subject enters the BRV Extension Period | Index j added for clarification of the newly inserted item "Dispense BRV dosing diary". |
| Footnote to Table 5-2 | Not applicable | The BRV dosing diary will be dispensed only if the subject enters the BRV Extension Period | Index I added for clarification of the newly inserted item "Dispense BRV dosing diary". |
| Table 5-3 | Not applicable | Review BRV dosing diary | Task added, which is part of the Investigators' drug accountability. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Table 5-3 | VEEG | 1-hour VEEG | The duration of video-EEGs recorded during Down-Titration was specified to clearly separate this assessment from the 24-hour continuous video-EEG performed during the Evaluation Period. |
| Footnote to Table 5-3 | Video-EEG will only apply to subjects of the Confirmatory Cohorts who complete the study after the Evaluation Period. | Video-EEG will only apply to subjects of the Confirmatory Cohorts who complete the study after the Evaluation Period. The video-EEG will be recorded for at least 1 hour on the final day of the Down-Titration Period. Additional video-EEGs can be performed at any time during the Down-Titration Period at the investigator's discretion. | Description of the video-EEG that will be recorded at the end of the Down-Titration Period was specified to clearly separate this assessment from the 24-hour continuous video-EEG performed during the Evaluation Period. Also, adding clarification that the protocol allows other video-EEGs to be performed during the Down-Titration Period at the discretion of the Investigator. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 6.2 | 7. Subject has 2x upper limit of normal (ULN) of any of the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP), according to the subject's GA and the site's normal range values for the respective GA. | 7a. Subject has 2x upper limit of normal (ULN) of any of the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP), with the following exception: For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable, if initial and peak elevation of liver function tests (LFTs) occurs within 5 days after birth, and the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia. The determination of ULN will be based on the subject's GA and the site's normal range values for the respective GA. | Based on Investigators' feedback, LFT values specified were modified to make them more age and indication specific. These changes are also intended to ensure a balanced enrollment of subjects, regardless of the cause/underlying disease of ENS. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 6.3 | 6. Subject has 3x ULN of any of the following: AST, ALT, and ALP, according to the subject's GA and the site's normal range values for the respective GA. | 6a. Subject has AST, ALT or ALP values 3x ULN, with the following exception: For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable for continuation in the study, if initial and peak elevation of LFTs occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within a few days after birth, and subsequent normalization until up to day 14 after birth). In case AST, ALT or ALP elevation ≥5x ULN occurs within 5 days after birth, study drug must be discontinued and LFTs retested within 24 hours. If AST, ALT and ALP are confirmed to be <5x ULN, the subject may restart study drug after consultation with and approval by the Medical Monitor. The determination of ULN will be based on the subject's GA and the site's normal range values for the respective GA. | Based on Investigators' feedback, LFT values specified in withdrawal criterion #6 were adapted in accordance with exclusion criteria changes (see Section 6.2). |

| Section<br>Impacted | Key components of previous text | K | ey components of amended text | Rationale |
|---|---|---|---|---|
| Section 6.3 | 1. Subject experiences prolongation of seizure duration, a worsening of seizure burden, or emergence of new seizure type or illness considered by the investigator to require intervention. | 7a. | Subject experiences prolongation of seizure duration, a worsening of seizure burden, or emergence of new seizure type considered by the investigator to require intervention. | Modified to delete redundant information which is covered by withdrawal criterion #8. Numbering changed to a consecutive numbering throughout section 6.3. |
| Section 6.3 | 2. Investigator may withdraw subject due to any medical condition, based on clinical judgment and discretion. | 8. | Investigator may withdraw subject due to any medical condition, based on clinical judgment and discretion. | Numbering changed to a consecutive numbering throughout section 6.3. |
| Section 6.3 | 3. The Investigator may withdraw the subject if AST/ ALT/ ALP levels are between >2x and 3x ULN, according to the subject's GA and the site's normal range values for the respective GA. | 9a. | values between >2x and ≤3x ULN, with the following exception: For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable for continuation in the study, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within a few days after birth, and subsequent normalization until up to day 14 after birth). The determinations of ULN will | Aligned with changes to exclusion criterion #7 and withdrawal criterion #6. Numbering changed to a consecutive numbering throughout section 6.3. |
| | calmot be | | be based on the subject's GA and<br>the site's normal range values for<br>the respective GA. | |
| Confidential | Jocument cannot | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 6.3 | 4. Subject has rapidly increasing total bilirubin without requiring or being expected to require phototherapy or exchange transfusion; the subject's withdrawal will be at the discretion of the Investigator. | 10. Subject has rapidly increasing total bilirubin without requiring or being expected to require phototherapy or exchange transfusion; the subject's withdrawal will be at the discretion of the Investigator. | Numbering changed to a consecutive numbering throughout section 6.3. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 6.3.1 | Subject has AST/ALT/ALP values >3x ULN according to the subject's GA and the site's normal values for that GA. | Subject has AST, ALT or ALP values >3x ULN, with the following exception: For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable for continuation in the study, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within few days after birth, and subsequent normalization until up to day 14 after birth). In case AST, ALT or ALP elevation ≥5x ULN occurs within 5 days after birth, study drug must be discontinued and LFTs retested within 24 hours. If AST, ALT and ALP are confirmed to be <5x ULN, the subject may restart study drug after consultation with and approval by the Medical Monitor. The determination of ULN will be based on the subject's GA and the site's normal range values for the respective GA. | The PDILI criterion was aligned with changes to exclusion criterion #7, withdrawal criterion #9a (former "may" withdrawal criterion #3). |
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.2 | For subjects who are switched to BRV oral solution, the dose will be measured using the appropriate syringes (1mL and 5mL) with an adaptor able to fit all the bottle sizes. | For subjects who are switched to BRV oral solution, the dose will be measured using the appropriate syringes (1mL, 3mL or 10mL) with an adaptor able to fit all the bottle sizes. | To avoid confusion and the risk of dosing errors in subjects transitioning to Follow-up study N01266, syringes used for the administration of oral BRV were aligned with those used in study N01266. |
| Section 7.3 | Brivaracetam 10mg/mL oral solution will be packaged in 300mL type-III amber glass bottles with child-resistant tamper evident polypropylene screw closures. Syringes of 1mL and 5mL will be provided with an adaptor able to fit all the bottle sizes. | Brivaracetam 10mg/mL oral solution will be packaged in 300mL type-III amber glass bottles with child-resistant tamper evident polypropylene screw closures. Syringes of 1mL, 3mL or 10mL will be provided with an adaptor able to fit all the bottle sizes. | To avoid confusion and the risk of dosing errors in subjects transitioning to Follow-up study N01266, syringes used for the administration of oral BRV were aligned with those used in study N01266. |
| Sections 7.7 and 8.1.4 | Not applicable | Hand out and return of a dosing diary<br>and documentation of drug use during<br>home administration of oral BRV<br>added to the description of the BRV<br>Extension Period (EPV1, EPV2) | Introduction of a dosing diary to facilitate parents' recording of BRV oral solution administered at home during the BRV Extension Period. Diaries will be returned to the site and reviewed by the site personnel to ensure correct use/dosing of BRV. |
| Section 7.8.2 | For the Exploratory Cohort, with the exception of MDZ as scheduled in the Protocol, if other BZDs are given prior to the first BRV administration, the subjects will be considered BRV nonresponders. | Removed | The Exploratory Cohort will not be analyzed for efficacy. For this reason it is unreasonable to classify subjects as "BRV nonresponders". |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.8.3 | For the analysis of the key efficacy variables, subjects must not have used >1 dose of rescue medication following the first 3 hours after initiation of BRV treatment to be considered BRV responders. | For the analysis of the key efficacy variables (other than the main efficacy variable) and other efficacy variables, subjects must not have used >1 dose of rescue medication following the first 3 hours after initiation of BRV treatment to be considered BRV responders. | Modified to clarify what is meant by the term "key efficacy variables". |
| Section 8.1.4 | Not applicable | In this case the parent(s) or legal representative(s) will receive a dosing diary to record the home administration of oral BRV. | Introduction of a dosing diary to facilitate parents' recording of BRV oral solution administered at home during the BRV Extension Period. Diaries will be returned to the site and reviewed by the site personnel to ensure correct use/dosing of BRV. |
| Sections 8.1.4 and 8.2.4 | Extension Period Visit 2 will be performed when the subject enters the long-term study (see Section 8.1.4.2). | Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study (see Section 8.1.4.2). | Modified to clarify that EPV2 will not only be performed if a subject transitions to the Follow-up study N01266 but on that particular day. |
| Sections<br>8.1.4.1,<br>8.1.4.2,<br>8.2.4.1 and<br>8.2.4.2 | <u> </u> | Review of BRV dosing diary (only if oral BRV is administered at home) | Introduction of a dosing diary to facilitate parents' recording of BRV oral solution administered at home during the BRV Extension Period. Diaries will be returned to the site and reviewed by the site personnel to ensure correct use/dosing of BRV. |
| Sections<br>8.1.4.3 and<br>8.2.4.3 | Not applicable Not applicable | Review of BRV dosing diary | Introduction of a dosing diary to facilitate parents' recording of BRV oral solution administered at home during the BRV Extension Period Diaries will be returned to the site and reviewed by the site personnel to ensure correct use/dosing of BRV. |
| | Deument canno | | |
| Confidential | Scn. | | |
| \his | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Sections<br>8.1.4.4 and<br>8.2.4.4 | Not applicable | Discussion of BRV dosing diary | Introduction of a dosing diary to facilitate parents' recording of BRV oral solution administered at home during the BRV Extension Period. Diaries will be discussed over the phone to ensure correct use/dosing of BRV. |
| Sections<br>8.1.4.2 and<br>8.2.4.2 | The EPV2 will be performed when the subject enters the long-term study. | The EPV2 will be performed on the same day when the subject enters the long-term study. | Modified to clarify that EPV2 will not only be performed if a subject transitions to the Follow-up study N01266 but on that particular day. |
| Section 8.2.5 | Video-EEG | At least a 1-hour video-EEG on the final day of the Down-Titration Period (during the Down-Titration Period, additional video-EEGs can be performed at the investigator's discretion) | Description of the video-EEG that will be recorded at the end of the Down-Titration Period was specified to clearly separate this assessment from the 24-hour continuous video-EEG performed during the Evaluation Period. Also, adding clarification that the protocol allows other video-EEGs to be performed in the Down-Titration Period at the discretion of the Investigator. |
| Section 9.1 | Pharmacokinetic samples will be obtained either through an existing central line or taken from routinely performed heel-pricks. | Pharmacokinetic samples will be obtained either through a venous or arterial catheter or taken from routinely performed heel-pricks. | Description of the method of blood drawing for<br>the PK analysis was specified based on<br>feedback received from investigators. The<br>former term "existing central line" was too<br>specific to cover all the different possible routes<br>of drawing blood from individual patients. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 11.1.1.3 | AST/ALT/ALP >3x ULN according to the subject's GA and the site's normal values for that GA | AST, ALT or ALP values ≥3x ULN according to the subject's GA and the site's normal values for that GA, with the following exception: | The description of AESI associated with PDILI was aligned with the PDILI criterion specified in section 6.3.1. |
| | | For subjects with perinatal asphyxia, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of the elevation of LFT is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within few days after birth, and subsequent normalization until up to day 14 after birth) only AST, ALT or ALP elevation ≥5x ULN must be reported as an AE of special interest. | and any extension |
| Figure 11-1 | Not applicable | Is the AE a PDILI event that leads to discontinuation? (see Section 11.2.1) | Information added for consistency with the change made to section 11.1.1.3 (description of AESI associated with PDILI) |
| Sections<br>11.1.6 and<br>13.8.3 | The DMC will consist of 3 voting members, none of whom will be involved in the conduct of the study, either by management or participation | The DMC will consist of 4 voting members, none of whom will be involved in the conduct of the study, either by management or participation. | The number of voting DMC members was increased to cover the medical expertise needed to assess PK and safety data for the evaluation of the risk-benefit profile in relation to the overall progress of the study. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section<br>11.2.1.1 | Potential drug-induced liver injury events require notification of the Medical Monitor within 24 hours, and the subject must be discussed with the Medical Monitor as soon as possible. If applicable, the subject must also be discussed with the local hepatologist. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. If determined necessary, this discussion should be followed by a full hepatology assessment (see Section 11.2.1.3) and SAE report (if applicable). | Potential drug-induced liver injury events require notification of the Medical Monitor within 24 hours, and the subject must be discussed with the Medical Monitor as soon as possible. If applicable, the subject may also be discussed with the local hepatologist. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist or neonatologist with relevant expertise. If determined necessary, this discussion should be followed by a full assessment (see Section 11.2.1.3) and SAE report (if applicable). | Modified based on feedback received from Investigators to better reflect the qualification of medical personnel needed and available on a local level to discuss cases of PDILI. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 11.2.1.3 | The measurements and additional information required for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are detailed in Table 11-3 (laboratory measurements) and Table 11-4 (additional information). Results of the laboratory measurements and information collected are to be submitted to the Sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other assessments not included below, these additional assessments should be completed and submitted, as applicable. All blood samples will be tested locally. Table 11-3 shows the PDILI laboratory measurements to be assessed. | The measurements and additional information recommended for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are detailed in Table 11-3 (laboratory measurements) and Table 11-4 (additional information). Results of the laboratory measurements and information collected are to be submitted to the Sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other assessments not included below, these additional assessments should be completed and submitted, as applicable. All blood samples will be tested locally. Table 11-3 shows the PDILI laboratory measurements recommended to be assessed. | Additional laboratory tests were included which cover causes of PDILI in neonates. In order to limit the extent of laboratory and other examinations to a minimum, these tests are considered as recommendations and leave it at the Investigator's discretion to decide which tests/measurements are appropriate within the given situation, taking into consideration the elinical status and medical history of subjects and their mothers. |
| Section 11.3.6 | Video-EEG monitoring will be assessed for the subject's reactivity, in addition to the interpretation of the N-PASS in terms of sedation status. | Video-EEG monitoring performed during the Evaluation Period will be assessed for the subject's reactivity, in addition to the interpretation of the N-PASS in terms of sedation status. | Description of the video-EEG assessed for the subject's reactivity was specified to clearly separate it from the 1-hour video-EEG recorded on the final day of the Down-Titration Period. |

In addition, the following intext tables were modified:

Table 11-2: Required investigations and follow-up for PDILI

| Laboratory value | | Immediate | | Follow-Up | |
|---|---|---|---|---|---|
| ALT/ AST/ALP | Conjugated<br>bilirubin <sup>a</sup> | Consultation requirements | Actions | Testing | Evaluation |
| ≥3xULN<br>according to the<br>subject's GA and<br>site's normal value | NA | Hepatology consultation. Medical Monitor must be notified within 24 hours (eg, laboratory alert) and subject | Immediate, permanent IMP discontinuation. | Essential: Must have repeat liver chemistry values and additional testing completed ASAP (see Section 11.2.1.1); recommended | Monitoring of liver<br>chemistry values at least<br>twice per week until values<br>normalize, stabilize, or |
| ≥2x and ≤3xULN<br>according to the<br>subject's GA and<br>site's normal value | ≥2mg/dL | discussed with Medical<br>Monitor ASAP <sup>b</sup> | aR <sup>A</sup> ac | to occur at the site with HCP. | return to within Baseline values. |
| NA | ≥2mg/dL | | CO Astion | | |

ASAP=as soon as possible; GA=gestational age; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug-induced liver injury; ULN=upper limit of normal

To align the investigations and follow-up for PDILI with the updated exclusion criterion #7, withdrawal criterion #6 and PDILI criterion, Table 11-2 was changed to:

a Any requirement for phototherapy or exchange transfusion due to elevated bilirubin necessitates withdrawal regardless of laboratory values.

b Details provided in Section 11.2.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist.

# Table 11-2: Required investigations and follow-up for PDILI

| Patient population | Laborato | ory value | Immediate | | Follow-Up | |
|---|---|---|---|---|---|---|
| | ALT/<br>AST/ALP | Conjugated<br>bilirubin <sup>a</sup> | Consultation requirements | Actions | Testing | Evaluation |
| Subjects<br>without<br>perinatal<br>asphyxia | ≥3xULN<br>according to<br>the subject's<br>GA and site's<br>normal value | NA | Hepatology<br>consultation (see<br>Section 11.2.1).<br>Medical Monitor<br>must be notified | Immediate, permanent IMP discontinuation. | additional testing twice per week until completed ASAP (see values normalize, stabilize, or return to | chemistry values at least<br>twice per week until<br>values normalize,<br>stabilize, or return to |
| Subjects with<br>perinatal<br>asphyxia <sup>c</sup> | ≥5xULN<br>according to<br>the subject's<br>GA and site's<br>normal value | NA | within 24 hours (eg,<br>laboratory alert) and<br>subject discussed<br>with Medical<br>Monitor ASAP <sup>b</sup> | all copy and its | recommended to occur at the site with HCP. | within Baseline values. |
| All subjects | NA | ≥2mg/dL | | 3 ithorn | | |

ASAP=as soon as possible; GA=gestational age; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug-induced liver injury; ULN=upper limit of normal

a Any requirement for phototherapy or exchange transfusion due to elevated bilirubin necessitates withdrawal regardless of laboratory values.

b Details provided in Section 11.2.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist.

<sup>&</sup>lt;sup>c</sup> For subjects with perinatal asphyxia, if initial and peak LFT elevation occurs within 5 days after birth, and if the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia (ie, peak LFT elevation within few days after birth, and subsequent normalization until up to day 14 after birth): in case AST, ALT or ALP elevation ≥5x ULN occurs within 5 days after birth in patients with perinatal asphyxia and suspected hepatic hypoxic injury, study drug must be discontinued and LFTs retested within 24 hours. If AST, ALT and ALP values confirmed <5x ULN, the subject may restart study medication after consultation with and approval by the Medical Monitor

# Table 11-3: PDILI laboratory measurements

| Virology-related | Hepatitis A IgM antibody |
|---|---|
| (virology tests dependent on local vaccination schedule) | Hepatitis E IgM antibody |
| , | Hepatitis C IgM |
| | HBsAg |
| | Cytomegalovirus testing (culture or polymerase chain reaction) of saliva/urine |
| | Epstein-Barr viral capsid antigen IgM antibody |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen |
| Chemistry | Amylase |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| Additional | Prothrombin time/INR |

Additional Prothrombin time/INR

CPK=creatine phosphokinase; HBsAg=hepatitis B virus surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury


To include additional laboratory tests which cover causes of PDILI in neonates and to limit the extent of laboratory and other examinations to a minimum, these tests are considered as recommendations and leave it at the Investigator's discretion to decide which tests/measurements are appropriate within the given situation, taking into consideration the clinical status and medical history of the subject and its mother, Table 11-3 was changed to:

Table 11-3: Recommended PDILI laboratory measurements<sup>a</sup>

| Virology-related | HSV blood PCR (or other testing: HSV IgM, viral culture of blood or CSF, CSF PCR) |
|---|---|
| (virology tests dependent on local vaccination schedule) | Enterovirus blood PCR (or other testing) |
| , | Hepatitis A IgM antibody <sup>b</sup> |
| | Hepatitis E IgM antibody <sup>b</sup> |
| | Hepatitis C IgM <sup>b</sup> |
| | HBsAg <sup>b</sup> |
| | Cytomegalovirus testing (culture or polymerase chain reaction) of saliva/urine |
| | Epstein-Barr viral capsid antigen IgM antibody |
| Hematology | Eosinophil count BL HI |
| Urinalysis | Toxicology screen |
| Chemistry | Amylase |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| | Lactate, pyruvate (mitochondrial screen) |
| | Plasma acylcarnitine profile (fatty acid oxidation defects) |
| | Ferritin (screen for gestational alloimmune liver disease [neonatal hemochromatosis]) |
| Confirm newborn screening results (galactosemia and tyrosinemia) | |
| | Serum amino acid profile (urea cycle and metabolic) |
| Additional | Prothrombin time/INR |

# Table 11-3: Recommended PDILI laboratory measurements<sup>a</sup>

CPK=creatine phosphokinase; CSF=cerebrospinal fluid; HBsAg=hepatitis B virus surface antigen; HSV=herpes simplex virus; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PCR=polymerase chain reaction; PDILI=potential drug-induced liver injury

- <sup>a</sup> Recommended testing is at the discretion of the Investigator and should be individualized appropriately based on clinical situation
- <sup>b</sup> Maternal viral hepatitis status may be considered


#### Table 11-4: PDILI information to be collected

#### New or updated information

Concomitant medications prescription with dosages and dates should be included.

Pertinent medical history, including the following:

- Adverse reactions to drugs
- Allergies
- Relevant family history or inheritable disorders (eg, Gilbert's syndrome, alpha-1 antitrypsin deficiency)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Any postmortem/pathology reports

PDILI=potential drug-induced liver injury

on in case of It copy and the used to support any marketing authorization and the used to support any marketing authorization. For the evaluation of potential cardiac dysfunction in case of PDILI, Table 11-4 was changed to

#### Table 11-4: PDILI information to be collected

#### New or updated information

Concomitant medications prescription with dosages and dates should be included.

Pertinent medical history, including the following:

- Adverse reactions to drugs
- Allergies
- Relevant family history or inheritable disorders (eg, Gilbert's syndrome, alpha-1 antitrypsin deficiency)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

This document cannot be used to support any marketing authorization applies. Results of Echocardiogram (for evaluation of potential cardiac dysfunction) and abdominal ultrasound with

#### 17.2 **Protocol Amendment 2**

#### Rationale for the amendment

ions of variations thereof The primary purpose of this non-substantial amendment is to adapt the definition of the subjects' age at enrollment based on a request from the European Medicines Agency's (EMA) Paediatric Committee (PDCO). In addition, editorial changes were made to clarify different aspects of the study design. Administrative and stylistic changes may not be included in the summary table of specific changes since they are considered minor.

Brivaracetam

## **Modifications and changes**

# Global changes

- The definition of the subjects' age at enrollment was adapted to a request from PDCO
- MDZ treatment in the Exploratory Cohort during the 3-hour interval prior to start of BRV treatment was clarified
- Timepoints for the dispense of BRV for subjects entering the BRV Extension Period were
- Timepoints for the collection of PK samples were specified
- Number of DMC voting members was decreased from 4 to 3 members
- Sections referring to Monitoring and Source Data were aligned with the updated UCB protocol template
- Parific Parific Support any managing the used to support any manager than the used to support and the used to support any manager than the used to support any Sections referring to the treatment with Permitted/Prohibited Concomitant Medication and Rescue Medication were edited for clarification

# Specific changes

| UCB<br>Clinical Study Pr | otocol | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|---|
| Specific ch | anges | | idio |
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| Sections<br>1, 2.3, 5.4.1,<br>6.1 | Subject is male or female, with an age at birth of at least 34 weeks of GA and up to 28 days of postnatal age at the time of enrollment. | Subject is male or female, with an age at birth of 34 weeks to less than 42 weeks of GA and up to 28 days of postnatal age at the time of enrollment. | The definition of the subject age at enrollment was adapted based on a request from PDCO. |
| Sections<br>1, 5.1, 7.2 | For the Exploratory Cohort (first step), enrolled subjects will receive a therapeutic dose of MDZ (dose of MDZ is at the discretion of the Investigator) prior to receiving BRV. | For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple therapeutic doses of MDZ (dose of MDZ is at the discretion of the Investigator) prior to receiving BRV. | Edited to clarify that MDZ treatment in the Exploratory Cohort during the 3 hours prior to the start of BRV treatment is not limited to a single MDZ dose. |
| Section 5.1.1 | Evaluation Period (in total, 51 hours: 3 hours for the evaluation of MDZ and 48 hours for the evaluation of BRV): Subjects will receive iv MDZ at a therapeutic dose (MDZ dose is at the discretion of the Investigator). | Evaluation Period (in total, 51 hours: 3 hours for the evaluation of MDZ and 48 hours for the evaluation of BRV): Subjects will receive iv MDZ (one or multiple therapeutic doses; MDZ dose is at the discretion of the Investigator). | Aligned with the change described above. |
| Section 4.2.1 | The use of rescue medication will affect the analysis of the key efficacy variables in the different study Cohorts (see Section 7.8.3). | The use of rescue medication will affect the analysis of the key efficacy variables in the different study Cohorts (see Section 13.5.1). | Reference to section 7.8.3 adjusted to the shift of text. |
| Table 5-1 | Not applicable | Dispense BRV for the BRV<br>Extension Period <sup>k</sup> | Row added to indicate BRV dispense at the end of the Evaluation Period (after 48 hours). |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Table 5-1 | Not applicable | k Dispensing of BRV is only applicable if the subject enters the BRV Extension Period | Footnote k added to further explain the addition of BRV dispensing at the end of the Evaluation Period. |
| Table 5-2 | Not applicable | Dispense BRV for the BRV<br>Extension Period <sup>m</sup> | Row added to indicate BRV is dispensed at the end of the Evaluation Period (after 96 hours). |
| Table 5-2 | Not applicable | m Dispensing of BRV is only applicable if the subject enters the BRV Extension Period | Footnote m added to further explain the addition of BRV dispensing at the end of the Evaluation Period. |
| Table 5-2 | b If subjects do not benefit from BRV treatment after 96 hours of BRV administration, BRV administration will be stopped and replaced by another AED; however, the subject's participation in the Evaluation Period will continue. | b If subjects do not benefit from BRV treatment after 96 hours of BRV administration, BRV administration will be stopped and replaced by another AED; however, the subject's participation in the study will continue. | In the Confirmatory Cohort all subjects will complete the Evaluation Period after 96 hours. Subjects who do not benefit from BRV at this point will enter the Down-Titration and Safety Follow-up Period. The subject's participation in the "study" will hence continue. |
| Table 5-3 | g If the subject enters the long-term study, no medication from N01349 will be dispensed in EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration | g If the subject enters the long-term study, no study drug from N01349 will be dispensed in EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration (only applicable to subjects from the Confirmatory Cohorts). | Footnote g aligned with modifications to sections 8.1.4.2 and 8.2.4.2. |
| Figure 5-4 | <sup>a</sup> Switching to another AED or addition of rescue medication is | <sup>a</sup> Switching to another AED or addition of rescue medication | Footnote a aligned with modifications to section 7.8.3. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | only permitted 3 hours after the first BRV administration. | should only occur following 3 hours after the first BRV administration. | ensions of |
| Section 7.8.1 | Prior to BRV administration, the following AEDs are permitted during the study: • PB • MDZ (Exploratory Cohort only) For the Exploratory Cohort, subjects will be permitted to receive any concomitant medications at any time during the study after BRV administration as deemed necessary by the Investigator. For the Confirmatory Cohorts, subjects will be permitted to receive AEDs only 3 hours following the first BRV administration. Other concomitant medications will be permitted as deemed necessary by the Investigator. | Concomitant treatment with non-AEDs is permitted for the Exploratory and Confirmatory Cohort(s) at any time throughout the study. Concomitant treatment with AEDs is permitted as follows: Prior to first BRV administration: PB MDZ (Exploratory Cohort only) After first BRV administration: Any AEDs (including MDZ) Exploratory Cohort: from first BRV administration Confirmatory Cohorts: from 3 hours following first BRV administration | Simplified to clarify 1) the concomitant treatment with non-AEDs and AEDs and 2) the treatment of concomitant AEDs relative to the first administration of BRV. |
| Section 7.8.2 | For the Confirmatory Cohorts only, subjects will not be permitted to receive treatments for neonatal seizures (other than the specified PB doses) prior to and for the first 3 | For the Exploratory Cohort, subjects will not be permitted to receive treatments for neonatal seizures (other than the specified PB doses and MDZ) prior to the first BRV administration. | Description of prohibited concomitant treatment in the Exploratory Cohort added for clarification. |

Confidential Hochmer


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | hours after the first BRV administration. | For the Confirmatory Cohorts, subjects will not be permitted to receive treatments for neonatal seizures (other than the specified PB doses) prior to and for the first 3 hours after the first BRV administration. | and any extensions of via |
| Section 7.8.3 | Rescue medication can be given at any time if considered necessary by the Investigator. However, it is prohibited for subjects to receive rescue medication prior to BRV dosing for the Exploratory Cohort (except for MDZ as scheduled in the Protocol) and during the 3 hours after the initial dose of BRV for the Confirmatory Cohorts. If this occurs, subjects will be considered BRV nonresponders. For the Confirmatory Cohorts this means: • For the analysis of the main efficacy variable, subjects must not have used any rescue medication (including BZDs) during the first 3 hours after initiation of BRV treatment to be considered BRV responders. | Rescue medication in this study is considered as any treatment with AEDs. Rescue medication can be given at any time if considered necessary by the Investigator. However, during the Evaluation Period rescue medication should not be administered—if possible—in the following time frames: Prior to BRV dosing for the Exploratory Cohort (except for MDZ as scheduled in the Protocol). During the first 3 hours after the initial dose of BRV for the Confirmatory Cohorts. If this occurs, subjects will be considered BRV nonresponders. | Edited for clarification. Text about the analysis of the main efficacy variable and key efficacy variables was moved to section 13.5.1 (Analysis of the key efficacy variables). |
| Confidential | Schuent | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | • For the analysis of the key efficacy variables (other than the main efficacy variable) and other efficacy variables, subjects must not have used >1 dose of rescue medication following the first 3 hours after initiation of BRV treatment to be considered BRV responders. A single dose of short-acting BZD as rescue medication is allowed, but only after 3 hours subsequent to the initiation of treatment with BRV. | COP tion application | and any extensions of varia |
| Sections<br>8.1.4 and<br>8.2.4 | Not applicable | For subjects entering the BRV Extension Period, study drug will be dispensed at the end of the Evaluation Period. | Added in conjunction with above described changes to Tables 5-1 and 5-2. |
| Sections<br>8.1.4.2 and<br>8.2.4.2 | BRV administration/dispense (If the subject enters the long-term study, no medication from N01349 will be dispensed in EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration). | BRV administration/dispense. If the subject enters the long-term study, no study drug from N01349 will be dispensed at EPV2. If the subject does not enter the long-term study, BRV from N01349 will be administered for down-titration (only applicable to subjects from the Confirmatory Cohorts). | Edited for clarification. |

| Section H<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| come coordinate coordi | or the determination of plasma oncentrations of BRV, BRV betabolites, and plasma oncentrations of concomitant AEDs PB and PHT), up to 6 blood dicrosamples (65µL/sample) will be ollected per subject in the exploratory (3 to 6 blood dicrosamples) and Confirmatory ohorts (up to 6 blood dicrosamples) at 3 predetermined dicrosamples) at 3 predetermined dicrosamples will be obtained either through a venous or deterial catheter or taken from outinely performed heel-pricks. Glood for PK samples should be die BRV infusion. Three PK samples of blood will be collected at the oblowing predetermined timepoints of the first day of the Evaluation deriod: 30 to 60 minutes, 2 to hours, and 8 to 12 hours after the lart of the most recent BRV offusion. For the Exploratory Cohort design is the first day of the 48-hour valuation Period. For the | For the determination of plasma concentrations of BRV and BRV metabolites, up to 6 blood microsamples (65µL/sample) will be collected per subject in the Exploratory (3 to 6 blood microsamples) and Confirmatory Cohorts (up to 6 blood microsamples) at 3 predetermined timepoints per day. An additional microsample (65µL) will be collected per subject for the determination of plasma concentrations of concomitant AEDs (PB and PHT). Pharmacokinetic samples will be obtained either through a venous or arterial catheter or taken from routinely performed heel-pricks. Blood for PK samples should be drawn from a line different to that of the BRV infusion. Three BRV PK samples of blood will be collected at the following predetermined timepoints at the first day of the Evaluation Period: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. For the Exploratory Cohort the same timepoints apply to the | and any extensions |

| 11.1.1.2.1 expected SAEs in babies with HIE: anticipated SAEs in babies with HIE: SAEs listed are anticipated to occur in b | Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|---|
| 11.1.1.2.1 expected SAEs in babies with HIE: anticipated SAEs in babies with HIE: SAEs listed are anticipated to occur in b | | at the same timepoints on 1 of the other days of the 96-hour Evaluation Period. It will be acceptable if these samples are drawn on different days. The timepoints for the collection of PK samples are described in Table 5–4 for the Exploratory Cohort and in Table 5–5 for the Confirmatory Cohorts. An additional microsample (65µL) will be collected for the determination of plasma concentrations of concomitant AEDs (PB and PHT). The AED PK sample should be collected 3 hours after the start of the | collected 3 hours after the start of the initial BRV administration. The timepoints for the collection of PK samples are described in Table 5–4 for the Exploratory Cohort and in Table 5–5 for the Confirmatory | and any extensions of v |
| With The macponain of enposare to be | | _ | | The term describing SAEs was clarified since SAEs listed are anticipated to occur in babies with HIE independent of exposure to BRV. |
| 11.1.6 and members, none of whom will be involved in the conduct of the study, either by management or participation. members, none of whom will be involved in the conduct of the study, either by management or participation. members, none of whom will be involved in the conduct of the study, either by management or participation. 4 voting DMC members will be supported to voting DMC members. Hence, the number voting DMC members was corrected. Single or statement of the study, either by management or participation. 3 voting DMC members are health | 11.1.6 and 13.8.3 | members, none of whom will be involved in the conduct of the study, | members, none of whom will be involved in the conduct of the study, either by management or | professionals, the medical expertise covered by |

| Section | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Impacted Section 12.2 | UCB (or designee) will monitor the study to meet the Sponsor's monitoring SOPs, ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. Monitoring of the study may be delegated by UCB to a contract research organization (CRO) or a contract monitor. | Monitoring of the study will be delegated by UCB to a CRO. The CRO will monitor the study to meet the CRO's monitoring Standard Operating Procedures (SOPs), ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. | Aligned with the updated UCB protocol template. |
| Section 12.2.1 | Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records or other printouts, completed scales, or quality of life questionnaires, for example. Source documents should be kept in a secure, limited access area. | Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records or other printouts, completed scales, quality of life questionnaires, or video, for example. Source documents should be kept in a secure, limited access area. | Aligned with the updated UCB protocol template. |
| Section 13.5.1 | Not applicable Scument cannot be used to suffer a suffer to suffe | For the Confirmatory Cohorts this means: • For the analysis of the main efficacy variable, subjects must not have used any rescue medication (including BZDs) | Moved from section 7.8.3. |
| Confidential | CHUBUT | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | during the first 3 hours after initiation of BRV treatment to be considered BRV responders. • For the analysis of the key efficacy variables (other than the main efficacy variable) and other efficacy variables, subjects must not have used >1 dose of rescue medication following the first 3 hours after initiation of BRV treatment to be considered BRV responders. A single dose of short-acting BZD as rescue medication is allowed, but only after 3 hours subsequent to the initiation of treatment with BRV. | and any extensions of the |
| Figure 11-1 | Does the AE meet any of the following? • Potentially related to BRV (see Section 11.1.1.2.1) | Does the AE meet any of the following? • Potentially related to BRV | Reference deleted since AEs described in section 11.1.1.2.1 are observed in babies and in babies with HIE regardless of study drug exposure. |

### Table 5-4: Schedule for PK Sampling (Exploratory Cohort) Table

| Assessment | MDZ | | 48-hour Evaluation Period | | | | |
|---|---|---|---|---|---|---|---|
| | | Time relat | Time relative to the start of the latest BRV infusion given per day | | | | |
| | | | Day 1 <sup>a</sup> | | Day 2 <sup>ab</sup> | | |
| | | 30-60min <sup>c</sup> | 2-4h | 8-12h | 30-60min | 2-4h | 8-12h |
| BRV PK samples <sup>d</sup> | | X | X | X | X | X | XIIIO |
| AED PK sample | | | Xe | | | C | o's |

AED=antiepileptic drug; BRV=brivaracetam; h=hours; MDZ=midazolam; min=minutes; PK=pharmacokinetic(s) Note: Blood for PK samples should be drawn from a line different to that of the BRV infusion.

- <sup>a</sup> Blood sample collection 8-12 hours is relative to BRV dosing only if BRV is administered once per day. In case of a second BRV dose on the same day, the third blood sample should be collected 30 to 60 minutes after the start of the second BRV infusion.
- <sup>b</sup> Blood sampling is only needed on Day 2 if subjects are dosed with BRV on Day 2.
- <sup>c</sup> The PK sample should be collected 30 to 60 minutes after the start of the BRV infusion.
- <sup>d</sup> The PK sampling timepoints for the first 3 samples of the Exploratory Cohorts are as follows: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. The second set of 3 samples will be collected at the same timepoints on the second day of the 48-hour Evaluation Period.
- <sup>e</sup> The AED PK sample should be collected 3 hours after the start of the initial BRV administration.

For clarification of timepoints at which PK blood samples will be collected in the Exploratory Cohort, Table 5-4 was changed to

Table 5-4: Schedule for PK Sampling (Exploratory Cohort)

| Assessment | | 48-hour Evaluation Period | | | | |
|---|---|---|---|---|---|---|
| | Time | Time relative to the start of the most recent BRV infusion | | | | |
| | , 4 | Day 1 | | Day 2ª | | |
| | 30-60min | 2-4h | 8-12h | 30-60min | 2-4h | 8-12h |
| BRV PK samples <sup>c</sup> | N. | X | X | X | X | X |
| AED PK sample | SNK. | X <sup>d</sup> | | | | |

AED=antiepileptic drug; BRV=brivaracetam; h=hours; MDZ=midazolam; min=minutes; PK=pharmacokinetic(s) Note: Blood for PK samples should be drawn from a line different to that of the BRV infusion.

<sup>&</sup>lt;sup>a</sup> Blood sampling is only needed on Day 2 if subjects are dosed with BRV on Day 2.

<sup>&</sup>lt;sup>b</sup> The first PK sample should be collected 30 to 60 minutes after the start of the BRV infusion.

<sup>&</sup>lt;sup>c</sup> The BRV PK sampling timepoints for the first 3 samples of the Exploratory Cohorts are as follows: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. The second set of 3 samples will be collected at the same timepoints on the second day of the 48-hour Evaluation Period.

d The AED PK sample should be collected 3 hours after the start of the initial BRV administration.

### Table 5-5: Schedule for PK Sampling (Confirmatory Cohorts)

| Assessment | | 96-hour Evaluation Period | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Time relative to the start of the latest BRV infusion given per day | | | | | | | | | | |
| | Da | ay 1 <sup>a</sup> | | D | ay 2ª | | D | ay 3 <sup>a</sup> | | D | ay 4ª | |
| | 30-60mi<br>n° | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h |
| BRV PK samp<br>les <sup>b</sup> | X | X | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| AED PK sample | | X <sup>d</sup> | | | | | | | | | JONS | |

AED=antiepileptic drug; BRV=brivaracetam; h=hours; PK=pharmacokinetic(s); min=minutes; (X)=optional for that day

Note: Blood for PK samples should be drawn from a line different to that of the BRV infusion.

- <sup>a</sup> Blood sample collection 8-12 hours is relative to BRV dosing only if BRV is administered once per day. In case of a second BRV dose on the same day, the third blood sample should be collected 30 to 60 minutes after the start of the second BRV infusion.
- b The PK sampling timepoints for the first 3 samples of the Confirmatory Cohorts are as follows: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. The second set of 3 PK samples will be collected within the same timeframes as the first set on one of the following days: either Day 2 (post-24 hours), OR Day 3 (post-48 hours) OR Day 4 (post-72 hours). It is acceptable if these samples are drawn on different days.
- <sup>c</sup> The first PK sample will be collected 30 to 60 minutes after the start of the BRV infusion.

For clarification of timepoints at which PK blood samples should be collected in the Confirmatory Cohorts, Table 5-5 was changed to

<sup>&</sup>lt;sup>d</sup> The AED PK sample should be collected 3 hours after the start of the initial BRV administration.

#### **Table 5-5:** Schedule for PK Sampling (Confirmatory Cohorts)

| Assessment | | 96-hour Evaluation Period | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Time relative to the start of the most recent Bl | | | | | | | | | | |
| | D | Day 1 Day 2 Day 3 | | | Day 2 | | | | D | ay 4 | | |
| | 30-60mi<br>n <sup>a</sup> | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h | 30-60m<br>in | 2-4<br>h | 8-12<br>h |
| BRV PK samp<br>les <sup>b</sup> | X | X | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| AED PK sample | | Xc | | | | | | | | | JONS | |

AED=antiepileptic drug; BRV=brivaracetam; h=hours; PK=pharmacokinetic(s); min=minutes; (X)=optional for that day

Note: Blood for PK samples should be drawn from a line different to that of the BRV infusion.

<sup>&</sup>lt;sup>a</sup> The first PK sample will be collected 30 to 60 minutes after the start of the BRV infusion.

<sup>&</sup>lt;sup>b</sup> The BRV PK sampling timepoints for the first 3 samples of the Confirmatory Cohorts are as follows: 30 to 60 minutes, 2 to 4 hours, and 8 to 12 hours after the start of the most recent BRV infusion. The second set of the 1 + (post-7)

If the start of the start 3 PK samples will be collected within the same timeframes as the first set on one of the following days: either Day 2 (post-24 hours), OR Day 3 (post-48 hours) OR Day 4 (post-72hours). It is acceptable if these samples are

<sup>°</sup> The AED PK sample should be collected 3 hours after the start of the initial BRV administration.

#### 17.3 Protocol Amendment 3

#### Rationale for the amendment

The primary purpose of this non-substantial amendment is to incorporate feedback and clarification based on IEC and Investigator requests. Administrative and stylistic changes may not be included in the summary table of specific changes since they are considered minor.

# **Modifications and changes**

## Global changes

- Modification of safety lab panel
- Alignment of language presented in the Pediatric Investigation Plan
- Safety labs from third parties considered as medical history
- Clarification of timepoints for weight measurements
- Alignment of ALP measurement
- Definition of BRV nonresponders
- Use of VEEG traces recorded before parents consented for the determination of the Baseline VEEG
- Continuous VEEG to be allowed interruption
- PB treatment permitted to start prior to the subject's admission into the study site, as well as allowed to be administered in 3 separate doses
- Recommendations for subjects discontinuing BRV treatment
- Blood sampling guidance
- Adverse event recording clarification
- Allowance of telephone consenting process
- Clarification about the transition from N01349 to follow-up study N01266
- Change in serious adverse event contact information
- Dosing and data modeling clarification

  This document cannot be

  This document.

# Specific changes

| UCB<br>Clinical Study Pro | otocol | Brivaracetam | 24 May 202<br>N0134 |
|---|---|---|---|
| Specific ch | anges | | idio |
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| STUDY<br>CONTACT<br>INFORMAT-<br>ION | 8010 Arco Corporate Drive, Raleigh, NC 27617 | UCB BioSciences, Inc.<br>8010 Arco Corporate Drive,<br>Raleigh, NC 27617 | The clinical trial biostatistician has changed. |
| STUDY<br>CONTACT<br>INFORMA-<br>TION | Neonatal Neurologist | Pediatric Neonatologist | A member of the DMC has changed. |
| SERIOUS<br>ADVERSE<br>EVENT<br>REPORTING | Europe: +32 2 386 24 21 DS_ICT@ucb.com | Europe: +32 238 66561 PSRapidalert@ucb.com | Change in serious adverse event contact information. |
| Section 1 | As the patient population of neonates with electroencephalographic neonatal seizures (ENS) is limited, N01349 is designed with a 2-step approach to allow for confirmation (or adjustment) of dosing based on results from the first step (Exploratory Cohort) and evaluation of BRV efficacy in the second step (Confirmatory Cohorts). | As the patient population of neonates with electroencephalographic neonatal seizures (ENS) is limited, N01349 is designed with a 2-step approach to allow for confirmation (or adjustment) of BRV dosing based on results from the first step (Exploratory Cohort) and evaluation of BRV efficacy in the second step (Confirmatory Cohorts). | Specification of drug dosing. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 1 | Subjects will first receive 1 or 2 doses of phenobarbital (PB) (total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion). | Subjects will first receive 1 to 3 doses of phenobarbital (PB) (total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion). | Based on Investigator feedback, the total PB dose of 20 to 40mg/kg may be administered over 3 separate doses. |
| Section 1 | For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple doses of a therapeutic dose of midazolam (MDZ) (dose of MDZ is at the discretion of the Investigator) prior to receiving BRV. | For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple doses or continuous infusion of a therapeutic dose of midazolam (MDZ) (dose and dosing frequency of MDZ are at the discretion of the Investigator) prior to receiving BRV. | Dose frequency and continuous infusion are also at the discretion of the Investigator. |
| Section 1 | This treatment represents the first use of BRV in neonates (0.5mg/kg bid), which is 4-fold less than the highest dosage of 4mg/kg/day that has been used previously in study N01263 (subjects ≥1 month old to | This treatment represents the first use of BRV in neonates (0.5mg/kg bid), which is 4-fold less than the highest dosage of 4mg/kg/day that has been used previously in study N01263 (Section 2.2). | Age specification not needed. Data modeling details added. |
| | <16 years of age; Section 2.2). | In BRV PK modeling studies CL0187 and N01331, PK profiles were extrapolated allometrically to the neonatal age group from the pediatric data collected in N01263 (age range of ≥1 month to <16 years). A total of 600 samples from 96 subjects were used for this modeling. The results of | |
| Confidential | Hochineti canno | this modeling suggest that a dosing | |
| This | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Impacted | | regimen of 2mg/kg bid in pediatric subjects ≥1 month to <16 years of age with a maximum of 100mg bid would result in plasma concentration profiles similar to those attained in older children and adults who received therapeutic doses of BRV (up to 100mg bid). Since extrapolation of data from subjects ≥1 month to subjects ≤2 weeks may be imprecise due to variability in ontogeny in the metabolic and excretory functions in neonates, actual PK measurements conducted in the Exploratory Cohort of N01349 will be used to confirm the relationship between dose and plasma concentration in neonates. | and any extensions of valid |
| Section 1 | The iv dose and dosing frequency of BRV selected for the Confirmatory Cohorts will be determined by the evaluation of BRV plasma concentrations from the Exploratory Cohort to be within the range of plasma concentrations observed in children ≥1 month old who received BRV 4mg/kg/day. | The iv dose and dosing frequency of BRV selected for the Confirmatory Cohorts will be determined by the evaluation of BRV plasma concentrations from the Exploratory Cohort, as well as by the PK modeling of N01263 data described above, to be within the range of plasma concentrations observed in children ≥1 month old who received BRV 4mg/kg/day. | Per agency recommendation, clarification that BRV dose and dosing frequency is also determined by previous PK modeling of N01263 data. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Sections 1, 5.1, 5.4.2 | Not applicable | The recommendation to confirm or adjust the originally calculated BRV dose of the Confirmatory Cohorts of study N01349 will be given by the DMC after review of PK and safety data of the Exploratory Cohort. | Clarification of DMC participation in determination of Confirmatory Cohort dosage. |
| Sections 1,<br>4.2.1, 10.1,<br>13.5.1 | Not applicable | Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to ≤30 minutes, >30 to ≤60 minutes, >60 to ≤90 minutes, and >90 to ≤120 minutes. | Clarification of 30-minute time intervals. |
| Section 4.2.1 | Absolute reduction and proportion of clinical seizures correlated with continuous VEEG from Baseline to the end of the 96-hour Evaluation Period, and each of the 3-hour intervals | Absolute and percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion | Alignment of language presented in the Pediatric Investigation Plan. |
| Section 4.3 | <ul> <li>Mechanical ventilation: <ul> <li>Number and percentage of subjects requiring ventilation during treatment with BRV over the Evaluation Period</li> <li>Number and percentage of subjects requiring ventilation during treatment with other</li> </ul> </li> </ul> | <ul> <li>Mechanical ventilation: <ul> <li>Number and percentage of subjects requiring mechanical ventilation during the Evaluation Period</li> <li>Duration of mechanical ventilation during the Evaluation Period</li> </ul> </li> </ul> | Alignment of language presented in the Pediatric Investigation Plan. |
| Confidential | Number and percentage of subjects requiring ventilation during treatment with other | | |

| | AEDs over the Evaluation | | 121 |
|---|---|---|---|
| | Period | | . Ors of |
| | <ul> <li>Absolute and relative duration of ventilation during the treatment with BRV</li> </ul> | | and any extensions of variations of variatio |
| | <ul> <li>Absolute and relative<br/>duration of ventilation<br/>during the treatment with<br/>other AEDs</li> </ul> | poplication | and |
| Section 5.1 | For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple therapeutic doses of MDZ (dose of MDZ is at the discretion of the Investigator) prior to receiving BRV. | For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple therapeutic doses or continuous infusion of MDZ (dose and dosing frequency of MDZ are at the discretion of the Investigator) prior to receiving BRV. | Dose frequency and continuous infusion are also at the discretion of the Investigator. |
| Section 5.1 | The iv dose of BRV selected for the Confirmatory Cohorts will be determined by the evaluation of BRV plasma concentrations from the Exploratory Cohort to be within the range of plasma concentrations observed in children ≥1 month old who received 4mg/kg/day. | The iv dose of BRV selected for the Confirmatory Cohorts will be determined by the evaluation of BRV plasma concentrations from the Exploratory Cohort, as well as by previous PK modeling of N01263 data, to be within the range of plasma concentrations observed in children ≥1 month old who received 4mg/kg/day. | Per agency recommendation, clarification that BRV dose and dosing frequency is also determined by previous PK modeling of N01263 data. |
| | Merit Co. | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1 | Not applicable | The recommendation to confirm or adjust the originally calculated BRV dose of the Confirmatory Cohorts of study N01349 will be given by the DMC after review of PK and safety data of the Exploratory Cohort. | Clarification of DMC participation in determination of Confirmatory Cohort dosage. |
| Section 5.1 | Not applicable Not applicable | Blood samples for routine assay of hematology, biochemistry, liver enzymes, and endocrinology will be collected in line with Section 13.2 of the "Ethical Considerations for Clinical Trials on Medicinal Products Conducted with the Paediatric Population" (European Union Commission ad hoc group, 2008), and according to the schedule of study assessments in Table 5-1 (Exploratory Cohort) and Table 5-2 (Confirmatory Cohorts). The local laboratories will perform the routine analysis of blood samples. For Screening and determination of eligibility, use of laboratory data acquired prior to Screening per standard of care inside or outside the study site within 36 hours prior to the start of the Evaluation Period is allowed. | Movement of text from Section 5.1.2 to Section 5.1, since information applied to both cohorts. Blood sampling guidance. Laboratory assessments are allowed to be administered at a separate site. Allowance of use of standard of care laboratory data. |
| This | , and the second | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1 | Not applicable | Paragraphs 17 to 21 were moved from Section 5.1.2 to Section 5.1. | Text was moved to Section 5.1 since information applied to both cohorts. |
| Section 5.1 | The independent central reader will be blinded from concomitant AED treatment that the subject has received. | The independent central reader will be blinded from site-specific information and the subject's medical history. | Blinding clarification. |
| Section 5.1 | Not applicable | Interruption of the VEEG is allowed up to 30 minutes per day. Depending on medical needs related to standard of care (eg, MRIs to be performed), interruptions longer than this are acceptable. However, every effort should be made to avoid VEEG interruption of the 2-hour Baseline VEEG and during the first 3 hours after the start of the initial BRV administration for the Confirmatory Cohorts. | Based on Investigator feedback, neonates with hypoxic ischemic encephalopathy may disconnect from the EEG for other assessments, therefore interruptions exist and are allowed. |
| Section 5.1.1 | For the Exploratory Cohort, at least 6 subjects who do not have adequate seizure control after receiving 1 or 2 doses of PB (total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the investigator's discretion) will be enrolled and dosed with one or multiple therapeutic doses of MDZ (dose of MDZ is at the discretion of the | For the Exploratory Cohort, at least 6 subjects who do not have adequate seizure control after receiving 1 to 3 doses of PB (PB treatment may have started prior to the subject's admission into the study site; total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion) will be enrolled and dosed with one or | Dose frequency and continuous infusion are also at the discretion of the Investigator. Based on Investigator feedback, the total PB dose of 20 to 40mg/kg may be administered over 3 separate doses. PB treatment is permitted to start prior to subject's admission into the study. |
| Confidential | oculture the discretion of the | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | Investigator). Phenobarbital treatment must be discontinued prior to entering the Evaluation Period. Approximately 3 hours after the MDZ dosing, an initial low dose of BRV (0.5mg/kg [bid]) will be administered according to the standard of care. | multiple therapeutic doses of MDZ (dose and dosing frequency of MDZ are at the discretion of the Investigator). Phenobarbital treatment must be discontinued prior to entering the Evaluation Period. Approximately 3 hours after the initiation of MDZ dosing, an initial low dose of BRV (0.5mg/kg [bid]) will be administered according to the standard of care. | and any extensions of val. |
| Section 5.1.1 | The first iv dose of PB (standard of care) can be administered between 36 hours and 2 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). The initial PB treatment may have been administered prior to the subject's enrollment in the study. | The Screening Period is up to 36 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). The PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the study site. | PB treatment is permitted to start prior to subject's admission into the study, as well as allowed to be administered at a separate site prior to the study admittance. |
| Section 5.1.1 | Baseline Period (included in the Screening Period): 2 hours immediately prior to the start of MDZ infusion. The occurrence of ENS during the 2-hour period must be confirmed either by the local or | Baseline Period (included in the Screening Period): 2 hours immediately prior to the start of MDZ infusion. The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |
| Confidential | be confirmed either by the local or | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | central VEEG reader prior to the start of MDZ treatment. | administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements (eg, ability for immediate cloud-based central review) can be used as part of the Baseline assessment VEEG. | and any extensions or var |
| Sections 5.1.1, 8.1.3 | Not applicable | The first MDZ infusion marks the starting point of the Evaluation Period. | Clarification of the initiation of the Evaluation Period. |
| Section 5.1.1 | Subjects will receive iv MDZ (one or multiple therapeutic doses; MDZ dose is at the discretion of the Investigator). | Subjects will receive iv MDZ (one or multiple therapeutic doses or continuous infusion; MDZ dose and dosing frequency are at the discretion of the Investigator). | Dose frequency and continuous infusion are also at the discretion of the Investigator. |
| Section 5.1.1 | Following the first BRV infusion, 3 to 6 PK blood microsamples (65µL/sample) will be collected during the 48-hour Evaluation Period from each subject for the determination of plasma concentrations of BRV and its metabolites, as described in Table 5-4. | Following the first BRV infusion, 3 to 6 PK blood microsamples (60µL/sample) will be collected during the 48-hour Evaluation Period from each subject for the determination of plasma concentrations of BRV and its metabolites, as described in Table 5-4. | Volume of microsample tubes is 60 μL. |
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1.2 | For the Confirmatory Cohorts, enrollment will only start after the dosing of BRV is determined based on the PK findings of the Exploratory Cohort. A total of at least 36 subjects without adequate seizure control after receiving 1 or 2 doses of PB (total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion) will enter the Confirmatory Cohorts. | For the Confirmatory Cohorts, enrollment will only start after the dosing of BRV is determined based on the PK findings of the Exploratory Cohort and an existing PK model from N01263. A total of at least 36 subjects without adequate seizure control after receiving 1 to 3 doses of PB (PB treatment may have started prior to the subject's admission into the study site; total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion) will enter the Confirmatory Cohorts. | Based on Investigator feedback, the total PB dose of 20 to 40mg/kg may be administered over 3 separate doses. Dosing frequency is also at the discretion of the Investigator. Per agency recommendation, clarification that BRV dose and dosing frequency is also determined by previous PK modeling of N01263 data. |
| Section 5.1.2 | The first iv dose of PB (standard of care) can be administered between 36 hours and 2 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). The initial PB treatment may have been administered prior to the subject's enrollment in the study. | The Screening Period is up to 36 hours prior to the first administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of BRV). The PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the study site. | PB treatment is permitted to start prior to subject's admission into the study, as well as allowed to be administered at a separate site prior to the study admittance. |
| Confidential | ocument camotibe | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1.2 | - Baseline Period (included in the Screening Period): 2 hours immediately prior to the start of BRV infusion. The occurrence of ENS during this 2 hour period must be confirmed either by the local or central VEEG reader prior to the start of MDZ treatment. | - Baseline Period (included in the Screening Period): 2 hours immediately prior to the start of BRV infusion. The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements (eg, ability for immediate cloud- based central review) can be used as part of the Baseline assessment VEEG. | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |
| Sections 5.1.2, 8.2.3 | Not applicable | The first administration of BRV marks the starting point of the Evaluation Period. | Clarification of the initiation of the Evaluation Period. |
| Section 5.1.2 | The BRV dose for subjects in the Confirmatory Cohorts will be determined based on the results of the PK analysis of the Exploratory Cohort (predicted to be | The BRV dose for subjects in the Confirmatory Cohorts will be determined based on the results of the PK analysis of the Exploratory Cohort (predicted to be approximately the | Per agency recommendation, clarification that BRV dose and dosing frequency is also determined by previous PK modeling of N01263 data. |
| Confidential | ocument | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | approximately the BRV plasma concentrations in the same range as those observed at the highest recommended dose in older children and adults who receive BRV 200mg/day). | BRV plasma concentrations in the same range as those observed at the highest recommended dose in older children and adults who receive BRV 200mg/day), as well as based on an existing PK model from N01263. | anyertensions of vio |
| Section 5.1.2 | Following the first BRV infusion, 6 PK blood microsamples (65µL/sample) will be collected during the 96-hour Evaluation Period for each subject for the determination of plasma concentrations of BRV and its metabolites, as described in Table 5-5. | Following the first BRV infusion, 6 PK blood microsamples (60µL/sample) will be collected during the 96-hour Evaluation Period for each subject for the determination of plasma concentrations of BRV and its metabolites, as described in Table 5-5. | Volume of microsample tubes is 60 μL. |
| Section 5.1.2 | Down-Titration Period (up to 1 week): A Down-Titration Period of up to 1 week is recommended for subjects in the Confirmatory Cohorts who do not proceed to the BRV Extension Period, or start the BRV Extension Period but do not enter the long-term study. | Down-Titration Period (up to I week): A Down-Titration Period of up to 1 week is recommended for subjects in the Confirmatory Cohorts who discontinue BRV treatment prior to completion of the Evaluation Period, who do not proceed to the BRV Extension Period, or start the BRV Extension Period but do not enter the long-term study. | Recommendations for subjects discontinuing BRV treatment. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1.2,<br>Table 5-2<br>footnote b | Not applicable | Subjects discontinuing BRV treatment during the Evaluation Period should start the Down-Titration Period while completing the Evaluation Period in parallel for the full 96 hours. | Recommendations for subjects discontinuing BRV treatment. |
| Table 5-1<br>footnote c,<br>Table 5-2<br>footnote d | The occurrence of ENS during the 2-hour period must be confirmed either by the local or central VEEG reader, prior to the start of MDZ treatment. | The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |
| Table 5-1 footnote d | Not applicable | d Measurement of body weight is optional at 24 and 48 hours. Dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the Evaluation Period. | Clarification of timepoints for weight measurements. |
| Table 5-1<br>footnote f,<br>Table 5-2<br>footnote h | Not applicable | f Video-EEGs that are acquired per<br>standard of care prior to consenting<br>and meet study-specific technical and<br>quality requirements can be used as | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |
| Confidential | Schlaghteathor | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | part of the Baseline assessment VEEG. | :OLE OL |
| Table 5-1 footnote g | g Following the first BRV infusion, 3 to 6 blood microsamples (65µL/sample) will be collected from each subject in the Exploratory Cohort. | g Following the first BRV infusion,<br>3 to 6 blood microsamples<br>(60μL/sample) will be collected from<br>each subject in the Exploratory<br>Cohort. | Volume of microsample tubes is 60 μL. |
| Table 5-1<br>footnote i,<br>Table 5-2<br>footnote k | Not applicable | i For Screening and determination of eligibility, use of laboratory data acquired prior to Screening per standard of care inside or outside the study site within 36 hours prior to the start of the Evaluation Period is allowed. | Allowance of use of standard of care laboratory data. |
| Table 5-2<br>footnote e | Not applicable | e Measurement of body weight is optional at 24, 48, 72, and 96 hours. Dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the Evaluation Period. | Clarification of timepoints for weight measurements. |
| Table 5-2 footnote i | i Following the first BRV infusion, 6 blood microsamples (65μL/sample) will be collected | i Following the first BRV infusion, 6 blood microsamples (60μL/sample) | Volume of microsample tubes is 60 μL. |

Confidential Hochmen


y 2021

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | during the Evaluation Period from each subject. | will be collected during the Evaluation Period from each subject. | ionsor |
| Table 5-3 footnote a | a i For Screening and determination of eligibility, use of laboratory data acquired prior to Screening per standard of care inside or outside the study site within 36 hours prior to the start of the Evaluation Period is allowed. A Down-Titration Period of up to 1 week applies only to subjects in the Confirmatory Cohorts. The Down-Titration Period is recommended for subjects who do not proceed to the BRV Extension Period, or start the BRV Extension Period but do not enter the long-term study. | a A Down-Titration Period of up to 1 week applies only to subjects in the Confirmatory Cohorts. The Down-Titration Period is recommended for subjects who discontinue BRV treatment prior to completion of the Evaluation Period, who do not proceed to the BRV Extension Period, or start the BRV Extension Period but do not enter the long-term study. Subjects discontinuing BRV treatment during the Evaluation Period can continue assessments pertaining to the Evaluation Period, except the collection of blood microsamples for the determination of BRV plasma concentrations. Those subjects should start the Down-Titration Period in parallel to completing the Evaluation Period. | Recommendations for subjects discontinuing BRV treatment. |
| Section 5.4.2 | The doses planned to be applied in this study are based on the available data in 96 pediatric subjects (overall, 1 month to 17 years of age with the following number of subjects per pediatric age group: 1 month to <2 years of age, 29 subjects; 2 years | The doses planned to be applied in this study are based on pediatric data collected in N01263 subjects (overall 96 subjects in the age range of 1 month to 17 years with the following number of subjects per pediatric age group: 1 month to <2 years of age, | Clarification of dosage selection. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | to <6 years of age, 26 subjects;<br>6 years to <12 years of age,<br>24 subjects; 12 years to <16 years of<br>age, 17 subjects). | 29 subjects; 2 years to <6 years of age, 26 subjects; 6 years to <12 years of age, 24 subjects; 12 years to <16 years of age, 17 subjects). | *tensions of vio |
| Section 5.4.2 | The dose of BRV to be administered in the Confirmatory Cohorts will be determined by the evaluation of plasma samples collected in the Exploratory Cohort and should not exceed the range of plasma concentrations observed in children ≥1 month old who received BRV 4mg/kg/day. | The dose of BRV to be administered in the Confirmatory Cohorts will be determined by the evaluation of plasma samples collected in the Exploratory Cohort, as well as by the PK modeling of N01263 data described above, and should not exceed the range of plasma concentrations observed in children ≥1 month old who received BRV 4mg/kg/day. The plasma concentration of BRV 4mg/kg/day for neonates is predicted to be approximately equivalent to the plasma concentrations observed in adults who receive BRV 200mg/day. The dose in neonates to reach the same plasma concentrations will be confirmed or adapted upon completion of enrollment and analysis of PK and safety data from the Exploratory Cohort involving the DMC. The BRV dose used in the Confirmatory Cohorts will be based | Per agency recommendation, clarification that BRV dose and dosing frequency is also determined by previous PK modeling of N01263 data. Clarification of DMC participation in determination of Confirmatory Cohort dosage. |

Confidentia

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | on recommendations made by the DMC. | ionsold |
| Section 6.1 | 2.Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the 2 hours prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite receiving PB (total therapeutic administered dose of 20 to 40mg/kg) for the treatment of repeated seizures. | 2a. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the 2 hours prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite receiving PB (total therapeutic administered dose of 20 to 40mg/kg) for the treatment of repeated seizures. The occurrence of ENS during the 2- hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. | Local and central reader preference clarification: |
| Section 6.2 | 1. Subject received AED treatment (other than the required 1 or 2 doses of PB [total therapeutic administered dose of 20 to 40mg/kg] for the treatment of repeated seizures) prior to entering the Evaluation Period. | 1a. Subject received AED treatment (other than the required 1 to 3 doses of PB [total therapeutic administered dose of 20 to 40mg/kg] for the treatment of repeated seizures) prior to entering the Evaluation Period. | Based on Investigator feedback, the total PB dose of 20 to 40mg/kg may be administered over 3 separate doses. |
| Section 6.2 | 8. Subject has conjugated bilirubin levels >2mg/dL. | 8a. Subject has direct (conjugated) bilirubin levels >2mg/dL. | Language correction. |
| Confidential | Jocithent Cos and | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 6.3 | 4. Subject has conjugated bilirubin levels >2mg/dL. | 4a. Subject has direct (conjugated) bilirubin levels >2mg/dL. | Language correction. |
| Section 6.3.1 | • Subject has conjugated bilirubin >2mg/dL. | • Subject has direct (conjugated) bilirubin >2mg/dL. | Language correction. |
| Section 7.2 | Subjects in the Exploratory Cohort will be dosed with iv MDZ (dosing of MDZ is at the discretion of the Investigator). | Subjects in the Exploratory Cohort will be dosed with iv MDZ (dosing and dosing frequency of MDZ are at the discretion of the Investigator). | Dose frequency and continuous infusion are also at the discretion of the Investigator. |
| Section 8.1.1 | The first iv dose of PB (standard of care) can be administered between 36 hours and 2 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). | The Screening Period is up to 36 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). | PB treatment is permitted to start prior to subject's admission into the study, as well as allowed to be administered at a separate site prior to the study admittance. |
| Sections<br>8.1.1, 8.2.1 | The initial PB treatment may have started prior to the subject's admission to the study. | The PB treatment may have started prior to the subject's admission to the study and/or at a location other than the study site but should be completed prior to the 2-hour Baseline Period. | PB treatment is permitted to start prior to subject's admission into the study, as well as allowed to be administered at a separate site prior to the study admittance. |
| Section 8.1.2 | Not applicable | Video-EEGs that are acquired per<br>standard of care prior to consenting<br>and meet study-specific requirements<br>(eg, ability for immediate cloud-based | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | central review) can be used as part of the Baseline assessment VEEG. | ionsol |
| Section 8.1.2 | The occurrence of ENS during this 2-hour period must be confirmed either by the local or central VEEG reader prior to the start of MDZ treatment. | The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |
| Section 8.1.2,<br>8.2.2 | Verification of inclusion/exclusion criteria. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the 2 hours prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite PB treatment | Verification of inclusion/exclusion criteria. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the 2 hours prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite PB treatment prior to Baseline | PB treatment is permitted to start prior to subject's admission into the study, as well as allowed to be administered at a separate site prior to the study admittance. |
| Section 8.1.2 | Not applicable Not applicable Real | Baseline laboratory measurements will be performed by local laboratories unless historical data is available. Historical safety laboratory assessments, previously collected as standard of care, may be accepted from referring hospitals as Baseline measurement if performed 36 hours prior to the start of the Evaluation Period. In this case, test results will be | Allowance of use of standard of care laboratory data. |
| Confidential | ocument cannot | | |
| This | • | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | considered medical history. Prior laboratory assessment results should already be available at Baseline and verified prior to initiation of the MDZ infusion. | l extensions of |
| Section 8.1.3 | Body weight (24 and 48 hours) | Body weight (optional [at 24 and 48 hours]; dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent weight measurement, upon discretion of the Investigator, if weight is measured during the Evaluation Period) | Clarification of timepoints for weight measurements. |
| Sections<br>8.1.4, 8.2.4 | Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study (see Section 8.1.3.2). | Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study N01266 (see Section 8.1.3.2). If study N01266 is performed outside the N01349 hospital, an interval of up to 3 days between the N01349 EPV2 and N01266 Entry Visit is allowed. | Clarification of visit intervals. |
| Section 8.2.1 | The Screening Period (up to 36 hours) will be from the signing and dating of the written ICF by the | The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal | Elimination of repetition. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | parent(s) or legal representative(s) of<br>the subject to the end of the Baseline<br>Period. | representative(s) of the subject to the end of the Baseline Period. | Sidnsor |
| Section 8.2.1 | The first iv dose of PB (standard of care) can be administered between 36 hours and 2 hours prior to the first administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of BRV). | The Screening Period is up to 36 hours prior to the first administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of BRV). | PB treatment is permitted to start prior to subject's admission into the study, as well as allowed to be administered at a separate site prior to the study admittance. |
| Section 8.2.2 | The occurrence of ENS during this 2-hour period must be confirmed either by the local or central VEEG reader prior to the start of BRV treatment. | The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements (eg, ability for immediate cloud-based central review) can be used as part of the Baseline assessment VEEG. | Permitted use of EEG traces recorded before parents consented for the determination of the Baseline EEG. |
| Section 8.2.2 | Not applicable | Baseline laboratory measurements will be performed by local laboratories unless historical data is available. Historical safety laboratory | Allowance of use of standard of care laboratory data. |
| Confidential | Schuleuteanhor | | |
| This d | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | assessments, previously collected as standard of care, may be accepted from referring hospitals as Baseline measurement if performed 36 hours prior to the start of the Evaluation Period. In this case, test results will be considered medical history. Prior laboratory assessment results should already be available at Baseline and verified prior to initiation of BRV administration. | and any extensions of vall |
| Section 8.2.3 | Not applicable | If subjects in the Confirmatory Cohort receive <8 BRV doses, those subjects are allowed to continue study participation and complete study assessments per Table 17-2, with the exception of PK blood sampling. Those subjects should start the Down-Titration Period while completing the Evaluation Period in parallel for the full 96 hours. | Recommendations for subjects discontinuing BRV treatment. |
| Section 8.2.3 | Body weight (at 24, 48, 72 and 96 hours). | Body weight (optional [at 24, 48, 72 and 96 hours]; dosage of BRV during the Evaluation Period will be based on the subject's weight measured prior to the start of the first BRV administration. However, dosage calculation can be adjusted to a more recent | Clarification of timepoints for weight measurements. |
| Confidential | ocument | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | weight measurement, upon<br>discretion of the Investigator, if<br>weight is measured during the<br>Evaluation Period) | ATENSIONS OF VIO |
| Section 8.2.5 | A Down-Titration Period of up to 1 week is recommended for subjects who complete the Evaluation Period, but do not enter the BRV Extension Period, or start the BRV Extension Period but do not continue into the long-term study for any reason. | A Down-Titration Period of up to 1 week is recommended for subjects who complete the Evaluation Period, but do not enter the BRV Extension Period, discontinue BRV during the Evaluation Period, or start the BRV Extension Period but do not continue into the long-term study for any reason. | Recommendations for subjects discontinuing BRV treatment. |
| Section 9.1 | For the determination of plasma concentrations of BRV and BRV metabolites, up to 6 blood microsamples (65µL/sample) will be collected per subject in the Exploratory (3 to 6 blood microsamples) and Confirmatory Cohorts (up to 6 blood microsamples) at 3 predetermined timepoints per day. An additional microsample (65µL) will be collected per subject for the determination of plasma concentrations of concomitant AEDs (PB and PHT). | For the determination of plasma concentrations of BRV and BRV metabolites, up to 6 blood microsamples (60µL/sample) will be collected per subject in the Exploratory (3 to 6 blood microsamples) and Confirmatory Cohorts (up to 6 blood microsamples) at 3 predetermined timepoints per day. An additional microsample (60µL) will be collected per subject for the determination of plasma concentrations of concomitant AEDs (PB and PHT). | Volume of microsample tubes is $60~\mu L$ . |
| Confidential | ocument com. | | |
| This | • | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Sections 10.1,<br>13.5.1 | Absolute reduction and proportion of clinical seizures correlated with continuous VEEG from Baseline to the end of the 96-hour Evaluation Period, and at each of the 3-hour intervals | Absolute and percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion | Alignment of language presented in the Pediatric Investigation Plan. |
| Section 11.1.1 | <ul> <li>Potential drug-induced liver injury as indicated by:</li> <li>Conjugated bilirubin &gt;2mg/dL</li> </ul> | <ul> <li>Potential drug-induced liver injury as indicated by:</li> <li>Direct (conjugated) bilirubin &gt;2mg/dL</li> </ul> | Language correction. |
| Section 11.1.2 | In line with GCP, from the signing of the ICF, the Investigator will record any AEs that occur to the subject, and will keep detailed records of all AEs that occur. All AEs will be recorded daily in each subject's medical notes. Serious AEs, AEs that are considered related to the medicinal (investigational) product, AEs leading to discontinuation, infusion site reactions, or AEs considered by the Investigator to be critical to the safety evaluation of the protocol will also be recorded on the Adverse Event eCRF. | In line with GCP, from the signing of the ICF, the Investigator will evaluate the subject for occurrence of any AEs based on continued observation and medical notes throughout the study. Serious AEs, AEs that are considered related to the medicinal (investigational) product, AEs leading to discontinuation, BRV infusion site reactions, or AEs considered by the Investigator to be critical to the safety evaluation of the protocol will also be recorded on the Adverse Event eCRF. | Adverse event recording clarification. |
| Confidential | Event eCRE. | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 11.2 | Not applicable | Blood samples will be collected in line with Section 13.2 of the "Ethical Considerations for Clinical Trials on Medicinal Products Conducted with the Paediatric Population" (European Union Commission ad hoc group, 2008). | Recommendations for subjects discontinuing BRV treatment. |
| Section 11.2 | All laboratory measurements, including laboratory assessments for PDILI, will be performed by local laboratories. | Laboratory measurements, including laboratory assessments for PDILI, will be performed by local laboratories unless historical data is available. Historical safety laboratory assessments, previously collected as standard of care, may be accepted from referring hospitals as Baseline measurement if performed 36 hours prior to the Evaluation Period. | Allowance of use of standard of care laboratory data. |
| Section 11.2 | As part of routine assessments performed by local laboratories, the parameters shown in Table 11-1 will be measured. | As part of routine assessments performed by local laboratories, the parameters shown in Table 11-1 and Table 11-2 will be measured. | Table addition. |
| Table 11-3 | Conjugated bilirubin | Direct (conjugate) bilirubin | Language correction. |
| Section 11.2.1.3 | Not applicable | Recommended testing is at the discretion of the Investigator and should be individualized | Testing recommendation clarification. |

Confidential Accument

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | appropriately based on clinical situation. | onsor |
| Section 11.3.8 | Not applicable | Withdrawal and rebound phenomena, if any, will be captured from data collected at the end of BRV exposure for subjects in both the Exploratory and Confirmatory Cohorts | Text was relocated. |
| Section 11.3.9 | Numbers and percentage of subjects requiring mechanical ventilation at the time they are treated with BRV will be recorded from Baseline through the 48-hour Evaluation Period for the Exploratory Cohort and the 96-hour Evaluation Period for the Confirmatory Cohorts and compared between subjects that required BRV only and subjects treated with BRV and receiving rescue medication or other AEDs. Absolute and relative duration of ventilation at the time subjects are treated with BRV will be recorded over the Evaluation Period and compared between subjects treated with BRV only and subjects treated with BRV and receiving rescue medication or other AEDs. | Numbers and percentage of subjects requiring mechanical ventilation will be recorded from Baseline through the 48-hour Evaluation Period for the Exploratory Cohort and the 96-hour Evaluation Period for the Confirmatory Cohort. Duration of mechanical ventilation will be recorded over the Evaluation Period. | Alignment of language presented in the Pediatric Investigation Plan. |

Confidentia

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 13.3 | Not applicable | The analysis of the PK parameters for<br>the Exploratory and Confirmatory<br>Cohorts will include a sub-analysis<br>for any concomitant use of<br>hypothermia. | Content consistency. Text was relocated. |
| Section 13.4 | The primary cause of seizure (HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes) may also be used to categorize the safety review. | The primary cause of seizure (eg, HIE, hemorrhage, or infarction; CNS malformations; CNS infections; undetermined causes) may also be used to categorize the safety review. | Typographical change. |
| Section 13.7 | Subjects in the Confirmatory Cohorts are withdrawn, are switched over to another AED treatment, prior to the Evaluation Period or are administered >1 dose of rescue medication (including BZDs) following the first 3 hours after initial BRV treatment started will be considered BRV nonresponders. | Subjects in the Confirmatory Cohorts who drop out due to lack of BRV efficacy, are switched over to another AED treatment, or are administered >1 dose of rescue medication (including BZDs) following the first 3 hours after initial BRV treatment started will be considered BRV nonresponders. | Recommendations for subjects discontinuing BRV treatment. |
| Section 13.8.1 | Upon the completion of the Exploratory Cohort, the DMC will be provided with the summaries and the listings of PK and safety data for review (see Section 13.8.3). | Upon the completion of the Exploratory Cohort, the DMC will be provided with the summaries and the listings of PK and safety data for review to make recommendations concerning the dosing of BRV in the Confirmatory Cohorts (see Section 13.8.3). | Clarification of DMC participation in determination of Confirmatory Cohort dosage. |
| Confidential | Delinent | | |
| Ki. | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 14.1 | Not applicable | An informed consenting process managed via telephone is allowed where applicable per local regulations. | Allowance of telephone consenting process. |
| References | Not applicable | European Union Commission ad hoc group. Recommendations of the ad hoc group for the development of implementing guidelines for Directive 2001/20/EC relating to good clinical practice in the conduct of clinical trials on medicinal products for human use. Ethical Considerations for Clinical Trials on Medicinal Products Conducted with the Paediatric Population. 2008; 13.2. https://ec.europa.eu/health/sites/health/files/files/eudralex/vol-10/ethical_considerations_en.pdf. | Reference addition. |


Figure 5-1: Schematic overview of the study for the Exploratory Cohort



BRV=brivaracetam; ICF=informed consent form; MDZ=midazolam; VEEG=(multichannel) video-electroencephalography

Note: A continuous consent process will be followed. Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the ICF after the occurrence of seizures has been confirmed by VEEG. During the course of the study, parent(s) or legal representative(s) will be updated about the care of their neonate, and continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s).

<sup>a</sup> The anticipated duration of the BRV Extension Period is up to 28 days of postnatal age (+7 days).


<sup>&</sup>lt;sup>b</sup> Subjects in the Exploratory Cohort will enter the Safety Follow-Up Period, if they complete the Evaluation Period or are discontinued from the BRV Extension Period.

For adjustment of dosing and time intervals, Figure 5-1 was changed to:

Figure 5-1: Schematic overview of the study for the Exploratory Cohort



BRV=brivaracetam; ICF=Informed Consent form; MDZ=midazolam; VEEG=(multichannel) video-electroencephalography

Note: A continuous consent process will be followed. Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the ICF after the occurrence of seizures has been confirmed by VEEG. During the course of the study, parent(s) or legal representative(s) will be updated about the care of their neonate, and continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s).

<sup>a</sup> The anticipated duration of the BRV Extension Period is up to 28 days of postnatal age (+7 days).


b Subjects in the Exploratory Cohort will enter the Safety Follow-Up Period if they complete the Evaluation Period or are discontinued from the BRV Extension Period.

Figure 5-2: Screening and Evaluation Periods (Exploratory Cohort)



BRV=brivaracetam; ICF=informed consent form; MDZ=midazolam; PB=phenobarbital

Note: The Screening Period is from signing and dating of the written ICF up to Cohort Assignment. The first iv dose of PB (standard of care) can be administered between 36 hours and 2 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). The PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the designated site.

- <sup>a</sup> Treatment with MDZ will continue in parallel with BRV.
- b Subjects enrolled in the Exploratory Cohort will receive a therapeutic dose of MDZ (dose and dosing frequency of MDZ are at the discretion of the Investigator) prior to receiving BRV. Subsequently, an initial low dose of iv BRV will be administered. At the discretion of the Investigator, 3 additional iv BRV doses can be administered, up to a total of 4 iv BRV doses (0.5mg/kg twice daily [bid]), during the 48-hour Evaluation Period.
- <sup>c</sup> If seizures are adequately controlled with previous AED treatment per SOC, subjects will be considered screen failures and will not be permitted to enter the Evaluation Period.

For adjustment of dosing and time intervals, Figure 5-2 was changed to:

Figure 5-2: Screening and Evaluation Periods (Exploratory Cohort)



BRV=brivaracetam; ICF=Informed Consent form; MDZ=midazolam; PB=phenobarbital

Note: The Screening Period is from signing and dating of the written ICF up to Cohort Assignment. The Screening Period is up to 36 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). The PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the study site.

<sup>&</sup>lt;sup>a</sup> Treatment with MDZ will continue in parallel with BRV.

b Subjects enrolled in the Exploratory Cohort will receive one or multiple therapeutic doses or continuous infusion of MDZ (dose and dose frequency of MDZ) are at the discretion of the Investigator) prior to receiving BRV. Subsequently, an initial low dose of iv BRV will be administered. At the discretion of the Investigator, 3 additional iv BRV doses can be administered, up to a total of 4 iv BRV doses (0.5mg/kg twice daily [bid]), during the 48-hour Evaluation Period.

<sup>&</sup>lt;sup>c</sup> If seizures are adequately controlled with previous AED treatment per SOC, subjects will be considered screen failures and will not be permitted to enter the Evaluation Period.

Figure 5-3: Schematic overview of the study for the Confirmatory Cohorts



BRV=brivaracetam; ICF=informed consent form; VEEG=(multichannel) video-electroencephalography Note: A continuous consent process will be followed. Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the ICF after the occurrence of seizures has been confirmed by VEEG. During the course of the study, parent(s) or legal representative(s) will be updated about the care of their neonate, and continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s).

<sup>a</sup> The anticipated duration of the BRV Extension Period is up to 28 days of postnatal age (+7 days).

For adjustment of dosing and time intervals, Figure 5-3 was changed to:

Figure 5-3: Schematic overview of the study for the Confirmatory Cohorts



BRV=brivaracetam; ICF=Informed Consent form; VEEG=(multichannel) video-electroencephalography Note: A continuous consent process will be followed. Parent(s) or legal representative(s) will be informed about the study as early as possible and asked to sign the ICF after the occurrence of seizures has been confirmed by VEEG. During the course of the study, parent(s) or legal representative(s) will be updated about the care of their neonate, and continuous consent will be ensured by meetings between the Investigator (or designee) and the subject's parent(s) or legal representative(s).

<sup>a</sup> The anticipated duration of the BRV Extension Period is up to 28 days of postnatal age (+7 days).

Figure 5-4: Screening and Evaluation Periods (Confirmatory Cohorts)



AED=antiepileptic drug; BRV=brivaracetam; ICF=informed consent form; PB=phenobarbital

Note: The Screening Period is from signing and dating of the written ICF up to Cohort Assignment. The first iv dose of PB (standard of care) can be administered between 36 hours and 2 hours prior to the first administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of BRV). The initial PB treatment may have been administered prior to the subject's enrollment in the study.

<sup>&</sup>lt;sup>a</sup> Switching to another AED or addition of rescue medication should only occur following 3 hours after the first BRV administration.

b If seizures are adequately controlled with previous AED treatment per SOC, subjects will be considered screen failures and will not be permitted to enter the Evaluation Period.

For adjustment of dosing and time intervals, Figure 5-4 was changed to:

Figure 5-4: Screening and Evaluation Periods (Confirmatory Cohorts)



AED=antiepileptic drug; BRV=brivaracetam; ICF=Informed Consent form; PB=phenobarbital

Note: The Screening Period is from signing and dating of the written ICF up to Cohort Assignment. The Screening Period is up to 36 hours prior to the first administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of BRV). The PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the study site.

<sup>&</sup>lt;sup>a</sup> Switching to another AED or addition of rescue medication should only occur following 3 hours after the first BRV administration.

b If seizures are adequately controlled with AED treatment per SOC, subjects will be considered screen failures and will not be permitted to enter the Evaluation Period.

Clinical Study Protocol

Table 11-1: Laboratory measurements

| Hematology | Biochemistry | Urinalysis | Endocrinology |
|----------------------|-------------------|------------|----------------|
| Basophils | Calcium | Albumin | TSH |
| Eosinophils | Chloride | Bacteria | T <sub>3</sub> |
| Lymphocytes | Potassium | Glucose | T <sub>4</sub> |
| Atypical lymphocytes | Sodium | рН | or vari |
| Monocytes | Glucose | RBC | ins |
| Neutrophils | BUN | WBC | "SILSIE |
| Hematocrit | Creatine kinase | | et |
| Hemoglobin | AST | | and |
| МСН | ALT | 95 | Š |
| MCHC | GGT | Zijol | |
| MCV | Total bilirubin | Oplice | |
| Platelet count | LDH | Ry Clay | |
| RBC count | Total cholesterol | 1211 | |
| WBC count | C AST LONG | C DIN II I | |

ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen;

GGT=gamma-glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin;

This document cannot be used to support any more MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell;

T3=triiodothyronine; T4=thyroxine; TSH=thyroid-stimulating hormone; WBC=white blood cell

For clarification of laboratory assessments, Table 11-1 was split into mandatory and optional measurements:

**Table 11-1: Mandatory laboratory measurements** 

| Hematology | Biochemistry |
|----------------------|-------------------------------|
| Basophils | Calcium |
| Eosinophils | Chloride |
| Lymphocytes | Potassium |
| Atypical lymphocytes | Sodium |
| Monocytes | Glucose |
| Neutrophils | Urea/BUN <sup>a</sup> |
| Hematocrit | Creatine kinase |
| Hemoglobin | AST |
| МСН | ALT |
| MCHC | ALP |
| MCV | GGT GGT |
| Platelet count | LDH |
| RBC count | Total bilirubin |
| WBC count | Direct (conjugated) bilirubin |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; GGT=gamma-glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; WBC=white blood cell

Table 11-2: Optional laboratory measurements

| Biochemistry | Urinalysis <sup>b</sup> | Endocrinology <sup>c</sup> |
|---|---|---|
| Total cholesterol <sup>a</sup> | Protein | TSH |
| 2,55 | Bacteria | $T_4$ |
| 0,00 | Glucose | |
| allin | рН | |
| CITY | RBC | |
| | WBC | |

RBC=red blood cell; T<sub>4</sub>=thyroxine; TSH=thyroid-stimulating hormone; WBC=white blood cell


<sup>&</sup>lt;sup>a</sup> Urea <u>or</u> BUN to be tested depending on the local lab's standard panel for neonates.

<sup>&</sup>lt;sup>a</sup> Total cholesterol to be measured if this is part of the local lab's standard panel for neonates.

<sup>&</sup>lt;sup>b</sup> Urinalysis to be performed only if a urine sample was obtained for clinical purposes.

<sup>&</sup>lt;sup>c</sup> TSH and T<sub>4</sub> to be recorded for the study only if measured for neonatal screening of congenital hypothyroidism prior to or during study participation.

### 17.4 **Protocol Amendment 4**

### Rationale for the amendment

The primary purpose of this nonsubstantial protocol amendment is to update the laboratory measurement section where creatinine was inadvertently not included as a mandatory laboratory measurement. Creatinine is needed for monitoring of renal function. Clarification for optional laboratory measurements has also been provided.

# Specific changes Change #1

Table 11-1

Creatinine has been added as a new laboratory parameter and in addition, the following footnote b was added:

<sup>b</sup> During the first days of life, creatinine will only be collected if the site assesses this parameter per standard of care.

## Change #2

Table 11-2 Footnote b

Urinalysis to be performed only if a urine sample was obtained for clinical purposes.

This document cannot be used to support any marketing atthorn. Urinalysis to be performed only if a urine sample was obtained for clinical purposes. A urine

### 17.5 Protocol Amendment 5

### Rationale for the amendment

The purpose of this substantial amendment is to implement the changes from the agreed Pediatric Investigation Plan for BRV in order to help improve enrollment rate (to date, 1 subject has been enrolled). The primary change is to remove restriction in terms of concomitant medication by replacing PB only with SOC for the Exploratory Cohort and one or more of the following AEDs: PB, MDZ, PHT, LEV (≤60mg/kg/day) or LDC for the Confirmatory Cohort. Also, the age range has been modified. Additionally, subjects will be proposed to enroll into a new long-term follow-up study.

A brief list of modifications to the protocol include the following:

- Age at enrollment modified
- Phenobarbital no longer required as first line treatment prior to BRV; replaced by "ENS treatment per SOC (first line, second line, or subsequent treatment; choice of treatment, dose and dosing at the Investigator's discretion)" for the Exploratory Cohort and "one or more of the following AEDs: PB, MDZ, PHT, LEV (≤60mg/kg/day) or LDC (first line, second line or subsequent treatment; dose and dosing at the Investigator's discretion)" for the Confirmatory Cohorts
- 2-hour Baseline EEG and 48-hour VEEG removed from the Exploratory Cohort; required ENS to be confirmed by the Investigator via local EEG
- Duration of the 2-hour Baseline Period shortened to up to 1 hour for the Confirmatory Cohorts and separated by seizure activity: "at least 1 hour" for subjects with intermittent ENS and "up to 30 minutes" for subjects in status epilepticus
- Definition of status epilepticus for neonates enrolled into this study was added
- Treatment with "MDZ only" during the first 3 hours of the Evaluation Period removed from the Confirmatory Cohort; duration of the Evaluation Period hence shortened from 51 to 48 hours
- Historical control changed from "MDZ" to "one or more AED treatments"
- The initiation of LEV treatment after the first time BRV is introduced is prohibited throughout the study for the Confirmatory Cohorts
- Inclusion Criteria 2a and 3, Exclusion Criteria 1a and 2 modified
- Use of concomitant medication and rescue medication adapted
- PK variables split into "primary" and "other" PK variables
- Safety variables categorized as "secondary safety variable" and "other safety variables"
- Reference to N01266 removed since this study will be closed before the last N01349 subject was able to participate in that study for 3 years. Those subjects may instead roll-over to EP0132. Study number replaced by generic term "long-term study"
- Clarified that enrollment will be put on hold during the first DMC (that was always the plan but not explicitly mentioned in the protocol)
- Marketing status of BRV updated

# Specific changes

| Specific ch | anges | | idio |
|---|---|---|---|
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| STUDY<br>CONTACT<br>INFORMAT-<br>ION | Removed study physican name, address, and contact information | Added relevant information | Study physician has changed |
| Section 1<br>Summary | Subjects will first receive 1 to 3 doses of phenobarbital (PB) (total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion). If they do not have adequate seizure control after receiving PB, they may be enrolled into N01349, but they must stop PB treatment. | Subjects will first receive antiepileptic drugs (AEDs) for the treatment of electroencephalographic neonatal seizures (ENS) (first-line, second-line, or subsequent treatment, which may have started prior to the subject's admission into the study site; dose and dosing regimen at the Investigator's discretion). If they do not have adequate seizure control after the treatment with AEDs, they may be enrolled into N01349. | PB no longer required as first-line treatment prior to BRV |
| Section 1<br>Summary | For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple doses or continuous infusion of a therapeutic dose of midazolam (MDZ) (dose and dosing frequency of MDZ is at the discretion of the Investigator) prior to receiving BRV | For the Exploratory Cohort (first step), enrolled subjects will receive 1 or more AEDs per standard of care (SOC) for the treatment of ENS (first-line, second-line, or subsequent treatment; choice of treatment, dose, and dosing frequency is at the discretion of the Investigator) prior to receiving BRV | Historical control changed from MDZ to "1 or more AED treatments" |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 1<br>Summary | The primary objective of this study is to evaluate the PK of BRV in neonates who have seizures that are not adequately controlled with PB treatment, and to identify the optimal BRV dose (Exploratory Cohort) for the treatment of subjects enrolled into the Confirmatory Cohorts of this study. Secondary objectives include the evaluation of the short-term safety and tolerability of BRV in neonates and the evaluation of the efficacy of BRV in severe and nonsevere seizure burden (defined as total minutes of ENS per hour) in neonates with seizures that are not adequately controlled with PB treatment | The primary objective of this study is to evaluate the PK of BRV in neonates who have seizures that are not adequately controlled with previous AED treatment, and to identify the optimal BRV dose (Exploratory Cohort) for the treatment of subjects enrolled into the Confirmatory Cohorts of this study. Secondary objectives include the evaluation of the short-term safety and tolerability of BRV in neonates and the evaluation of the efficacy of BRV in severe and nonsevere seizure burden (defined as total minutes of ENS per hour) in neonates with seizures that are not adequately controlled with previous AED treatment | PB no longer required as first line treatment prior to BRV |
| Section 1<br>Summary | Subjects must be of 34 weeks to less than 42 weeks of gestational age (GA) at birth and up to 28 days of postnatal age at the time of enrollment. | At enrollment, subjects must be at least 34 weeks of corrected gestational age (CGA). In addition, term neonates up to 27 days of postnatal age (PNA) and preterm neonates up to 40 weeks of postmenstrual age (PMA) and 27 days of PNA can be enrolled. | Age at enrollment was modified |
| Confidential | Hocumant canne | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 1<br>Summary | Subjects must have a confirmed diagnosis of ENS by multichannel video-electroencephalography (VEEG) of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the 2 hours prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite receiving PB for the treatment of repeated seizures. The maximum study duration per subject will be up to 75 days, which consists of a Screening Period, Baseline Period, Evaluation Period, BRV Extension Period, Down-Titration Period (Confirmatory Cohorts only), and Safety Follow-Up Period. All subjects who participate in the BRV Extension Period must be offered entry into the long-term study N01266, if they meet the eligibility criteria. Before entering the long-term study, subjects must be on oral BRV | Subjects must have a confirmed diagnosis of ENS by multichannel video-electroencephalography (VEEG) of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS prior to entering the Evaluation Period (ENS is defined as a seizure lasting for at least 10 seconds on VEEG), despite receiving AED treatment. The maximum study duration per subject will be up to 75 days, which consists of a Screening Period, Baseline Period (Confirmatory Cohorts only), Evaluation Period, BRV Extension Period, Down-Titration Period (Confirmatory Cohorts only), and Safety Follow-Up Period. All subjects who participate in the BRV Extension Period must be offered entry into a long-term study, if they meet the eligibility criteria. Before entering the long-term study, subjects must be on oral BRV | Clarification Clarification And any extensions of the state of the s |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 1<br>Summary | The PK variables are the plasma concentrations of BRV, the area under the curve (AUC), volume of distribution, and clearance of BRV in neonates. Further, PK assessments will include plasma concentrations of concomitant antiepileptic drugs (AEDs) (PB and phenytoin [PHT]). | The PK variables are the plasma concentrations of BRV, the area under the curve (AUC), volume of distribution, and clearance of BRV in neonates. Further, PK assessments will include plasma concentrations of concomitant phenobarbital (PB) and phenytoin (PHT) if administered | Clarification of and any extensions |
| Section 1<br>Summary | The efficacy of BRV will be analyzed based on the following variables: | The efficacy of BRV will be analyzed for the Confirmatory Cohorts based on the following variables: | Clarification |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 1<br>Summary | A BRV responder is defined as a subject who achieves a reduction in seizure burden (ENS in minutes per hour), compared to the seizure burden measured during the 2-hour Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment. Reduction in seizure burden is defined as at least 80% reduction in nonsevere seizure burden (nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in any 30-minute timespan) or at least 50% reduction in severe seizure burden (severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan); timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to ≤30 minutes, >30 to ≤60 minutes, >60 to ≤90 minutes, and >90 to ≤120 minutes. | A BRV responder is defined as a subject who achieves a reduction in seizure burden (ENS in minutes per hour), without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment. Reduction in seizure burden is defined as at least 80% reduction in nonsevere seizure burden (nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in all 30-minute timespans) or at least 50% reduction in severe seizure burden (severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan). Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to ≤30 minutes, >30 to ≤60 minutes, >60 to ≤90 minutes, and >90 to ≤120 minutes. | Clarification Clarification And any extensions of the state of the s |
| Section 1<br>Summary | Key efficacy variables | Secondary efficacy variables | Changed key efficacy variables to efficacy variables |
| Confidential | document canno | | variables |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 2.1<br>Epidemology<br>and treatment<br>of targeted<br>disease | Minor editorial changes | Accepted | Not applicable of a service of |
| Section 2.2<br>Background<br>information<br>regarding<br>product | Removed outdated background information | Updated with new background information | To provide more current marketing information |
| Section 2.2<br>Background<br>information<br>regarding<br>product | The following text was removed: The study was amended to allow direct enrollment of at least 100 subjects 4 years to <17 years of age who have focal epilepsy. Subject participation in N01266 will extend from study entry for | No additional text was added | Removed study information for N01266 |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 2.3 Rationale for the study | N01349 represents the first study of BRV in neonatal subjects, and will evaluate the PK, efficacy, and safety of BRV in neonates (with an age of 34 weeks to less than 42 weeks of GA at birth and up to 28 days of postnatal age at the time of enrollment) with repeated EEG seizures. A historical control group treated with MDZ from literature (matched in age and condition) will be used for the evaluation of efficacy. | N01349 represents the first study of BRV in neonatal subjects, and will evaluate the PK, efficacy, and safety of BRV in neonates (up to 27 days of PNA and preterm neonates up to 40 weeks of PMA and 27 days of PNA. | Age at enrollment was modified |
| Section 3.1 Primary objective and Section 3.2 Secondary objectives | Removed "PB" | Added "previous AED" | PB no longer required as first line treatment prior to BRV |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 4.1<br>PK variables<br>(Exploratory<br>and<br>Confirmatory<br>Cohorts) | The PK variables, all of which are primary, are as follows: • Plasma concentrations of BRV and its metabolites ucb-42145 (acid), ucb-100406-1 (hydroxy), and ucb-107092-1 (hydroxyacid) • AUC, volume of distribution, and clearance of BRV • Plasma concentrations of concomitant AEDs (PB and PHT) | Section 4.1.1 Primary PK variable The primary PK variable is as follows: Plasma concentrations of BRV following first dose on Day 1 Section 4.1.2 Other PK variables Plasma concentrations of BRV on other occasions Plasma concentrations of BRV metabolites ucb-42145 (acid), ucb-100406-1 (hydroxy), and ucb-107092-1 (hydroxyacid) AUC, volume of distribution, and clearance of BRV Plasma concentrations of concomitant AEDs if administered | PK variables were split into "Primary and Other PK variables" |
| Section 4.2.1 | Title: Key efficacy variables | Title: Secondary efficacy variables | Clarification throughout Section 4.2.1 |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 4.2.1<br>Secondary<br>efficacy<br>variables | A BRV responder is defined as a subject who achieves the following reduction in seizure burden (ENS in minutes per hour) compared to the seizure burden measured during the 2-hour Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment: - At least 80% reduction in nonsevere seizure burden (Nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in any 30-minute timespan) | <ul> <li>A BRV responder is defined as a subject who achieves the following reduction in seizure burden (ENS in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment: <ul> <li>At least 80% reduction in nonsevere seizure burden (Nonsevere seizure burden is defined as ≤50% seizure activity on VEEG in all</li> </ul> </li> </ul> | Updated the definition of a BRV responder |

30-minute timespans)

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 4.2.1<br>Secondary<br>efficacy<br>variables | For this study, an ENS is defined as an EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of 2 hours immediately prior to the first administration of study drug. | For this study, an ENS is defined as an EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug. | For this study, updated the ENS definition |
| Section 4.2.1<br>Secondary<br>efficacy<br>variables | <ul> <li>Absolute and percentage reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period</li> <li>Proportion of BRV responders during the 96-hour Evaluation Period (measured at the end of the 96-hour Evaluation Period)</li> </ul> | <ul> <li>Absolute reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period</li> <li>Percent reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period</li> <li>Proportion of BRV responders at the end of the 96-hour Evaluation Period</li> </ul> | "Absolute and percentage reduction in average seizure burden" were given 2 separate bullet points. Clarified that the proportion of BRV responders "at the end of the 96-hour Evaluation Period". |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 4.2.1<br>Secondary<br>efficacy<br>variables | <ul> <li>Proportion of subjects who are seizure-free by time interval at 3 hours, at 3-hour intervals thereafter through 24 hours, and every 12 hours to 24 hours following the start of the initial BRV treatment</li> <li>Absolute and percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion</li> </ul> | and every 12 hours to 24 hours | Timepoint clarifications and "absolute and percent difference in clinical seizures" were given 2 separate bullet points |


inclusion

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 4.2.2<br>Other<br>efficacy<br>variables | • Absolute and percentage reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment | <ul> <li>Absolute reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, &gt;3 hours to 6 hours, &gt;6 hours to 12 hours, &gt;12 hours to 24 hours, &gt;24 hours to 36 hours, &gt;36 hours to 48 hours, &gt;48 hours to 72 hours, and &gt;72 hours to 96 hours after the start of initial BRV treatment</li> <li>Percent reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, &gt;3 hours to 6 hours, &gt;6 hours to 12 hours, &gt;12 hours to 24 hours, &gt;24 hours to 36 hours, &gt;36 hours to 48 hours, &gt;48 hours to 72 hours, and &gt;72 hours to 96 hours after the</li> </ul> | "Absolute and percentage reduction from Baseline in seizure burden" were given 2 separate bullet points. |


start of initial BRV treatment

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 4.3<br>Safety | The safety variables are as follows: | Section 4.3.1 Secondary safety variable | Separated safety variables into "Secondary" and "Other" |
| variables<br>(Exploratory<br>and | AEs as reported by the<br>Investigator | The secondary safety variable is as follows: | and "Other" |
| Confirmatory<br>Cohorts) | EEG-parameters | AEs as reported by the<br>Investigator | and and |
| | (assessment of sedation) to the end of the Evaluation Period | Section 4.3.2 Other safety variables | |
| | 2 manusin 1 en eu | Change from Baseline in<br>EEG-parameters | Clarification |
| | | (assessment of sedation) to the end of the Evaluation | |
| | | Period (Confirmatory Cohorts only) | |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1<br>Study<br>description | N01349 consists of 2 steps including a comparison with a historical control from literature (MDZ treatment from literature of subjects matched in age and condition) for the evaluation of efficacy. For the Exploratory Cohort (first step), enrolled subjects will receive one or multiple therapeutic doses or continuous infusion of MDZ (dose and dosing frequency of MDZ are at the discretion of the Investigator) prior to receiving BRV. | N01349 consists of 2 steps including a comparison with a historical control group (matched in age and condition) treated with AEDs comparable SOC and diagnostic methods from literature will be used for the evaluation of efficacy. For the Exploratory Cohort (first step), enrolled subjects will receive one or more AEDs for the treatment of ENS per SOC (first-line, second-line, or subsequent treatment; choice of treatment, dose, and dosing frequency are at the discretion of the Investigator) prior to receiving BRV. | Historical control changed from "MDZ" to "one or more AED treatments" |
| Section 5.1<br>Study<br>description | Removed reference to N01266 | Not applicable | Reference to N01266 removed since this study will be closed before the last N01349 subject was able to participate in that study for 3 years. |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1<br>Study<br>description | Interpretation of the VEEGs will be done by local readers but may be supported by the blinded central reader, as needed. Subjects will be evaluated with VEEG monitoring at least during the Baseline, Evaluation, and Down-Titration (Confirmatory Cohorts only) Periods. | Interpretation of VEEGs recorded for the Confirmatory Cohorts will be done by local readers but may be supported by the blinded central reader, as needed. Subjects assigned to the Confirmatory Cohorts will be evaluated with VEEG monitoring at least during the Baseline, Evaluation, and Down-Titration Period. | Clarification Of and any extensions |
| Section 5.1<br>Study<br>description | However, every effort should be made to avoid VEEG interruption of the 2-hour Baseline VEEG and during the first 3 hours after the start of the initial BRV administration for the Confirmatory Cohort. | However, every effort should be made to avoid VEEG interruption of the Baseline VEEG and during the first 3 hours after the start of the initial BRV administration. | Clarification |
| Section 5.1<br>Study<br>description | The schedule of assessments during the BRV Extension, Down-Titration, and Safety Follow-Up Periods for both the Exploratory and Confirmatory Cohorts are presented in Table 5-3 | The schedule of assessments during the BRV Extension, Down-Titration (Confirmatory Cohorts only), and Safety Follow-Up Periods for both the Exploratory and Confirmatory Cohorts are presented in Table 5-3. | Clarification |

| UCB<br>Clinical Study Pro | otocol | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|---|
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| Section 5.1.1 | For the Exploratory Cohort, at | For the Exploratory Cohort, at | PB no longer required as first line treatment |

enrolled and dosed with one or multiple therapeutic doses of MDZ (dose and dosing frequency of MDZ are at the discretion of the Investigator). Phenobarbital treatment must be discontinued prior to entering the Evaluation Period. Approximately 3 hours after the initiation of MDZ dosing, an initial low dose of BRV administered according to the (0.5mg/kg [bid]) will be standard of care. Treatment with MDZ will continue in parallel with BRV treatment. After the Exploratory Cohort completes the study, a PK and safety data review will be performed by the

least 6 subjects who do not have

receiving 1 to 3 doses of PB (PB

treatment may have started prior to the subject's admission into the

40mg/kg; dosing regimen at the

Investigator's discretion) will be

adequate seizure control after

study site; total therapeutic

administered dose of 20 to

For the Exploratory Cohort, at least 6 subjects who do not have adequate seizure control after they received one or more AEDs per SOC for the treatment of ENS (first-line, second-line, or subsequent treatment, which may have started prior to the subject's admission into the study site; choice of treatment, dose, and dosing regimen at the Investigator's discretion) will be enrolled. The AED treatment per SOC can be continued when BRV dosing is initiated. Alternatively, another AED treatment (choice of treatment, dose, and dosing regimen at the Investigator's discretion) must be initiated and continue in parallel with BRV treatment.

At any time after AED treatment per SOC for the treatment of ENS (first-line, second-line, or subsequent treatment) was initiated, an initial low dose of BRV (0.5mg/kg [bid]) will be administered at the Investigator's discretion. After the Exploratory Cohort completes the study, a PK

PB no longer required as first line treatment prior to BRV. Historical control changed from "MDZ" to "one or more AED treatments". Clarification that enrollment will be put on hold during the first DMC


**Exploratory** 

Cohort


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | Data Monitoring Committee (DMC). | and safety data review will be performed by the DMC. During the review of data from the Exploratory Cohort, the enrollment of subjects will be on hold. | anyextensions or |
| Section 5.1.1<br>Exploratory<br>Cohort | Screening Period: from<br>signing and dating of the<br>written Informed Consent<br>form (ICF) up to Cohort<br>Assignment. | Screening Period: from signing and dating of the written ICF up to initiation of the first BRV dose. | For consistency, "Cohort Assignment" changed globally to "up to initiation of the first BRV dose". |
| Section 5.1.1<br>Exploratory<br>Cohort | The Screening Period is up to 36 hours prior to the first administration of MDZ (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of MDZ). The PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the study site. - Baseline Period (included in the Screening Period): 2 hours immediately prior to the start of MDZ infusion. The occurrence | The Screening Period starts up to 36 hours prior to the first administration of BRV. Phenobarbital, MDZ, PHT, LEV, or LDC may have been administered prior to the subject's enrollment into the study and/or at a location other than the study site. Subjects will enter the Evaluation Period and start BRV treatment as soon as the occurrence of ENS per inclusion criterion 2a is confirmed by the Investigator based on local EEG. | Two-hour Baseline EEG and 48-hour VEEG removed from the Exploratory Cohort; required ENS to be confirmed by the Investigator via local EEG |
| Confidential | Chuent | | |

| | of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical | OP Tion application | and any extensions of ve |
|---|---|---|---|
| | (eg, ability for immediate cloud-based central review) can be used as part of the Baseline assessment VEEG. | PUBLIC Contrain | |
| Confidential | Iment cannot be used to support a | Rey components of amended text Copy and the state of the | |

| Evaluation Period (in | Evaluation Period | Treatment with "MDZ only" during the |
|---|---|---|
| total, 51 hours: 3 hours for the evaluation of MDZ and 48 hours for the evaluation of BRV): The first MDZ infusion marks the starting point of the Evaluation Period. Subjects will receive iv MDZ (one or multiple therapeutic doses or continuous infusion; MDZ dose and dosing frequency are at the discretion of the Investigator). Three hours after the initial dose of MDZ, a low dose of BRV (0.5mg/kg) will be administered as an approximately 15-minute iv infusion; additional 3 doses of BRV(0.5mg/kg) can be administered every 12 hours for 48 hours (at the discretion of the Investigator). | (48 hours): The first BRV infusion marks the starting point of the Evaluation Period. At any time after AED treatment per SOC for the treatment of ENS (first-line, second-line, or subsequent treatment) was initiated, a low dose of BRV (0.5mg/kg) will be administered as an approximately 15-minute iv infusion; additional 3 doses of BRV(0.5mg/kg) can be administered every 12 hours for 48 hours (at the discretion of the Investigator). The AED treatment per SOC can be continued when BRV dosing is initiated. Otherwise, another AED treatment (choice of treatment, dose, and dosing regimen at the Investigator's discretion) must be initiated and continue in parallel with BRV treatment. | first 3 hours of the Evaluation Period removed from the Confirmatory Cohort; duration of the Evaluation Period hence shortened from 51 to 48 hour. Historical control changed from "MDZ" to "one or more AED treatments". Other updates for clarification purposes. |
| S. | | |
| | approximately 15-minute iv infusion; additional 3 doses of BRV(0.5mg/kg) can be administered every 12 hours for 48 hours (at the discretion of the Investigator). | approximately 15-minute iv infusion; additional 3 doses of BRV(0.5mg/kg) can be administered every 12 hours for 48 hours (at the discretion of the Investigator) The discretion of the Investigator is discretion of the Investigator is discretion of the Investigator is discretion in must be initiated and continue in parallel with |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.1.2<br>Confirmatory<br>Cohorts | A total of at least 36 subjects without adequate seizure control after receiving 1 to 3 doses of PB (PB treatment may have started prior to the subject's admission into the study site; total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion) will enter the Confirmatory Cohorts. Phenobarbital treatment must be discontinued prior to entering the Evaluation Period. | A total of at least 36 subjects without adequate seizure control after receiving one or more of the following AEDs prior to or at the time of enrollment: PB, MDZ, PHT, LEV (≤60mg/kg/day), or LDC (first-line, second-line, or subsequent treatment, which may have started prior to the subject's admission into the study site; dose and dosing regimen at the Investigator's discretion) will enter the Confirmatory Cohorts. The AED treatment can be continued if the subject is on a stable dose for at least 1 hour at the time the first BRV infusion is initiated. | Phenobarbital no longer required as first line treatment prior to BRV; replaced by "one or more of the following AEDs: PB, MDZ, PHT, LEV (≤60mg/kg/day) or LDC (first-line, second-line or subsequent treatment; dose and dosing at the Investigator's discretion)" for the Confirmatory Cohorts. Other edits for clarification purposes. |
| Section 5.1.2<br>Confirmatory<br>Cohorts | Screening Period: from signing and dating of the written ICF up to Cohort Assignment. • The Screening Period is up to 36 hours prior to the first administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first administration of BRV). The | Screening Period: from signing and dating of the written ICF up to initiation of the first BRV dose. • The Screening Period starts up to 36 hours prior to the first administration of BRV. Phenobarbital, MDZ, PHT, LEV (≤ 60mg/kg/day), or LDC may have been administered prior to the subject's enrollment into the | Clarified to define Baseline Period as part<br>of Screening Period. Definition of status<br>epilepticus for neonates enrolled into this<br>study was added |
| Confidential | administration of BRV (depending on the number of PB doses and time between PB doses and the interval between PB treatment and first | administration of BRV. Phenobarbital, MDZ, PHT, LEV (≤ 60mg/kg/day), or LDC may have been administered prior to | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | PB treatment may have been administered prior to the subject's enrollment in the study and/or at a location other than the study site. • Baseline Period (included in the Screening Period): 2 hours immediately prior to the start of BRV infusion. The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. | study and/or at a location other than the study site. Baseline Period (included in the Screening Period): For subjects with intermittent ENS: at least 1 hour prior to entering the Evaluation Period For subjects in status epilepticus: up to 30 minutes prior to entering the Evaluation Period. At least 15 minutes of continuous seizures, or 50% of cumulative seizure activity during a 30-minute interval are to be confirmed on EEG before | and any extensions of |
| nfidential | ocument co | | |
| This | | | |

| | | | , S |
|---|---|---|---|
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| | | dilution of BRV solution for iv infusion), even if the required EEG recording is not completed by that time. | ad any extensions or s |
| | | • Status epilepticus in neonates for the purpose of this study is defined as follows: | and any or |
| | | o 15 minutes of continuous or cumulative electrographic or | |
| | | electroclinical<br>seizure within 30<br>minutes | |
| | | The occurrence of ENS during the Baseline Period must be confirmed either by the local or | |

central VEEG reader prior to BRV

administration.

| Section | | | alio |
|---|---|---|---|
| Impacted | Key components of previous text | Key components of amended text | Rationale |
| Section 5.1.3 | The maximum study duration per | The maximum study duration per | Clarification |
| Study | subject will be up to 75 days | subject will be up to 75 days | 25 |
| duration per | (Screening Period, Baseline | (Screening Period [including | sio' |
| subject | Period, Evaluation Period, BRV | Baseline Period (Confirmatory | Clarification of |
| 3 | Extension Period, Down-Titration | Cohorts only)], Evaluation Period, | et |
| | Period, and Safety Follow-Up | BRV Extension Period, | the state of the s |
| | Period). The individual study | Down-Titration Period | 72 |
| | duration will be shorter | [Confirmatory Cohorts only], and | alle |
| | depending on the type of cohort | Safety Follow-Up Period). The | |
| | to which subjects will be | individual study duration will be | |
| | assigned, the age at enrollment, | shorter depending on the type of | |
| | and the decision to enter into the | cohort to which subjects will be | |
| | BRV Extension Period. | assigned, the age at enrollment, | |
| | | and the decision to enter the BRV | |
| | | Extension Period. | |
| Table 5-1 | Column heading 2: | Column heading 2: | Updated to reflect changes throughout |
| Schedule of | -36h to -2h | -36h to 0h | protocol |
| assessments - | Column Heading 3: | Column heading 3: | |
| Screening | Baseline Period | Timepoint immediately before first | |
| and | MDZ | BRV administration | |
| Evaluation | -2h to 0h | 4 | |
| Periods | × | | |
| (Exploratory | | | |
| Cohort) | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Table 5-1 Schedule of assessments - Screening and Evaluation Periods (Exploratory Cohort) | Not applicable | Time point immediately before first BRV administration: Vital signs Physical and neurological examination Sarnat scale for subjects with HIE Body weight Added the following to -36h to 0h: Primary cause of seizure Psychometric parameters: N-PASS and EEG-parameters | Updates based on updates made throughout the protocol |
| Table 5-1 Schedule of assessments - Screening and Evaluation Periods (Exploratory Cohort) | PB infusion VEEG-removed AEDs-removed AED PK sample | AED PK sample (only when PB and PTH are used) | Change as reflected throughout protocol |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Table 5-1 | Footnote a | Footnote a | Change as reflected throughout protocol |
| Schedule of | Screening Period is from signing and dating of the written ICF up | Screening Period is from signing and dating of the written ICF up to | Change as reflected throughout protocol |
| assessments - Screening | to Cohort Assignment. | initiation of the first BRV dose. | elisi |
| and | Footnote c | Footnote c | O. T. |
| Evaluation | The occurrence of ENS during | The occurrence of ENS prior to | M |
| Periods | the 2-hour Baseline Period must | entering the Evaluation Period | 200 |
| (Exploratory | be confirmed either by the local | minute of committee of the recur | al. |
| Cohort) | or central VEEG reader prior to drug administration. Preferably, | VEEG reader prior to initial BRV administration. | |
| | the central VEEG reader should | administration. | |
| | confirm the required ENS. | 1 200 | |
| | Footnote d | Footnote d | |
| | Measurement of body weight is | Measurement of body weight is | |
| | optional at 24 and 48 hours. | mandatory prior to BRV treatment | |
| | Dosage of BRV during the | and optional at 24 and 48 hours. | |
| | Evaluation Period will be based | Dosage of BRV during the | |
| | on the subject's weight measured prior to the start of the first BRV | Evaluation Period will be based on the subject's weight measured | |
| | administration. However, dosage | prior to the start of the first BRV | |
| | calculation can be adjusted to a | administration. However, dosage | |
| | more recent weight measurement, | calculation can be adjusted to a | |
| | upon discretion of the | more recent weight measurement, | |
| | Investigator, if weight is | upon discretion of the Investigator, | |
| | measured during the Evaluation | if weight is measured during the | |
| | Period. | Evaluation Period. | |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Table 5-2 Schedule of assessments - Screening and Evaluation Periods (Confirmatory Cohorts) | | Column 2: -36h to up to -1h Column 3: Up to -1h to 0h | Change as reflected throughout protocol |
| Table 5-2<br>Schedule of<br>assessments -<br>Screening and<br>Evaluation<br>Periods<br>(Confirmatory<br>Cohorts) | | AED treatment (PB, MDZ, PHT, LEV [≤60mg/kg/day], or LDC) <sup>n</sup> Assessment to be completed during the Screening Period (both visits) and at all timepoints after 6h during the Evaluation Period AED PK sample (only when PB and PHT are used) | Change as reflected throughout protocol |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Table 5-2 Schedule of assessments - Screening and Evaluation Periods (Confirmatory Cohorts) | Footnote a: Screening Period is from signing and dating of the written ICF up to Cohort Assignment. Not applicable | Footnote a: Screening Period is from signing and dating of the written ICF up to initiation of the first BRV dose. Footnote b added: The duration of the Baseline EEG depends on seizure activity. Subjects with intermittent seizures will enter the Evaluation Period based on at least 1 hour of EEG recording. Subjects in status epilepticus will enter the Evaluation Period based on up to 30 minutes of EEG recording, ie, as soon as 15 minutes of continuous seizures or 50% of cumulative seizure activity is confirmed on EEG. Subsequent footnotes were | Change as reflected throughout protocol |
| Confidential | Footnote d: The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. | re-alphabetized. Footnote e: The occurrence of ENS during the Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.3<br>Schematic | Figure 5-1, Figure 5-2, Figure 5-3, and Figure 5-4 | Figure 5-1, Figure 5-2, Figure 5-3, and Figure 5-4 | All figures updated to reflect protocol changes |
| diagrams | s, and rigure s | and Figure 3 | risioni |
| Section 5.4.1 | Thus, study N01349 was | Thus, study N01349 was designed | PB no longer required as first line treatment |
| Rationale for | designed to include PB as the first | for a flexible treatment of ENS, | prior to BRV |
| study design | line of treatment, and only those | and only those subjects who do not | ad all |
| | subjects who do not have | have adequate seizure control with | 210 |
| | adequate seizure control with PB | previous AED treatment will be | 0. |
| | will be permitted to continue in | permitted to continue in the study | |
| | the study | ica | |
| Section 5.4.1 | Thus, only neonates with an age | At enrollment, subjects must be at | Age at enrollment has been modified |
| Rationale for | at birth of 34 weeks to less than | least 34 weeks of CGA. In | |
| the study | 42 weeks of GA (and up to | addition, term neonates up to | |
| design | 28 days of postnatal age at the | 27 days of PNA and preterm | |
| | time of enrollment) with repeated | neonates up to 40 weeks of PMA | |
| | neonatal seizures (assessed by | and 27 days of PNA can be | |
| | VEEG) will be enrolled in | enrolled. | |
| 1 | N01340 | | |


| Section | | | id dio |
|---|---|---|---|
| Impacted | Key components of previous text | <b>Key components of amended text</b> | Rationale |
| Section 6.1 | 2a. Confirmation on VEEG of | 2a. Confirmation on VEEG of | Based on agency recommendation, the |
| Inclusion | ≥2 minutes of cumulative ENS or | ≥2 minutes of cumulative ENS or | 2-hour Baseline EEG has been removed. |
| Criteria | ≥3 identifiable ENS within the | ≥3 identifiable ENS prior to | ėjo, |
| | 2 hours prior to entering the | entering the Evaluation Period | * Cl |
| | Evaluation Period (ENS is | (ENS is defined as a seizure | 2-hour Baseline EEG has been removed. |
| | defined as a seizure lasting for at | lasting for at least 10 seconds on | to |
| | least 10 seconds on VEEG), | VEEG), despite receiving previous | 700 |
| | despite receiving PB (total | AED treatment for the treatment of | Dille |
| | therapeutic administered dose of | electroencephalographic seizures. | |
| | 20 to 40mg/kg) for the treatment | alle | |
| | of repeated seizures. | 7 applic | |
| | The occurrence of ENS during | The occurrence of ENS during an | For clarification 2-hour period was replaced |
| | the 2-hour period must be | up to 1-hour period must be | with up to 1-hour period |
| | confirmed either by the local or | confirmed either by the local or | - |
| | central VEEG reader prior to drug | central VEEG reader prior to drug | |
| | administration. Preferably, the | administration. Preferably, the | |
| | central VEEG reader should | central VEEG reader should | |
| | confirm the required ENS. | confirm the required ENS | |
| Section 6.1 | 3. Subject is male or female, with | 3. Subject is male or female and | Based on feedback from Investigators, the |
| Inclusion | an age at birth of 34 weeks to less | must be at least 34 weeks of CGA. | age of subjects allowed to participate in the |
| Criteria | than 42 weeks of GA and up to $\sqrt{2}$ | In addition, term neonates up to | study will be extended to help with |
| | 28 days of postnatal age at the | 27 days of PNA and preterm | enrollment. |
| | time of enrollment. | neonates up to 40 weeks of PMA | |
| | | and 27 days of PNA can be | |
| | | enrolled | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 6.2<br>Exclusion<br>Criteria | 1a. Subject received AED treatment (other than the required 1 to 3 doses of PB [total therapeutic administered dose of 20 to 40mg/kg] for the treatment of repeated seizures) prior to entering the Evaluation Period. | 1a. Subject receiving AED treatment other than PB, MDZ, PHT, LEV (≤60mg/kg/day), or LDC for the treatment of seizures prior to or at the time of enrollment (Confirmatory Cohorts only). | Phenobarbital no longer required as first line treatment prior to BRV |
| Section 6.2<br>Exclusion<br>Criteria | 2. Subject with seizures responding to PB (total therapeutic administered dose of 20 to 40mg/kg), pyridoxine treatment, or correction of metabolic disturbances (hypoglycemia, hypomagnesemia or hypocalcemia). | 2. Subject with seizures responding to previous AED treatment immediately prior to BRV treatment, pyridoxine treatment, or correction of metabolic disturbances (hypoglycemia, hypomagnesemia, or hypocalcemia). | Phenobarbital no longer required as first line treatment prior to BRV |
| Section 7.1<br>Description of<br>investigational<br>medicinal<br>products | Tartifer actains on the manaring or | Refer to the IMP Handling Manual for further details on the handling of BRV. | Clarification |
| Section 7.1<br>Description of<br>investigational<br>medicinal<br>products | | After the completion of the study, BRV treatment per SOC may be continued as prescribed but will not be provided by the Sponsor. | Clarification |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.2<br>Treatments to<br>be<br>administered | Subjects in the Exploratory Cohort will be dosed with iv MDZ (dosing and dosing frequency of MDZ are at the discretion of the Investigator). Three hours after the start of MDZ infusion, BRV dosing (0.5mg/kg bid) will start according to the standard of care. Treatment with MDZ will continue in parallel with BRV treatment. | Subjects in the Exploratory Cohort will be dosed with BRV (0.5mg/kg bid) according to the sites standard procedures. Treatment with AEDs per SOC (first-line, second-line, or subsequent treatment) will continue in parallel with BRV treatment. | Historical control changed from "MDZ". |
| Section 7.2<br>Treatments to<br>be<br>administered | Not applicable | Treatment with previous AEDs (PB, MDZ, PHT, LEV [≤60mg/kg/day], or LDC) is permitted to continue if the subject is on a stable dose from 1 hour prior to initiation of the BRV treatment. | Clarification |
| Section 7.3 Packaging | Commercial MDZ will be used for this study and will not be provided by the Sponsor. | Other AED treatments will be used for this study and will not be provided or covered by the Sponsor. | Historical control changed from "MDZ". |
| Confidential | Schuent cannot be | | |
| This | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.5 Handling and storage requirements | Appropriate storage conditions must be ensured either by controlling the temperature (eg, room, refrigeration unit) or by completing a temperature log in accordance with local requirements on a regular basis (eg, once a week), showing actual minimum/maximum temperatures reached over the time interval. | Appropriate storage conditions must be ensured either by controlling the temperature (eg, room, refrigeration unit) or by completing a temperature log in accordance with local requirements on a regular basis (eg, once per working day), showing actual minimum/maximum temperatures reached over the time interval. | Clarification of and any extensions |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.8.1 Permitted concomitant treatments (medications and therapies) | Concomitant treatment with AEDs is permitted as follows: Prior to first BRV administration: | For the Exploratory Cohort, concomitant treatment with AEDs is permitted at any time. For the Confirmatory Cohorts, concomitant treatment with AEDs is permitted to continue in parallel with BRV treatment if subjects are on a stable dose from 1 hour prior to initiation of BRV treatment. Changes to concomitant AEDs are permitted from 3 hours onward following first BRV administration. | PB is no longer required as first-line treatment prior to BRV; historical control changed from MDZ. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.8.2<br>Prohibited<br>concomitant<br>treatments<br>(medications<br>and therapies) | receive treatments for neonatal seizures (other than the specified PB doses and MDZ) prior to the first BRV administration. | For the Confirmatory Cohorts, subjects will not be permitted to change concomitant treatment for neonatal seizures for the first 3 hours after the first BRV administration. The initiation of LEV treatment after the first time BRV is introduced is prohibited throughout the study for the Confirmatory Cohorts. | Clarification and any extensions and any extensions |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| 7.8.3 Rescue medication | Rescue medication in this study is considered as any treatment with AEDs. Rescue medication can be given at any time if considered necessary by the Investigator. However, during the Evaluation Period rescue medication should not be administered – if possible – in the following time frames: • Prior to BRV dosing for the Exploratory Cohort (except for MDZ as scheduled in the Protocol). • During the first 3 hours after the initial dose of BRV for the Confirmatory Cohorts. If this occurs, subjects will be considered BRV nonresponders. | Any treatment initiation with a new AED, or any increase of dose or frequency of an existing concomitant AED for the treatment of seizures during the Evaluation Period is considered rescue treatment. Rescue medication can be given at any time if considered necessary by the Investigator. However, during the Evaluation Period rescue medication should not be administered if possible in the following time frames: • During the first 3 hours after the initial dose of BRV for the Confirmatory Cohorts. If this occurs, subjects will be considered BRV nonresponders for the evaluation of the main efficacy variable. | Clarification of and any extensions of and any extensions |
| Section 8.1.1<br>Screening<br>Period | The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal representative(s) of the subject to the end of the Baseline Period. Any AEs, AEDs, | The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal representative(s) up to initiation of the first BRV dose. Any AEs, AEDs, concomitant | Text has been updated to reflect the changes to the study schedule of assessments. Other text changes were also made to provide consistent language throughout the protocol. Section heading 8.1.2 Baseline Period was deleted and text |
| Confidential | written ICF by the parent(s) or legal representative(s) of the subject to the end of the Baseline Period. Any AEs, AEDs, | | |

| · | | | |
|---|---|---|---|
| Section | | | n i dill |
| Impacted | <b>Key components of previous text</b> | Key components of amended text | Rationale |
| | concomitant medications, and | medications, and medical | merged with Section 8.1.1. All subsequent |
| | medical procedures will be | procedures will be collected after | section headings were updated. |
| | collected after the ICF is signed. | the ICF is signed. The subject's | sio. |
| | The subject's eligibility to | eligibility to participate in this | *eile |
| | participate in this study will be | study will be assessed. The subject | et |
| | assessed. The subject | identification card will be | to |
| | identification card will be | dispensed. | section headings were updated. |
| | dispensed. | The Screening Period starts up to | arie |
| | The Screening Period is up to 36 | 36 hours prior to the first | |
| | hours prior to the first | administration of BRV. | |
| | administration of MDZ | Phenobarbital, MDZ, PHT, REV | |
| | (depending on the number of PB | (≤ 60mg/kg/day), or LDC may | |
| | doses and time between PB doses | have been administered prior to | |
| | and the interval between PB | the subject's enrollment into the | |
| | treatment and first administration | study and/or at a location other | |
| | of MDZ). Body weight | than the study site. | |
| | measurements can be taken | 7 0 | |
| | between 36 hours and 2 hours for | Subjects will enter the Evaluation | |
| | the determination of PB | Period and start BRV treatment as | |
| | dosage (mg/kg). The PB | soon as the occurrence of ENS per | |
| | treatment may have started prior | inclusion criterion 2a is confirmed | |
| | to the subject's admission to the | by the Investigator based on local | |
| | study and/or at a location other | EEG. | |
| | than the study site but should be | The following assessments will be | |
| | completed prior to the 2-hour | performed immediately before the | |
| | Baseline Period. | first administration of BRV is | |
| | - Walter Tario and Tario | initiated: | |
| | Baseline Period. | Verification of | |
| | 10, | inclusion/exclusion criteria. | |
| | cain. | Confirmation on VEEG of | |
| | , O | | |

Confidential document

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | At the determination of the Investigator, subjects achieving adequate seizure control after initial PB treatment (total therapeutic administered dose of 20 to 40mg/kg; dosing regimen at the Investigator's discretion) will be considered PB responders. Those subjects will be classified as screen failures and will not be assigned to BRV treatment | <ul> <li>Vital signs (blood pressure, pulse rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature)</li> <li>Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity)</li> </ul> | and any extensions of |
| Confidential | 30cument cannot | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | liver enzymes, and endocrinology) | ans of |
| | | • Thompson score (for subjects with HIE) | Rationale value of value and any extensions of value and any extension and any extensions of value and any extensions of value and any extensions of value and any extensions of value and any extensi |
| | | Mechanical ventilation | M |
| | | AEs as reported by the Investigator | and o |
| | | Recording of AEDs,<br>concomitant medications, and<br>medical procedures | |
| | | Laboratory measurements will be performed by local laboratories | |
| | | unless historical data is available.<br>Historical safety laboratory | |
| | | assessments, previously collected as standard of care, may be | |
| | | accepted from referring hospitals | |
| | | as measurement prior to first use | |
| | X. | of BRV if performed 36 hours prior to the start of the Evaluation | |
| | 2801 | Period. In this case, test results | |
| | SILL. | will be considered medical history. | |
| | 20 | Prior laboratory assessment results | |
| | Les Control of the Co | should be available and verified | |
| | X Ve V | prior to initiation of the first BRV infusion. | |
| | camot be used to support of | At the determination of the Investigator, subjects achieving | |


| 0 |
|------------|
| May 2021 |
| 1VIay 2021 |
| N01349 |
| 1.010.7 |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | adequate seizure control following | ok . |
| | | AED treatment per SOC will be | 1,5 |
| | | considered AED responders. | sio' |
| | | Those subjects will be classified as | *ells |
| | | screen failures and will not be | et |
| | | assigned to BRV treatment. | (i) |


| Section 8.1.2 | The Baseline Period is included | Not applicable | This section heading was deleted, and text |
|---|---|---|---|
| Baseline<br>Period | in the Screening Period; the period begins 2 hours before and ends at the initiation of the MDZ infusion. The occurrence of ENS during the 2-hour Baseline Period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS. Video-EEGs that are acquired per standard of care prior to consenting and meet study-specific technical and quality requirements (eg, ability for immediate cloud-based central review) can be used as part of the Baseline assessment VEEG. The following assessments will be performed during the Baseline Period: • Verification of inclusion/exclusion criteria. Confirmation on VEEG of ≥2 minutes of cumulative ENS or ≥3 identifiable ENS within the 2 hours prior to entering the Evaluation Period (ENS is defined as a seizure | Not applicable COPT and application Not applicable Not applicable | merged into Section 8.1.7. Subsequent headings were renumbered |
| Confidential | (ENS is defined as a seizure | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| • | on VEEG), despite PB treatment prior to Baseline | V X | ans of the |
| | Demographic data Medical<br>history (including Apgar<br>score) | | Rationale Jan's Of Jan's and any extensions of Jan's Of J |
| | Vital signs (blood pressure, pulse rate, respiratory rate, oxygen saturation [pulse oximetry] including apneas, and body temperature) | Oplication | andair |
| | Physical and neurological examination (Sarnat scale for subjects with HIE; physical examination will include a check for the presence of skin rash and skin hypersensitivity) | Nymarketing authorization application | |
| | • Length | Mali | |
| | Body weight | A Company of the Comp | |
| | • Head circumference (Baseline measurement should be taken within 7 days prior to drug administration, or at birth for subjects ≤7 days old) | | |
| | Primary cause of seizure<br>(HIE, hemorrhage, or<br>infarction; CNS | | |
| | cent | | |
| Confidential | chu. | | |
| (his | | - | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | malformations; CNS infections; undetermined causes) | | asions of |
| | • N-PASS and EEG parameters for the assessment of sedation | | detiel. |
| | • Video-EEG | | Par. |
| | Heart rate monitoring | ~ | |
| | • Safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology) | Key components of amended text COPT and application application application authorization application | |
| | • Thompson score (for subjects with HIE) | .BLL "horizati | |
| | Mechanical ventilation | box any | |
| | • AEs as reported by the Investigator | aiketines | |
| | Baseline laboratory measurements will be performed by local laboratories unless historical data is available. Historical safety laboratory assessments, previously collected as standard of care, may be accepted from referring hospitals as Baseline measurement if performed 36 hours prior to the start of the Evaluation Period. In | B. Carrier | |

Confidential documer


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | this case, test results will be considered medical history. Prior laboratory assessment results should already be available at Baseline and verified prior to initiation of the MDZ infusion. | | anyetiensions or |
| Section 8.1.4<br>Evaluation<br>Period | The first MDZ infusion marks the starting point of the Evaluation Period. The Evaluation Period will last for 51 hours in total (3 hours for the evaluation of MDZ and 48 hours for the evaluation of BRV). After the enrollment of subjects, the weight of the subject will be measured and MDZ will be administered. The following assessments will be performed at the start of and 3 hours after the initial MDZ administration: Vital signs (blood pressure, pulse rate, respiratory rate, oxygen saturation [pulse oximetry] including apneas, and body temperature); only at the start of MDZ administration Video-EEG | Section 8.1.3 Evaluation Period The first BRV infusion marks the starting point of the 48-hour Evaluation Period. An initial iv dose of BRV (0.5mg/kg) will be administered as an approximately 15-minute infusion. At the discretion of the Investigator, 3 additional iv BRV doses can be administered, up to a total of 4 iv BRV doses (0.5mg/kg bid) during the 48-hour BRV Evaluation Period. The following assessments will be performed after the end of the first BRV infusion: | Text has been updated to reflect the changes to the study schedule of assessments. Other text changes were also made to provide consistent language throughout the protocol. |
| Confidential | CHUEUT | | |
| \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Impacted | Heart rate monitoring | They components of unionaed text | O. A. |
| | AEs as reported by the<br>Investigator | | ansions |
| | AEDs, concomitant<br>medications, and medical<br>procedures | | ad any exte |
| | • Infusion site reaction monitoring | Oijo | |
| | 7 | Key components of amended text COPT and application a | |
| | The following assessments will be performed after the first BRV administration: | | |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section<br>8.1.4.2<br>Extension<br>Period Visit 2 | The EPV2 will be performed on the same day when the subject enters the long-term study. The following assessments will be performed: | The EPV2 should be performed on the same day when the subject enters the long-term study. The following assessments will be performed: | Clarification |
| Section 8.2.1<br>Screening<br>Period | The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal representative(s) of the subject to the end of the Baseline Period. Any AEs, AEDs, concomitant medications, and medical procedures will be collected after the ICF is signed. The subject's eligibility to participate in this study will be assessed. The subject identification card will be dispensed. | The Screening Period will be from the signing and dating of the written ICF by the parent(s) or legal representative(s) of the subject up to initiation of the first BRV dose. Any AEs, AEDs, concomitant medications, and medical procedures will be collected after the ICF is signed. The subject's eligibility to participate in this study will be assessed. The subject identification card will be dispensed. The Screening Period starts up to 36 hours prior to the first administration of BRV. The treatment with one or more of the following AEDs prior to or at the time of enrollment: PB, MDZ, PHT, LEV (≤60mg/kg/day), or LDC (first-line, second-line, or subsequent treatment; choice of treatment, dose, and dosing | Text has been updated to reflect the changes to the study schedule of assessments. Other text changes were also made to provide consistent language throughout the protocol. |
| This | , | - | |

| Period is up to 36 the first of BRV the number of PB between PB doses al between PB first administration y weight can be taken urs and 2 hours for ion of PB t). The PB have started prior s enrollment in the t a location other | regimen at the Investigator's discretion) may have started prior to the subject's enrollment in the study and/or at a location other than the study site. At the determination of the Investigator, subjects achieving adequate seizure control following any of the following AEDs: PB, MDZ, PHT, LEV (≤60mg/kg/day), or LDC will be considered AED responders. | and any extensions of you |
|---|---|---|
| site but should be or to the 2-hour d. nation of the ubjects achieving are control after ment (total ministered dose of gidosing regimen at or's discretion) will PB responders. | or LDC will be considered AED responders. | |
| Period will<br>nediately prior to<br>V infusion. | Section 8.2.1.1 Baseline Period The Baseline Period will be up to | Section heading numbering changed<br>because Baseline is part of Screening. Text<br>has been updated to reflect the changes to<br>the study schedule of assessments. Other |
| P | B responders. eriod will ediately prior to | B responders. Period will Section 8.2.1.1 Baseline Period ediately prior to |

| Section | IV | Warrange and a farmer deal to at | Defined viality |
|---|---|---|---|
| Impacted | Key components of previous text | Key components of amended text | Rationale |
| | | 1 hour immediately prior to the | text changes were also made to provide |
| | | start of initial BRV infusion and | consistent language throughout the |
| | | depend on seizure activity: | protocol. |
| | | - For subjects with intermittent | *ell_ |
| | | ENS: at least 1 hour prior to | et |
| | | entering the Evaluation Period | ta |
| | | - For subjects in status epilepticus: | consistent language throughout the protocol. |
| | | up to 30 minutes prior to entering | 3/1° |
| | | the Evaluation Period. At least 15 | |
| | | minutes of continuous seizures, or | |
| | | 50% of cumulative seizure activity | |
| | | during a 30-minute interval are to | |
| | | be confirmed on EEG before the | |
| | | administration of BRV can start. | |
| | | As soon as subjects are considered | |
| | | to be in status epilepticus, steps | |
| | | required for the preparation of the | |
| | | initial BRV infusion can be | |
| | | initiated (eg, assignment of BRV | |
| | | kits through interactive IRT and | |
| | . 2 | the dilution of BRV solution for iv | |
| | | infusion), even if the required | |
| | 100 | EEG recording is not completed | |
| | SV. | by that time. | |
| | The occurrence of ENS during | The occurrence of ENS during the | |
| | the 2-hour Baseline Period must | Baseline Period must be confirmed | |
| | be confirmed either by the local | either by the local or central | |
| | or central VEEG reader prior to | VEEG reader prior to drug | |
| | drug administration. | administration. | |
| | - (N) | | |

Confidential Hocument of

N01349

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | • Verification of | • Verification of | o's |
| | inclusion/exclusion criteria. | inclusion/exclusion criteria. | 15 |
| | Confirmation on VEEG of | Confirmation on VEEG of | extensio" |
| | ≥2 minutes of cumulative | ≥2 minutes of cumulative ENS | *ells |
| | ENS or ≥3 identifiable ENS | or ≥3 identifiable ENS within | et |
| | within the 2 hours prior to | the 1 hour prior to entering the | know h |
| | entering the Evaluation Period | Evaluation Period (ENS is | 9,0 |
| | (ENS is defined as a seizure | defined as a seizure lasting for | all |
| | lasting for at least 10 seconds | at least 10 seconds on VEEG) | |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 8.2.3<br>Evaluation<br>Period | Not applicable | The AED treatment initiated prior to first administration of BRV can be continued if the subject is on a stable dose for at least 1 hour at the time the first BRV infusion is initiated. | Text has been updated to reflect the changes to the study schedule of assessments. Other text changes were also made to provide consistent language throughout the protocol. |
| Section 8.2.4<br>BRV<br>Extension<br>Period | Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study N01266 (see Section 8.2.4.2). If study N01266 is performed outside the N01349 hospital, an interval of up to 3 days between the N01349 EPV2 and N01266 Entry Visit is allowed. | Extension Period Visit 2 will be performed on the same day when the subject enters the long-term study (see Section 8.2.4.2). If the long-term study is performed outside the N01349 hospital, an interval of up to 3 days between the N01349 EPV2 and long-term study Entry Visit is allowed. | Text changes were made to provide consistent language throughout the protocol. |
| Section<br>8.2.4.2<br>Extension<br>Period Visit 2 | This visit will be performed on the same day when the subject enters the long-term study. | This visit should be performed on<br>the same day when the subject<br>enters the long-term study. | Text changes were made to provide consistent language throughout the protocol. |
| Section 10.1 | Title: Assessment of the key efficacy variables | Title: Assessment of secondary efficacy variables (Confirmatory Cohort[s] only) | Text changes were made to provide consistent language throughout the protocol. |
| Section 10.1 | The main efficacy variable is: | The main secondary efficacy variable is: | Text changes were made to provide consistent language throughout the protocol. |
| Confidential | Ment | | |
| Confidential | SC, | | |
| This | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | | A BRV responder is defined as a | Rationale And any extensions of the angle and any extensions o |
| | A BRV responder is defined as a | subject who achieved the | 1,50 |
| | subject who achieved the | following reduction in seizure | si <sup>0</sup> |
| | following reduction in seizure | burden (ENS in minutes per hour) | *ells |
| | burden (ENS in minutes per hour) | without need for rescue | et |
| | compared to the seizure burden | medication, compared to the | (I) |
| | measured during the 2-hour | seizure burden measured during | 20,0 |
| | Baseline Period immediately | | all. |
| | prior to BRV administration, | prior to BRV administration, | |
| | evaluated for a 2-hour period | evaluated for a 2-hour period | |
| | starting 1 hour after the start of | starting 1 hour after the start of | |
| | initial BRV treatment | initial BRV treatment | |
| | | cor ijor. | |
| | | (Nonsevere seizure burden is | |
| | (Nonsevere seizure burden is | defined as ≤50% seizure activity | |
| | defined as ≤50% seizure activity | on VEEG in all 30-minute | |
| | on VEEG in any 30-minute | timespans) | |
| | timespan) | | |
| | | For this study on ENC is defined | |
| | For this study, an ENS is defined | For this study, an ENS is defined as EEG seizure lasting for at least | |
| | as EEG seizure lasting for at least | 10 seconds on VEEG. Baseline | |
| | 10 seconds on VEEG. Baseline | seizure burden is defined as | |
| | seizure burden is defined as | seizure burden is defined as seizure burden measured on the | |
| | seizure burden measured on the | continuous VEEG (total ENS in | |
| | continuous VEEG (total ENS in | minutes per hour) during a period | |
| | minutes per hour) during a period | of up to 1 hour immediately prior | |
| | of 2 hours immediately prior to | to the first administration of study | |
| | the first administration of study | drug. | |
| | drug | | |
| | Jocument Call | | |
| Confidential | cui. | | |

| Key components of previous text For the analysis of the main efficacy variable (Section 4.2.1), subjects that are switched to another AED or have been administered any rescue medication (including BZDs) during the first 3 hours after initiation of BRV treatment will be considered BRV nonresponders. Subjects must not have switched to another AED or used >1 dose of rescue medication (including | For the analysis of the main secondary efficacy variable (Section 4.2.1), subjects who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS during the first 3 hours after initiation of BRV | Rationale and any extensions of and any extensions |
|---|---|---|
| BZDs) following the first 3 hours after initiation of BRV treatment to be considered BRV responders for the analysis of the following key efficacy variables: | treatment will be considered BRV nonresponders. For the analysis of the following secondary efficacy variables, subjects who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS following the first 3 hours after initiation of BRV treatment will be considered BRV responders: • Absolute reduction in average seizure burden measured by continuous VEEG from | |
| ziment | | |
| | after initiation of BRV treatment<br>to be considered BRV responders<br>for the analysis of the following<br>key efficacy variables: | after initiation of BRV treatment to be considered BRV responders for the analysis of the following key efficacy variables: For the analysis of the following secondary efficacy variables, subjects who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS following the first 3 hours after initiation of BRV treatment will be considered BRV responders: |

| Section | | | idio |
|---|---|---|---|
| | reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period Proportion of BRV responders during the 96-hour Evaluation Period (measured at the end of the 96-hour Evaluation Period) | Baseline to the end of the 96-hour Evaluation Period Percent reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period Proportion of BRV responders at the end of the 96-hour Evaluation Period Seizure freedom at the end of the Down-Titration Period Proportion of subjects who are seizure-free by time interval at 3 hours, at 3-hour intervals | Rationale Jakination of Jakination and any extensions of Jakination and any extensions of Jakination and Jakina |
| • | are seizure-free by time interval at 3 hours, at 3-hour intervals thereafter through 24 hours, and every 12 hour to 24 hours following the start of the initial BRV treatment Absolute and percent difference in clinical seizures at the end of the 24-hour Evaluation Period from | thereafter through 24 hours, and every 12 hours to 24 hours following the start of the initial BRV treatment • Absolute difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion | |
| Confidential doci | Inella | | |
| This | | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | Baseline for neonates with motor seizures at the time of inclusion | Percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion | anyextensions or vo |
| Section 10.2<br>Assessment of<br>other efficacy<br>variables | To further evaluate BRV efficacy, a descriptive comparison will be conducted of the main efficacy variable data from N01349 with published responder rates for MDZ (historical control group matched in age and condition) effective for the treatment of neonatal seizures in subjects of similar age (<29 days of postnatal age) and condition (neonatal seizures as noted in N01349 eligibility criteria). A recent study (Weeke et al, 2016) provides response rates for second line MDZ treatment of neonatal seizures in a similar population and with primary endpoints comparable to N01349. | To further evaluate BRV efficacy, a descriptive comparison will be conducted of the main efficacy variable data from N01349 with published responder rates for one or more AED treatments from literature (historical control group matched in age and condition) effective for the treatment of neonatal seizures in subjects of similar age (<29 days of postnatal age) and condition (neonatal seizures as noted in N01349 eligibility criteria). A recent study (Weeke et al, 2016) provides response rates for second line AED treatment of neonatal seizures in a similar population and with primary endpoints comparable to N01349. | Historical control changed from "MDZ" to "one or more AED treatments" |
| Section 10.3<br>Seizure<br>burden | Seizure burden is defined as the total minutes of ENS per hour. Seizure burden information will | Seizure burden is defined as the total minutes of ENS per hour. Seizure burden information will be | Clarification |
| Confidential | CHURCH | | |

| UCB<br>Clinical Study Protocol | | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|---|
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| | be recorded via a continuous | recorded for the Confirmatory | Ol Ol |
| | VEEG. Seizure burden at | Cohorts via a continuous VEEG. | ,5 |
| | Baseline will be evaluated over a | Seizure burden at Baseline will be | si <sup>0</sup> |
| | 2-hour period. | evaluated over a period of at least | exension |
| | | 1 hour (subjects with intermittent | et |
| | | seizures) or up to 30 minutes | tin |
| | | (subjects in status epilepticus). | 70, |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| 11.1.1.1<br>Adverse event | Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the Investigator from the subject's history or the Baseline Period. | Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the Investigator from the subject's history or based on assessments performed prior to the first administration of BRV. | Clarification of and any extensions of and any extensions |
| Section 11.3.3<br>Vital signs | Vital sign measurements, including systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, oxygen saturation (pulse oximetry), and body temperature, should be measured at the study timepoints as described in | Vital sign measurements, including systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate (including apneas), oxygen saturation (pulse oximetry), and body temperature, should be measured at the study timepoints as described in | Text changes were made to provide consistent language throughout the protocol. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 13.1<br>Definition of<br>analysis sets | The Pharmacokinetic Per-Protocol Set will consist of all subjects who provide at least 1 measureable post-Baseline plasma sample (with recorded sampling time) on at least 1 post-Baseline visit with documented study drug intake times. This analysis set will be used for the Exploratory Cohort and the Confirmatory Cohort(s). | The Pharmacokinetic Per-Protocol Set will consist of all subjects who provide at least 1 measurable plasma sample (with recorded sampling time) on at least 1 post-Baseline visit with documented study drug intake times. This analysis set will be used for the Exploratory Cohort and the Confirmatory Cohort(s). | Clarification Or To the Clarification of the Clari |
| | The Full Analysis Set will be used for the analysis of seizure data and will consist of all subjects in the SS who have a minimum of 2 hours of interpretable VEEG data from both the Baseline period and the first 3 hours of the post-Baseline period after initial BRV treatment. | The Full Analysis Set will be used for the analysis of seizure data (efficacy) and will consist of all subjects in the SS who have a minimum of 2 hours of interpretable VEEG data from both the Baseline period and the first 3 hours of the post-Baseline period after initial BRV treatment. | |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| 13.3.1<br>Exploratory<br>Cohort | Based on the plasma samples collected for the Exploratory Cohort, relevant PK parameters including AUC, C <sub>max</sub> , volume of distribution, and clearance, will be estimated using noncompartmental methods. | Based on the plasma samples collected for the Exploratory Cohort, relevant PK parameters including AUC, C <sub>max</sub> , volume of distribution, and clearance, will be estimated using noncompartmental methods, with sub-analysis by concomitant use of hypothermia. | Text changes were made to provide consistent language throughout the protocol. |
| Section 13.5.1 | Title: Analysis of key efficacy variables | Title: Analysis of secondary efficacy variables | Text changes were made to provide consistent language throughout the protocol. |
| Section 13.5.1<br>Analysis of<br>the key<br>efficacy<br>variables | proportion of responders to BRV treatment from Baseline to 3 hours after the initial BRV dose. A BRV responder is defined as a subject who achieves at least 80% reduction in nonsevere seizure burden ("nonsevere" seizure burden being defined as ≤50% seizure activity on VEEG in any 30-minute timespan), or at least 50% reduction in severe seizure burden ("severe" seizure burden being defined as >50% seizure activity on VEEG in any 30-minute timespan) compared to | The main secondary efficacy variable is as follows: • Proportion of responders to BRV treatment from Baseline to 3 hours after the initial BRV dose. A BRV responder is defined as a subject who achieves the following reduction in seizure burden (ENS in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period | Text changes were made to provide consistent language throughout the protocol. |
| Confidential | Chuent | | |

| the scizure burden measured during the 2-hour Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment. Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to ≤30 minutes, >30 to ≤60 minutes, >60 to ≤90 minutes. The main efficacy variable will be analyzed using descriptive statistics. Baseline seizure burden is defined as seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of 2 hours immediately prior to the first administration of BRV. Confidential | Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|---|
| of up to 1 hour immediately prior | | during the 2-hour Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment. Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to ≤30 minutes, >30 to ≤60 minutes, >60 to ≤90 minutes, and >90 to ≤120 minutes. The main efficacy variable will be analyzed using descriptive statistics. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of 2 hours immediately prior to the first administration of BRV. | OR - At least 50% reduction in severe seizure burden (Severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan). Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to ≤30 minutes, >30 to ≤60 minutes, >60 to ≤90 minutes, and >90 to ≤120 minutes. For this study, an ENS is defined as an EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period | and any extensions of |
| | Confidential | 30Climent | | |

| UCB<br>Clinical Study | Protocol | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|---|
| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
| | Subjects with at least 80% | to the first administration of study | Ol . |
| | reduction in nonsevere seizure | drug. | and any extensions or |
| | burden or at least 50% reduction | | ėjo, |
| | in severe seizure burden from | | *ells |
| | Baseline will be categorized as | | et |
| | BRV responders. Subjects who | | to |
| | drop out due to lack of BRV | | 900 |
| | efficacy, are switched over to | | affe |
| | another AED treatment, or are | · | |
| | administered any rescue | · call | |
| | medication (including BZDs) will | olile | |
| | be considered BRV | ot application | |
| | nonresponders. | 70° × 10° | |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 13.5.1<br>Analysis of<br>secondary<br>efficacy<br>variables | <ul> <li>For the Confirmatory Cohorts this means:</li> <li>For the analysis of the main efficacy variable, subjects must not have used any rescue medication (including BZDs) during the first 3 hours after initiation of BRV treatment to be considered BRV responders.</li> <li>For the analysis of the key efficacy variables (other than the main efficacy variable) and other efficacy variables, subjects must not have used &gt;1 dose of rescue medication following the first 3 hours after initiation of BRV treatment to be considered BRV responders. A single dose of short-acting BZD as rescue medication is allowed, but only after 3 hours subsequent to the initiation of treatment with BRV.</li> </ul> | <ul> <li>For the Confirmatory Cohorts this means:</li> <li>For the analysis of the main secondary efficacy variable, subjects must not have used any rescue medication for the treatment of ENS during the first 3 hours after initiation of BRV treatment to be considered BRV responders.</li> <li>For the analysis of the secondary efficacy variables (other than the main secondary efficacy variable) and other efficacy variables, subjects must not have used any rescue medication for the treatment of ENS following the first 3 hours after initiation of BRV treatment to be considered BRV responders.</li> </ul> | Text changes were made to provide consistent language throughout the protocol. |
| Section 13.5.1<br>Analysis of<br>secondary | Descriptive statistics will be presented for the following key efficacy variables: | Descriptive statistics will be presented for the following secondary efficacy variables: | Text changes were made to provide consistent language throughout the protocol. |
| Confidential | CHURENT | | |

| Section | | | |
|---|---|---|---|
| Impacted | <b>Key components of previous text</b> | Key components of amended text | Rationale |
| efficacy<br>variables | <ul> <li>Absolute and percentage reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period</li> <li>Proportion of BRV responders during the 96-hour Evaluation Period (measured at the end of the 96-hour</li> </ul> | <ul> <li>Absolute reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period</li> <li>Percent reduction in average seizure burden measured by continuous VEEG from Baseline to the end of the 96-hour Evaluation Period</li> </ul> | and any extensions of |
| | Absolute and percent difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion | <ul> <li>Proportion of BRV responders at the end of the 96-hour Evaluation Period</li> <li>Absolute difference in clinical seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion</li> <li>Percent difference in clinical</li> </ul> | |
| | inclusion Jead to Support | seizures at the end of the 24-hour Evaluation Period from Baseline for neonates with motor seizures at the time of inclusion | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 13.5.2 Analysis of the other efficacy variables | • Absolute and percentage reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, >3 hours to 6 hours, >6 hours to 12 hours, >12 hours to 24 hours, >24 hours to 36 hours, >36 hours to 48 hours, >48 hours to 72 hours, and >72 hours to 96 hours after the start of initial BRV treatment | <ul> <li>Absolute reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, &gt;3 hours to 6 hours, &gt;6 hours to 12 hours, &gt;12 hours to 24 hours, &gt;24 hours to 36 hours, &gt;36 hours to 48 hours, &gt;48 hours to 72 hours, and &gt;72 hours to 96 hours after the start of initial BRV treatment </li> <li>Percentage reduction from Baseline in seizure burden at evaluation periods of 0 hours to 3 hours, &gt;3 hours to 6 hours, &gt;6 hours to 12 hours, &gt;12 hours to 24 hours, &gt;24 hours to 36 hours, &gt;36 hours to 48 hours, &gt;48 hours to 72 hours, and &gt;72 hours to 96 hours after the start of initial BRV treatment</li> </ul> | Text changes were made to provide consistent language throughout the protocol. |


| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 13.7<br>Handling of<br>dropouts or<br>missing data | For subjects who drop out during the Evaluation Period, the number of hours from the start of the Evaluation Period to the time of withdrawal (in hours) will be considered for analysis. Subjects in the Confirmatory Cohorts who drop out due to lack of BRV efficacy, are switched over to another AED treatment, or are administered >1 dose of rescue medication (including BZDs) following the first 3 hours after initial BRV treatment started will be considered BRV nonresponders. The impact of missing data on the assessment of the main efficacy variable will be evaluated with sensitivity analyses with further details to be included in the SAP. | For subjects who dropped out during the Evaluation Period, the number of hours from the start of the Evaluation Period to the time of withdrawal (in hours) will be considered for analysis. Subjects in the Confirmatory Cohorts who started another AED, increased the dose or frequency of administration of an AED ongoing at the time the first BRV infusion started, or are switched to another AED, or have been administered any rescue medication for the treatment of ENS during the first 3 hours after initiation of BRV treatment will be considered BRV nonresponders. The impact of missing data on the assessment of the main secondary efficacy variable will be evaluated with sensitivity analyses with further details to be included in the SAP. | Clarification And any extensions of the article and any extensions of the article and article |
| Section 13.8.1<br>Exploratory<br>Cohort | That applicable 1/39 | During the DMC review of PK and safety data, the enrollment of subjects will be on hold. | Clarification |
| Confidential | Schlught Califor | | |

| Section<br>Impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 13.9 | No formal sample size calculation has been performed as a single treatment BRV arm is planned for descriptive summary of results and for comparison with the 6 MDZ-treated subjects from the Exploratory Cohort. | No formal sample size calculation has been performed as a single treatment BRV arm is planned for descriptive summary of results and for comparison with the 6 subjects from the Exploratory Cohort. | Text changes were made to provide consistent language throughout the protocol. |


### 17.6 **Protocol Amendment 6**

### Rationale for the amendment

The purpose of this non-substantial amendment is to correct minor inconsistencies of Protocol Amendment 5 identified after finalization.

- Measurement of length before the first administration of BRV was erroneously removed from the Exploratory Cohort in Protocol Amendment 5, and this measurement has been re-inserted.
   The text indicating that Investigation
- before subjects can enter the Evaluation Period was removed in Protocol Amendment 5 from the Exploratory Cohort, but for clarity this has been re-inserted.

## The specific changes include the following:

## Change #1

## **Sponsor Study Physician**

Added to address

## Change #2

## Section 5.1 Study description

COPY and application and any committee of the contraction and any committee of the contraction and any committee of the contraction and any committee of the contraction and any committee of the contraction and any contraction and contraction N01349 consists of 2 steps including a comparison with a historical control group (matched in age and condition) treated with AEDs comparable SOC and diagnostic methods from literature will be used for the evaluation of efficacy.

## Has been changed to:

N01349 consists of a 2-step design and includes a descriptive comparison with a historical control group (matched in age and condition) from literature treated with AEDs per SOC and diagnostic methods.

## Change #3

## **Section 5.1.1 Exploratory Cohort**

The Screening Period starts up to 36 hours prior to the first administration of BRV. Phenobarbital, MDZ, PHT, LEV (≤ 60mg/kg/day), or LDC may have been administered prior to the subject's enrollment into the study and/or at a location other than the study site.

## Has been changed to:

The Screening Period starts up to 36 hours prior to the first administration of BRV. Phenobarbital, MDZ, PHT, LEV, or LDC may have been administered prior to the subject's enrollment into the study and/or at a location other than the study site.

### Change #4

## **Section 5.1.1 Exploratory Cohort**

Table 5-1:

Length during the Screening Period (immediately before first BRV administration) was reinserted as an assessment for the Exploratory Cohort.

Change #6

Section 8.1.1 Screening Period

The following sentence was re-inserted

Preferred by the Inserted Specific Action of the eriod
as re-inserted:
avestigator, the central VEEG reader can be consulted to confirm the control of the control of the confirmation of the confi

### 17.7 **Protocol Amendment 7**

### Rationale for the amendment

The purposes of this substantial amendment are:

- Update the protocol for the new UCB company name (UCB Biopharma SRL).
- Specify the BRV dose recommended by the DMC for the Confirmatory Cohorts.
- Incorporate the measures described in UCB's COVID-19 Contingency Plan for N01349.
- test eclosed.

  .oughout the p.
  .oughout the p. Prolong the BRV Extension Period for up to 90 days postnatal age for sites that may not be
  - Correct minor inconsistencies and apply uniform terminology throughout the protocol.


# Specific changes

| UCB<br>Clinical Study Protocol | | Brivaracetam | 24 May 2021<br>N01349 |
|---|---|---|---|
| Specific changes | | | idiot |
| Section impacted | Key components of previous text | Key components of amended text | Rationale |
| Title page Study contact information | Sponsor: UCB Biopharma<br>SPRL | Sponsor: UCB Biopharma SRL | Sponsor name update |
| Study contact information | Pediatric Neonatologist: | Pediatric Neonatologist: | Change in DMC member |
| Section 1, Summary Section 5.1, Study description Section 5.1.1, Exploratory Cohort | Added text to specify the AEDs enrolled subjects will receive for the Exploratory and Confirmatory Cohorts per SOC. | Per SOC, the AEDs include PB, MDZ, PHT, LEV, or LDC | Alignment with text in Sections 5.1.2 and 8.2.1 |
| Section 1, Summary Section 5.1, Study description Section 5.1.2, Confirmatory Cohort Section 5.4.2, Rationale for dose selection Section 7.2, Treatments to be administered | Added details regarding determination of the BRV dose was determined by the DMC at a meeting held on 05 Nov 2020. | The BRV dose and frequency selected by the DMC for the Confirmatory Cohorts is 1mg/kg bid (2mg/kg/day). Based on data from the Confirmatory Cohorts, the BRV dose may be further adjusted in a staggered approach per DMC discretion. | Specily the BRV dose for the Confirmatory Cohorts as selected by the DMC |
| Section 1, Summary Section 2.3, Rationale for the study Section 5.4.1, Rationale for study design Section 6.1, Inclusion criteria | Present current terminology for corrected gestational age (CGA). | Removed all prior references to postmenstrual age (PMA) and replaced consistently with CGA. | Consistency of terminology throughout the protocol |

| Section impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 1, Summary | No previous text. | Added text describing the possible prolongation of the BRV Extension Period for sites in certain regions that must pause enrollment into N01349 from early Sep 2021 onwards since they may not be ready to transition subjects to the long-term study (EP0156) at the time enrollment into N01266 will be closed. | Flexibility in allowing subjects to remain in N01349 until a long-term study is available. |
| Section 1, Summary Section 8.2.3, BRV Extension Period (Confirmatory Cohorts) | Original text stated that the maximum study duration would be up to 75 days and the maximum BRV exposure would be up to 42 days. | Clarified text to state that the maximum study duration and the maximum BRV exposure are <b>expected to be</b> up to 75 days and up to 42 days, respectively, for most subjects; the exceptions are subjects who remain in the Extension Period for a prolonged duration. New text added to provide the maximum study duration for subjects who remain in the study for up to 90 days of PNA (ie, 130 days [90 days of PNA+ up to 7 days for the Down-Titration Period + up to 33 days for the Safety Follow-Up Period]) | Provide study duration information for subjects who may remain in N01349 for a prolonged Extension Period. |


| variables Exploratory Cohort: Section 8.1.1, Screening Period Section 8.1.2, Evaluation | Heart rate and pulse rate were used interchangeably throughout the protocol. | Heart rate to be presented consistently throughout. | Consistency of terminology |
|---|---|---|---|
| Period In Section 8.1.2, Evaluation | | | throughout the protocol |
| Section 8 1 3 2 Extension | Vital signs (blood pressure, pulse rate, respiratory rate, oxygen saturation [pulse oximetry] including apneas, and body temperature; at 0, 3, 6, 12, 24, and 48 hours) | Vital signs (blood pressure, heart rate, respiratory rate [including apneas], oxygen saturation [pulse oximetry], and body temperature; at 0, 3, 6, 12, 24, and 48 hours) | Revised misleading wording to provide clarification on apneas |
| Section 8.1.3.3,<br>Unscheduled Visits<br>Section 8.1.4, Safety<br>Follow-Up Period | | COPT ion application | |
| Confirmatory Cohorts: Section 8.2.1.1, Baseline Period | | PUBLIC Orland | |
| Section 8.2.2, Evaluation Period Section 8.2.3.2, Extension Period 2 | | Leginos . | |
| Section 8.2.3.3,<br>Unscheduled Visits<br>Section 8.2.4, Down-<br>Litration Period | support and | | |
| Section 8.2.5, Safety<br>Follow-Up Period | ised to | | |
| description | A DMC will be in place for<br>the duration of this study and | Due to the low enrollment rate, the interval between DMC meetings may exceed 6-month intervals, at the discretion of the DMC. | Scheduling flexibility |

| Section impacted | Key components of previous text | Key components of amended text | Rationale Addition |
|---|---|---|---|
| | month intervals between meetings. | | , cs of 1 |
| Section 5.1.2, Confirmatory<br>Cohorts<br>Section 7.2, Treatments to<br>be administered | The dose for subjects in the Confirmatory Cohort was yet to be determined. | Subjects in the Confirmatory Cohorts will receive iv BRV 1mg/kg bid (2mg/kg/day), as recommended by the DMC on 05 Nov 2020. The DMC will continue to monitor the PK and safety of subjects and dosing may be further adjusted in a staggered approach as determined by the DMC. | Updated the previous text to reflect the dose recommended by the DMC on 05 Nov 2020 and to note that the dose may be further adjusted per DMC discretion. |
| Section 5.1.2, Confirmatory<br>Cohorts<br>Section 8.2.3, BRV<br>Extension Period<br>(Confirmatory Cohorts) | The maximum anticipated duration of the BRV Extension Period per subject is up to 28 days of postnatal age (+7 days). | In the event that a long-term study is temporarily not available, subjects are allowed to remain in the BRV Extension Period until they reach a PNA of up to 90 days. For those subjects, the assessments planned for Unscheduled Visits (see Section 8.1,3,3) will be conducted in intervals of approximately 30 days during the prolonged Extension Period. The treatment with BRV will be managed through IVRS. Before subjects can roll-over to the long-term study, they must have switched to BRV oral solution. | Clarification that most subjects will remain in the BRV Extension Period for up to 28 (+7 days) of PNA but that subjects may have a prolonged Extension Period for up to 90 days of PNA if the long-term study is not available at the time planned for the subject's transition. |
| Section 5.1.3, Study<br>duration per subject | The maximum study duration per subject is expected to be up to 75 days | In the event that a long-term study is not available at the time of a subject's planned transition, the maximum study duration for subjects who remain in the study for up to 90 days of PNA and do not enter the long-term study will then be up to 130 days (90 days of PNA, up to 1 week for the Down-Titration Period, and up to 33 days for the Safety Follow-Up Period). | Completeness; added maximum study duration for the subjects who remain for a prolonged BRV Extension Period. |
| Confidential Ancilment Can | | | |
| This | | 1 450 243 01 234 | |

| Section impacted | Key components of previous text | Key components of amended text | Rationale Additional |
|---|---|---|---|
| Section 5.1.3, Study duration per subject | The maximum BRV exposure per subject is expected to be up to 42 days | For subjects who remain in the study for up to 90 days of PNA and do not enter the long-term study, maximum BRV exposure per subject is expected to be up to 97 days (up to 90 days of PNA and up to 1 week for the Down-Titration Period). | Completeness; added maximum BRV exposure for the subjects who remain for a prolonged BRV Extension Period. |
| Section 5.2, Table 5-1<br>Schedule of study | Medical history including<br>Apgar score | Medical history including Apgar score and HIE | Clarification |
| assessments - Screening and Evaluation Periods | AED treatment | Added the specific AEDs per SOC | Clarification |
| (Exploratory Cohort) | Footnote 'j': The recording of AEDs will include BZDs and opiates taken by the mother at the time of delivery. | Added that COVID-19 vaccination will also be recorded as concomitant medication if the mother was pregnant or breastfeeding when vaccinated. | Alignment with the BRV Program Contingency Plan. |
| Section 5.2, Table 5-2<br>Schedule of study | Medical history including Apgar score | Medical history including Apgar score and HIE | Clarification |
| assessments – Screening<br>and Evaluation Periods<br>(Confirmatory Cohorts) | No previously included assessment for neurodevelopmental testing. | Added the Bayley-III assessment at the 96-hour timepoint of the Evaluation Period. | Clarification that subjects completing the Evaluation Period in 28 days of PNA and directly roll over to the long-term study will require that the Bayley assessment be performed at the 96-hour assessment of the Evaluation Period. |
| | Footnote 'h': Subjects are expected to receive IB BRV bid. The dose and dosing frequency of BRV will be adjusted based on the data collected for the analysis of the Exploratory Cohort. | Subjects will receive iv BRV 1mg/kg bid (2mg/kg/day), as recommended by the DMC on 05 Nov 2020 based on the results of the PK analysis of the Exploratory Cohort as well as an existing PK model from N01263. | Updated dose information based on DMC recommendation. |

| Section impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| | Footnote 'n': The recording of AEDs will include BZDs and opiates taken by the mother at the time of delivery. | Added that COVID-19 vaccination will also be recorded as concomitant medication if the mother was pregnant or breastfeeding when vaccinated. | Alignment with the BRV Program Contingency Plan. |
| Section 5.2, Table 5-3 Schedule of study assessments - BRV Extension Period and Safety Follow-Up Period (Exploratory and Confirmatory Cohorts) | Footnote 'b': Subjects will enter the Safety Follow-Up Period if they withdraw from the study at any time, or do not proceed to the BRV Extension Period, or complete the Down-Titration Period. This visit will occur 30±3 days after the last administration of BRV. | Added the following text to the existing footnote text: For subjects unable to return to the hospital due to COVID-19, the Safety Follow-up visit can be performed remotely. In this case vital signs, the physical and neurological examination, biometric and psychometric parameters, and the laboratory assessment may not be performed. | Alignment with the BRV Program Contingency Plan. |
| | Footnote 'k': The recording of AEDs will include BZDs and opiates taken by the mother at the time of delivery. | Added that COVID-19 vaccination will also be recorded as concomitant medication if the mother was pregnant or breastfeeding when vaccinated. | Alignment with the BRV Program Contingency Plan. |
| | Confirmation/diagnosis of epilepsy is planned for EPV1 and EPV2. | Confirmation/diagnosis of epilepsy is only conducted at EPV2 to confirm that the subject qualifies for N01266 or EP0156. | Correction and alignment across sections. |

| Section impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 5.2, Table 5-3 Schedule of study assessments - BRV Extension Period and Safety Follow-Up Period (Exploratory and Confirmatory Cohorts) Section 8.1.3.1, Safety Follow-Up Period (Exploratory Cohort) Section 8.2.3.1, Safety Follow-Up Period (Confirmatory Cohorts) | Footnote 'c': Subjects will attend EPV1 at 7±2 days after completion of the Evaluation Period. | Added the following text to the existing footnote text: For subjects unable to return to the hospital due to COVID-19, EPV1 can be performed remotely if BRV oral solution was dispensed at the time when the subject completed the Evaluation Period. | Alignment with the BRV Program Contingency Plan. |
| Section 5.2, Table 5-3 Schedule of study assessments - BRV Extension Period and Safety Follow-Up Period (Exploratory and Confirmatory Cohorts) Section 8.2.3.3, Unscheduled Visits (Confirmatory Cohorts) | No previous safety laboratory assessments were planned for Unscheduled Visits. | Added footnote 'n' to state "Laboratory assessments (safety) only required for Unscheduled Visits performed during the BRV Extension Period. Added safety laboratory assessments (hematology, biochemistry, liver enzymes, and endocrinology) to Unscheduled Visits. | Alignment with other BRV studies. |
| Section 5.3, Schematic diagrams Figure 5-1, Schematic Overview of the study (Exploratory Cohort) | Presents Evaluation Period as 96 hours and is missing the Screening Period timeframe. | The Evaluation Period is 48 hours and the Screening Period is up to 36 hours in duration. | Error correction and addition of additional information |
| Figure 5-2, Screening and Evaluation Periods (Exploratory Cohort) | Administration of AED per SOC first line-, second line-, and third line-treatments | Administration of one or more of the following AEDs: PB, MDZ, PHT, LEV, or LDC | Consistency with updated text describing AED administration per SOC |

Confidential Currient

| Section impacted | Key components of previous text | Key components of amended text | Rationale Addition |
|---|---|---|---|
| Figure 5-3, Schematic overview of the study (Confirmatory Cohorts) | Missing Screening Period timeframe. Missing duration of BRV Extension Period for subjects with a prolonged duration of up to 90 days of PNA. | The Screening Period is up to 36 hours in duration. Added duration of BRV Extension Period for subjects with a prolonged duration. | Error correction New information. |
| Figure 5-4, Screening and Evaluation Periods (Confirmatory Cohorts) | Administration of AED per<br>SOC first line-, second line-,<br>and third line-treatments | Administration of one or more of the following AEDs: PB, MDZ, PHT, LEV (≤60mg/kg/day), or LDC | Consistency with updated text describing AED administration per SOC |
| Section 6.2, Exclusion criteria | Exclusion criterion #2: Subjects with seizures responding to previous AED treatment immediately prior to BRV treatment, pyridoxine treatment, or correction of metabolic disturbances (hypoglycemia, hypomagnesemia, or | Subject with seizures <u>responding</u> to any of the following; previous AED treatment immediately prior to BRV treatment, pyridoxine treatment, or correction of metabolic disturbances (hypoglycemia, hypomagnesemia, or hypocalcemia). | Clarify that previous pyridoxine treatment is not an exclusion criterion; subjects are excluded if they responded to pyridoxine treatment. |


| Section impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 7.2, Treatments to be administered | Subjects in the Exploratory Cohort will be dosed with BRV (0.5mg/kg bid) according to the sites standard procedures. Administration of BRV is proposed as approximately 15-minute iv infusions. Treatment with previous AEDs (PB, MDZ, PHT, LEV [≤60mg/kg/day], or LDC) is permitted to continue if the subject is on a stable dose from 1 hour prior to initiation of the BRV treatment. | Subjects in the Exploratory Cohort will be dosed during the Evaluation Period with BRV (0.5mg/kg bid) according to the sites standard procedures. Administration of BRV is proposed as approximately 15-minute iv infusions. Treatment with previous AEDs (PB, MDZ, PHT, LEV [≤60mg/kg/day], or LDC) during the Evaluation Period is permitted to continue if the subject is on a stable dose from 1 hour prior to initiation of the BRV treatment. | Clarify that the dosing of subjects in the Exploratory Cohort with BRV 0.5mg/kg bid will occur during the Evaluation Period. Clarify that treatment with previous AEDs is permitted during the Evaluation Period |
| Section 8.1.3, BRV<br>Extension Period<br>(Exploratory Cohort) | No previous text describing the purpose of the BRV Extension Period. | The BRV Extension Period is intended to bridge the time until subjects are old enough to participate in the long-term study. Subjects completing the Evaluation Period at a PNA of at least 28 days may directly roll over to the long-term study, if they meet the eligibility criteria. Those patients are not required to enter the BRV Extension Period. | Clarify the purpose of the BRV<br>Extension Period |
| | Added text clarifying that subjects not continuing BRV treatment after the Evaluation Period will enter the Safety Follow-Up Period and not the BRV Extension Period | Subjects not continuing the BRV treatment after they completed the Evaluation Period will not enter the BRV Extension Period but proceed immediately to the Safety Follow-Up Period | Clarification of study design |
| Confidential Hochmant Call | | | |

| Section impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 8.1.4, Safety Follow-Up Visit (Exploratory Cohort) Section 8.2.5, Safety Follow-Up Visit (Confirmatory Cohort) | No previous text | For subjects unable to return to the hospital due to COVID-19, the Safety Follow-Up Visit can be performed remotely. In this case vital signs, the physical and neurological examination, biometric and psychometric parameters, and the laboratory assessment may not be performed. | Alignment with the BRV Program Contingency Plan. |
| Section 8.2.2 Evaluation<br>Period (Confirmatory<br>Cohort) | No previous text describing the number of doses administered in the Confirmatory Cohorts. | Up to 8 iv doses of BRV (1mg/kg bid) will be administered as an approximately 15-minute infusion during the 96-hour BRV Evaluation Period. | Clarify the number of BRV doses administered in the Confirmatory Cohorts. |
| Section 8.2.2 Evaluation<br>Period (Confirmatory<br>Cohort) | BRV infusion (dose and dosing frequency of BRV to be confirmed after analysis of the data collected for the Exploratory Cohort). | Evaluation Period. Text removed. | Text no longer applicable since<br>the DMC has determined the dose<br>for the Confirmatory Cohorts |
| Section 8.2.2 Evaluation<br>Period (Confirmatory<br>Cohorts) | No previous text | Added Bayley-III as an assessment to be performed following BRV administration during the Evaluation Period for subjects in the Confirmatory Cohort who are continuing into the long-term study and enrolled in countries where a validated translation is available. | Clarification that subjects completing the Evaluation Period in 28 days of PNA and directly roll over to the long-term study will require that the Bayley assessment be performed at the 96-hour assessment of the Evaluation Period. |
| Confidential Hochment can | not be used to support any mai | | |
| Confidential ACUIT | | | |
| This | | | |

| Section impacted | Key components of previous text | Key components of amended text | Rationale |
|---|---|---|---|
| Section 8.2.3 BRV<br>Extension Period<br>(Confirmatory Cohorts) | No previous text describing the purpose of the BRV Extension Period. | The BRV Extension Period is intended to bridge the time until subjects are old enough to participate in the long-term study. Subjects completing the Evaluation Period at a PNA of at least 28 days may directly roll over to the long-term study, if they meet the eligibility criteria. Those patients are not required to enter the BRV Extension Period. | Clarify the purpose of the BRV Extension Period |
| | Subjects not entering the BRV Extension Period will proceed immediately to the Down-Titration Period (see Section 8.2.4). | Subjects not continuing the BRV treatment after they completed the Evaluation Period will not enter the BRV Extension Period but proceed immediately to the Down-Titration Period | Clarification |
| Section 8.2.3.3,<br>Unscheduled Visit<br>(Confirmatory Cohort) | No previous text | For subjects who remain in the BRV Extension Period for a prolonged duration (ie, until they reach a PNA of 90 days), these assessments will be conducted at intervals of 30 (±3 days). | Provide the assessment schedule for subjects who remain for a prolonged BRV Extension Period. |
| Confidential Hochment Can | not be used to support any man | | |
| Confidential Action | | | |
| Klyis | | | |

## 18 DECLARATION AND SIGNATURE OF INVESTIGATOR

I confirm that I have carefully read and understood this protocol and agree to conduct this clinical study as outlined in this protocol, according to current Good Clinical Practice and local laws and requirements.

I will ensure that all subinvestigators and other staff members read and understand all aspects of this protocol.

I have received and read all study-related information provided to me.

The objectives and content of this protocol as well as the results deriving from it will be treated confidentially and will not be made available to third parties without prior authorization by UCB.

All rights of publication of the results reside with UCB, unless other agreements were made in a separate contract.

| Investigator: | ad and exte |
|---|---|
| Printed name | Date/Signature Date/Signature Ratheting authorization are a second control of the seco |
| | all cortation at |
| | Rolling arithe |
| the s. | Mark |
| A to SUPPOI | |
| othe used | |
| at canine | |

This document compute seed to support any more support support any more support and support any more support any more support any more support and support any more support and support any more support and support and support any more support and sup


# **Approval Signatures**

| Version: | 2. 0 | |
|---|---|---|
| Document Number: | CLIN-000174213 | Approvals |
| Title: | n01349 Protocol Amendmer | ot 7 |
| | | E OI VO |
| Approved Date: | 25 May 2021 | nsions |
| | | oties. |
| | | ad and |
| | | in our of |
| | Document | Approvals |
| Approval | | Name: |
| Verdict: Approved | | Capacity: Clinical Date of Signature: 25-May-2021 14:37:55 GMT+0000 |
| Approval | EURPORT any marketing authorities | Name: Capacity: Subject Matter Expert |
| Verdict: Approved | de lines | Date of Signature: 25-May-2021 14:40:08 GMT+0000 |
| Approval | Musi | Name: Capacity: Clinical |
| Verdict: Approved | - A A A A A A A A A A A A A A A A A A A | Date of Signature: 25-May-2021 14:55:14 GMT+0000 |
| cument cannot be used to | SUPP | |
| .sed* | ) | |
| * pe Jis | | |
| Edinor | | |
| nento | | |
| CITA | | |